CLINICAL TRIAL: NCT01218113
Title: Efficacy and Safety of HIV Vaccine 732462 in ART-naïve HIV-1 Infected Persons
Brief Title: Efficacy and Safety of GSK Biologicals HIV Vaccine in Antiretroviral Therapy (ART)-naïve HIV-1 Infected Persons
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111679
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-03

CONDITIONS: AIDS
Keywords: Human Immunodeficiency Virus (HIV)-1; safety; vaccine; immunogenicity; reactogenicity; HIV infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 3D_HIV Group (Experimental): HIV-1 infected male and female subjects, between and including 18 to 55 years of age at the time of first vaccination, who received 3 doses of the HIV Vaccine 732462 at Weeks 0, 4 and 28, administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: GSK Biologicals HIV Vaccine 732462
- 2D_HIV Group (Experimental): HIV-1 infected male and female subjects, between and including 18 to 55 years of age at the time of first vaccination, who received 2 doses of the HIV Vaccine 732462 at Weeks 0 and 4 and one dose of placebo (saline solution) at Week 28, administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: GSK Biologicals HIV Vaccine 732462; Drug: Placebo
- Control Group (Placebo Comparator): HIV-1 infected male and female subjects, between and including 18 to 55 years of age at the time of first vaccination, who received 3 doses of placebo (saline solution) at Weeks 0, 4 and 28, administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: GSK Biologicals HIV Vaccine 732462 — 2 or 3 doses according to protocol schedule
  Arms: 2D_HIV Group; 3D_HIV Group
Drug: Placebo — 1 or 3 doses according to protocol schedule
  Arms: 2D_HIV Group; Control Group

SUMMARY:
This study is designed to determine whether administration of the GSK Biologicals HIV vaccine 732462 can lead to a reduction in viral load, and impact on the course of human immunodeficiency virus type 1 (HIV-1) infection. In HIV-1 infected persons who have not yet started antiretroviral therapy (ART), such a vaccine would potentially lead to a delay in the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to any study procedure.
* A male or female between and including 18-55 years at the time of first vaccination.
* Known to be HIV-1 infected and under the care of an HIV physician for a minimum of 6 months. However, subjects who initially presented with a clinical diagnosis of primary HIV infection need to have been diagnosed and under care for at least 12 months.
* ART-naïve. Individuals must never have received ART after HIV diagnosis, including lamivudine used for chronic hepatitis B infection, with the exception of short-term ART for prevention of mother-to-child transmission (PMTCT) at least 12 months prior to enrollment.
* Commencement of ART is not expected, based on current assessment, within the next 12 months.
* Viral load level of 2,000-80,000 copies/mL at screening.
* CD4 count >= 500 cells per mm3 at screening.
* If the subject is female, she must be of non-childbearing potential, i.e. have a current tubal ligation, hysterectomy, ovariectomy or be post-menopausal. Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test at screening, and
  * has agreed to continue adequate contraception during the entire study period.

Exclusion Criteria:

The following criteria should be checked at the time of screening and before vaccination. If ANY exclusion criterion applies, the subject must not be included in the study:

* Infection with HIV-2. This includes patients with dual infection with HIV-1/HIV-2.
* Had an Acquired Immune Deficiency Syndrome (AIDS) defining clinical illness.
* Use of any investigational or non-registered product within 4 weeks preceding the first dose of study vaccine/placebo, or planned use of any investigational or non-registered product other than the study vaccine during the study period.
* Drug therapy with immunomodulators or steroids within the 12 weeks preceding the first dose of study vaccine/placebo or planned administration during the study period. Acute use of steroids up to 4 weeks preceding the first dose for treatment of hypersensitivity reactions is not an exclusion criterion. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/ or any blood products within the 12 weeks preceding the first dose of study vaccine/placebo or planned administration during the study period.
* Planned administration of a vaccine not foreseen by the study protocol during

  * the period starting 2 weeks before the first dose of study vaccine/placebo and ending at Visit 3 (Week 6) (after blood sampling),
  * the period starting from 2 weeks prior to Visit 5 (Week 28) and ending at Visit 6 (Week 30) (after blood sampling)
  * the period starting from 2 weeks prior to Visit 8 (Week 48) and ending at Visit 8 (Week 48) (after blood sampling), with the exception of non-adjuvanted influenza vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any previous vaccination or immunotherapy against HIV.
* A family history of hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute or chronic infective hepatitis.
* Acute or chronic, clinically relevant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination and/or medical history at screening.
* Grade 3 or grade 4 laboratory abnormality, as defined by Division od AIDS (DAIDS) grading table, at screening
* Pregnant or lactating female.
* Any condition which, in the opinion of the investigator, could compromise the subject's safety or adherence to the study protocol.
* History of medically confirmed autoimmune disease.
* History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure.
* Unstable asthma
* Food or wine induced asthma.
* Known sensitivity to sulfites or aspirin.
* Known sensitivity to aminoglycoside antibiotics.
* Contraindication to intramuscular injection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 191 (Actual)
Dates: Start 2010-11-08 (Actual); Primary Completion 2012-11-05 (Actual); Study Completion 2012-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (16):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Seattle, Washington
- France (4):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (6):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
- Spain (5):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles, Madrid
  - GSK Investigational Site, Valencia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 191 subjects originally enrolled in the study, only 190 subjects received vaccination and were hence included in the Total Vaccinated Cohort.
Period: Overall Study
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Started | 62 | 64 | 64
Completed | 57 | 63 | 58
Not Completed | 5 | 1 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 4 | 1 | 4
Not completed — Protocol Deviation Eligibility Criteria | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group | Total
Number analyzed (Participants) | 62 | 64 | 64 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.9 (7.6) | 37.0 (8.2) | 35.9 (8.4) | 35.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 29
  Male | 53 | 54 | 54 | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African heritage/African American | 11 | 10 | 15 | 36
  Race/Ethnicity: American Indian or Alaskan Native | 0 | 0 | 2 | 2
  Race/Ethnicity: White-Arabic/North African heritage | 4 | 3 | 3 | 10
  Race/Ethnicity: White-Caucasian/European heritage | 43 | 51 | 42 | 136
  Race/Ethnicity: Other | 4 | 0 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Change in Human Immunodeficiency Virus Type 1 (HIV-1) Viral Load (VL) From Baseline
Description: Changes from baseline in HIV-1 viral load (ratio of each value over baseline value) were obtained using crude values and expressed in RNA copies/milliliter [copies/mL]. Baseline of HIV-1 viral load was defined as geometric mean of values measured in blood samples taken at Screening and at Week 0. The HIV type 1, represents the more aggressive virus form, largely responsible for the AIDS pandemic.
Time Frame: At Week 48, post-Dose 3
Population: The analysis was performed on the Modified Total vaccinated cohort, which included all subjects with at least one vaccine administration documented who complied with the protocol-defined criteria and with sufficient data to perform the efficacy analysis.
Measure: Geometric Mean (Standard Deviation); unit: RNA copies/mL
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 46 | 55 | 50
RNA copies/mL | 1.0 (0.35) | 1.5 (0.38) | 1.3 (0.34)
Statistical Analysis 1: Comparison: 3D_HIV Group vs Control Group; To show the difference in change from baseline of HIV-1 VL at week 48 between persons who received 3 doses of the HIV vaccine 732462 and persons who received placebo alone; Test type: Non-Inferiority — Crierion for non-inferiority evaluation: The upper limit (UL) of the two-sided 97.5% confidence interval (CI) for the difference in change between the two arms (3D_HIV Group - Control Group) is below 0; Repeated-measures mixed model; Geometric Mean Ratio = 0.801, 97.5% CI 2-sided [0.553 to 1.162]
Statistical Analysis 2: Comparison: 2D_HIV Group vs Control Group; To show the difference in change from baseline of HIV-1 VL at week 48 between persons who received 2 doses of the HIV Vaccine 732462 and persons who received placebo alone; Test type: Non-Inferiority — Crierion for non-inferiority evaluation: The upper limit (UL) of the two-sided 97.5% confidence interval (CI) for the difference in change between the two arms (2D_HIV Group - Control Group) is below 0; Repeated-measures mixed model; Geometric Mean Ratio = 1.184, 97.5% CI 2-sided [0.816 to 1.717]

2. Primary Outcome: Geometric Mean Change in HIV-1 VL From Baseline
Description: Changes from baseline in HIV-1 viral load (difference of each value minus baseline value) were obtained using log10-transformed values and expressed in log10-RNA copies/mL. Baseline of HIV-1 viral load was defined as geometric mean of values measured in blood samples taken at Screening and at Week 0. The HIV type 1, represents the more aggressive virus form, largely responsible for the AIDS pandemic.
Time Frame: At Week 48, post-Dose 3
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: log10(RNA copies/mL)
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 46 | 55 | 50
log10(RNA copies/mL) | 0.0 (0.35) | 0.2 (0.38) | 0.1 (0.34)
Statistical Analysis 1: Comparison: 3D_HIV Group vs Control Group; To show the difference in change from baseline of HIV-1 VL (log10-transformed values) at week 48 between persons who received 3 doses of the HIV Vaccine 732462 and persons who received placebo alone; Test type: Non-Inferiority — Criterion for non-inferiority evaluation: The upper limit (UL) of the two-sided 97.5% confidence interval (CI) for the difference in change between the two arms (3D_HIV Group - Control Group) is below 0; Repeated-measures mixed model; Mean Difference = -0.096, 97.5% CI 2-sided [-0.257 to 0.065]
Statistical Analysis 2: Comparison: 2D_HIV Group vs Control Group; To show the difference in change from baseline of HIV-1 VL (log10-transformed values) at week 48 between persons who received 2 doses of the HIV Vaccine 732462 and persons who received placebo alone; Test type: Non-Inferiority — Criterion for non-inferiority evaluation: The upper limit (UL) of the two-sided 97.5% confidence interval (CI) for the difference in change between the two arms (2D_HIV Group - Control Group) is below 0; Repeated-measures mixed model; Mean Difference = 0.073, 97.5% CI 2-sided [-0.088 to 0.235]

3. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of symptom regardless of intensity. Grade 3 Pain = pain that prevented normal every day activities. Grade 3 Redness/Swelling = redness or swelling associated with ulceration or secondary infection/phlebitis/sterile abscess/drainage. Medically attended (MA) Pain = pain causing inability to perform basic self-care function or Hospitalization indicated for management of pain. Medically attended Redness/Swelling = redness or swelling associated with necrosis.
Time Frame: During the 7-day (Days 0-6) period following Dose 1
Population: The analysis was performed on the Total Vaccinated cohort, which included subjects with at least one vaccine administration documented, who had their symptom sheets filled in. For the purpose of the analysis, 3D_HIV Group and 2D_HIV Group were combined into a single group (HIV Group), since Dose 1 vaccination was identical for both groups.
Measure: Count of Participants; unit: Participants
Groups:
- HIV Group: HIV-1 infected male and female subjects, between and including 18 to 55 years of age at the time of first vaccination, who received 2 doses of the HIV Vaccine 732462 at Weeks 0 and 4, administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 125 | 63
Participants
  Any Pain, Dose 1 | 112 | 12
  Grade 3 Pain, Dose 1 | 9 | 0
  Medically attended Pain, Dose 1 | 0 | 0
  Any Redness, Dose 1 | 16 | 0
  Grade 3 Redness, Dose 1 | 0 | 0
  Medically attended Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 7 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0
  Medically attended Swelling, Dose 1 | 0 | 0

4. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: as for outcome 3
Time Frame: During the 7-day (Days 0-6) period following Dose 2
Population: The analysis was performed on the Total Vaccinated cohort, which included subjects with at least one vaccine administration documented, who had their symptom sheets filled in. For the purpose of the analysis, 3D_HIV Group and 2D_HIV Group were combined into a single group (HIV Group), since Dose 2 vaccination was identical for both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 120 | 61
Participants
  Any Pain, Dose 2 | 98 | 5
  Grade 3 Pain, Dose 2 | 11 | 0
  Medically Attended Pain, Dose 2 | 0 | 0
  Any Redness, Dose 2 | 15 | 0
  Grade 3 Redness, Dose 2 | 0 | 0
  Medically Attended Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2 | 6 | 0
  Grade 3 Swelling, Dose 2 | 0 | 0
  Medically Attended Swelling, Dose 2 | 0 | 0

5. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: as for outcome 3
Time Frame: During the 7-day (Days 0-6) period following Dose 3
Population: The analysis was performed on the Total Vaccinated cohort, which included subjects with at least one vaccine administration documented, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 55 | 58 | 54
Participants
  Any Pain, Dose 3 | 42 | 9 | 3
  Grade 3 Pain, Dose 3 | 6 | 0 | 0
  Medically attended Pain, Dose 3 | 0 | 0 | 0
  Any Redness, Dose 3 | 10 | 0 | 0
  Grade 3 Redness, Dose 3 | 0 | 0 | 0
  Medically attended Redness, Dose 3 | 0 | 0 | 0
  Any Swelling, Dose 3 | 3 | 0 | 0
  Grade 3 Swelling, Dose 3 | 0 | 0 | 0
  Medically attended Swelling, Dose 3 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: as for outcome 3
Time Frame: During the 7-day (Days 0-6) post-vaccination period, across doses
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 62 | 64 | 64
Participants
  Any Pain, Across doses | 58 | 57 | 14
  Grade 3 Pain, Across doses | 15 | 6 | 0
  Medically Attended Pain, Across doses | 0 | 0 | 0
  Any Redness, Across doses | 17 | 14 | 0
  Grade 3 Redness, Across doses | 0 | 0 | 0
  Medically Attended Redness, Across doses | 0 | 0 | 0
  Any Swelling, Across doses | 4 | 8 | 0
  Grade 3 Swelling, Across doses | 0 | 0 | 0
  Medically Attended Swelling, Across doses | 0 | 0 | 0

7. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms(smt.)were abdominalpain,anorexia,diarrhoea,fatigue,headache,myalgia,nausea,sweating,temperature(Temp.)orally=temp.37.7degreesCelsius(°C)&vomiting.Any=occurrene of smt.regardless of intensity.Grade3(G3)Abdominal pain/fatigue/myalgia/sweating/headache=symp.causing inability to perform usual social&functional activities.Medicallyattended(MA)Abdominalpain/fatigue/myalgia/sweating/headache=smt.causing inability to perform basic self-care activities.G3Anorexia=loss of appetite associated with significant weight loss.MAanorexia=aggressive intervention indicated.G3diarrhoea=blood/increased≥7stools per24hours(h)/4fluid replacement.G3nausea=persistent nausea resulting in minimal oral intake for more than48h/with aggressive rehydration indicated.G3vomiting=persistent vomiting resulting in orthostatic hypotension/aggressive.MAdiarrhoea/nausea/vomiting=smt.with life threatening consequences.Related=smt.assessed by the investigator as being related to vaccination
Time Frame: During the 7-day (Days 0-6) period following Dose 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 124 | 63
Participants
  Any Abdominal pain, Dose 1 | 14 | 3
  Grade 3 Abdominal pain, Dose 1 | 0 | 0
  Related Abdominal pain, Dose 1 | 2 | 0
  Grade 3 Related Abdominal pain, Dose 1 | 0 | 0
  Medically Attended Abdominal pain, Dose 1 | 1 | 0
  Any Anorexia, Dose 1 | 7 | 2
  Grade 3 Anorexia, Dose 1 | 0 | 0
  Related Anorexia, Dose 1 | 4 | 0
  Grade 3 Related Anorexia, Dose 1 | 0 | 0
  Medically Attended Anorexia, Dose 1 | 0 | 0
  Any Diarrhoea, Dose 1 | 16 | 5
  Grade 3 Diarrhoea, Dose 1 | 1 | 0
  Related Diarrhoea, Dose 1 | 1 | 0
  Grade 3 Related Diarrhoea, Dose 1 | 0 | 0
  Medically Attended Diarrhoea, Dose 1 | 1 | 0
  Any Fatigue, Dose 1 | 56 | 16
  Grade 3 Fatigue, Dose 1 | 3 | 1
  Related Fatigue, Dose 1 | 24 | 7
  Grade 3 Related Fatigue, Dose 1 | 1 | 0
  Medically Attended Fatigue, Dose 1 | 0 | 0
  Any Headache, Dose 1 | 40 | 14
  Grade 3 Headache, Dose 1 | 4 | 1
  Related Headache, Dose 1 | 16 | 8
  Grade 3 Related Headache, Dose 1 | 4 | 0
  Medically Attended Headache, Dose 1 | 0 | 1
  Any Myalgia, Dose 1 | 44 | 9
  Grade 3 Myalgia, Dose 1 | 2 | 0
  Related Myalgia, Dose 1 | 26 | 4
  Grade 3 Related Myalgia, Dose 1 | 1 | 0
  Medically Attended Myalgia, Dose 1 | 0 | 0
  Any Nausea, Dose 1 | 17 | 5
  Grade 3 Nausea, Dose 1 | 1 | 0
  Related Nausea, Dose 1 | 4 | 2
  Grade 3 Related Nausea, Dose 1 | 0 | 0
  Medically Attended Nausea, Dose 1 | 0 | 0
  Any Sweating, Dose 1 | 16 | 6
  Grade 3 Sweating, Dose 1 | 1 | 0
  Related Sweating, Dose 1 | 3 | 1
  Grade 3 Related Sweating, Dose 1 | 0 | 0
  Medically Attended Sweating, Dose 1 | 0 | 0
  Any Temperature, Dose 1 | 8 | 2
  Grade 3 Temperature, Dose 1 | 1 | 0
  Related Temperature, Dose 1 | 3 | 0
  Grade 3 Related Temperature, Dose 1 | 0 | 0
  Medically Attended Temperature, Dose 1 | 1 | 0
  Any Vomiting, Dose 1 | 2 | 1
  Grade 3 Vomiting, Dose 1 | 0 | 0
  Related Vomiting, Dose 1 | 1 | 0
  Grade 3 Related Vomiting, Dose 1 | 0 | 0
  Medically Attended Vomiting, Dose 1 | 0 | 0

8. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: as for outcome 7
Time Frame: During the 7-day (Days 0-6) period following Dose 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 120 | 61
Participants
  Any Abdominal pain, Dose 2 | 9 | 1
  Grade 3 Abdominal Pain, Dose 2 | 1 | 0
  Related Abdominal Pain, Dose 2 | 3 | 0
  Grade 3 Related Abdominal Pain, Dose 2 | 0 | 0
  Medically Attended Abdominal Pain, Dose 2 | 1 | 0
  Any Anorexia, Dose 2 | 7 | 2
  Grade 3 Anorexia, Dose 2 | 1 | 0
  Related Anorexia, Dose 2 | 3 | 0
  Grade 3 Related Anorexia, Dose 2 | 0 | 0
  Medically Attended Anorexia, Dose 2 | 1 | 0
  Any Diarrhoea, Dose 2 | 13 | 7
  Grade 3 Diarrhoea, Dose 2 | 0 | 0
  Related Diarrhoea, Dose 2 | 2 | 1
  Grade 3 Related Diarrhoea, Dose 2 | 0 | 0
  Medically Attended Diarrhoea, Dose 2 | 0 | 0
  Any Fatigue, Dose 2 | 56 | 10
  Grade 3 Fatigue, Dose 2 | 6 | 2
  Related Fatigue, Dose 2 | 25 | 4
  Grade 3 Related Fatigue, Dose 2 | 4 | 1
  Medically Attended Fatigue, Dose 2 | 2 | 0
  Any Headache, Dose 2 | 34 | 8
  Grade 3 Headache, Dose 2 | 5 | 1
  Related Headache, Dose 2 | 15 | 3
  Grade 3 Related Headache, Dose 2 | 3 | 0
  Medically Attended Headache, Dose 2 | 1 | 0
  Any Myalgia, Dose 2 | 42 | 6
  Grade 3 Myalgia, Dose 2 | 6 | 1
  Related Myalgia, Dose 2 | 26 | 1
  Grade 3 Related Myalgia, Dose 2 | 6 | 0
  Medically Attended Myalgia, Dose 2 | 1 | 1
  Any Nausea, Dose 2 | 11 | 0
  Grade 3 Nausea, Dose 2 | 0 | 0
  Related Nausea, Dose 2 | 4 | 0
  Grade 3 Related Nausea, Dose 2 | 0 | 0
  Medically Attended Nausea, Dose 2 | 1 | 0
  Any Sweating, Dose 2 | 17 | 3
  Grade 3 Sweating, Dose 2 | 2 | 0
  Related Sweating, Dose 2 | 8 | 0
  Grade 3 Related Sweating, Dose 2 | 2 | 0
  Medically Attended Sweating, Dose 2 | 1 | 0
  Any Temperature, Dose 2 | 11 | 3
  Grade 3 Temperature, Dose 2 | 0 | 0
  Related Temperature, Dose 2 | 7 | 0
  Grade 3 Related Temperature, Dose 2 | 0 | 0
  Medically Attended Temperature, Dose 2 | 1 | 1
  Any Vomiting, Dose 2 | 2 | 1
  Grade 3 Vomiting, Dose 2 | 0 | 0
  Related Vomiting, Dose 2 | 0 | 0
  Grade 3 Related Vomiting, Dose 2 | 0 | 0
  Medically Attended Vomiting, Dose 2 | 0 | 0

9. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: as for outcome 7
Time Frame: During the 7-day (Days 0-6) period following Dose 3
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 56 | 58 | 54
Participants
  Any Abdominal pain, Dose 3 | 4 | 4 | 2
  Grade 3 Abdominal pain, Dose 3 | 0 | 2 | 0
  Related Abdominal pain, Dose 3 | 1 | 1 | 0
  Grade 3 Related Abdominal pain, Dose 3 | 0 | 1 | 0
  Medically Attende Abdominal pain, Dose 3 | 1 | 1 | 0
  Any Anorexia, Dose 3 | 7 | 3 | 3
  Grade 3 Anorexia, Dose 3 | 0 | 0 | 0
  Related Anorexia, Dose 3 | 3 | 0 | 0
  Grade 3 Related Anorexia, Dose 3 | 0 | 0 | 0
  Medically Attended Anorexia, Dose 3 | 0 | 0 | 0
  Any Diarrhoea, Dose 3 | 8 | 12 | 5
  Grade 3 Diarrhoea, Dose 3 | 0 | 0 | 1
  Related Diarrhoea, Dose 3 | 4 | 3 | 1
  Grade 3 Related Diarrhoea, Dose 3 | 0 | 0 | 0
  Medically Attended Diarrhoea, Dose 3 | 1 | 0 | 0
  Any Fatigue, Dose 3 | 25 | 11 | 8
  Grade 3 Fatigue, Dose 3 | 3 | 2 | 1
  Related Fatigue, Dose 3 | 15 | 3 | 2
  Grade 3 Related Fatigue, Dose 3 | 1 | 0 | 0
  Medically Attended Fatigue, Dose 3 | 0 | 0 | 0
  Any Headache, Dose 3 | 16 | 17 | 7
  Grade 3 Headache, Dose 3 | 1 | 1 | 0
  Related Headache, Dose 3 | 8 | 5 | 1
  Grade 3 Related Headache, Dose 3 | 1 | 0 | 0
  Medically Attended Headache, Dose 3 | 2 | 1 | 0
  Any Myalgia, Dose 3 | 19 | 9 | 4
  Grade 3 Myalgia, Dose 3 | 2 | 1 | 0
  Related Myalgia, Dose 3 | 13 | 3 | 1
  Grade 3 Related Myalgia, Dose 3 | 1 | 0 | 0
  Medically Attended Myalgia, Dose 3 | 0 | 1 | 0
  Any Nausea, Dose 3 | 7 | 2 | 3
  Grade 3 Nausea, Dose 3 | 0 | 0 | 0
  Related Nausea, Dose 3 | 3 | 0 | 0
  Grade 3 Related Nausea, Dose 3 | 0 | 0 | 0
  Medically Attended Nausea, Dose 3 | 0 | 0 | 0
  Any Sweating, Dose 3 | 7 | 8 | 2
  Grade 3 Sweating, Dose 3 | 0 | 0 | 0
  Related Sweating, Dose 3 | 4 | 1 | 0
  Grade 3 Related Sweating, Dose 3 | 0 | 0 | 0
  Medically Attended Sweating, Dose 3 | 0 | 0 | 0
  Any Temperature, Dose 3 | 5 | 3 | 1
  Grade 3 Temperature, Dose 3 | 1 | 0 | 0
  Related Temperature, Dose 3 | 4 | 0 | 0
  Grade 3 Related Temperature, Dose 3 | 1 | 0 | 0
  Medically Attended Temperature, Dose 3 | 0 | 0 | 0
  Any Vomiting, Dose 3 | 2 | 0 | 1
  Grade 3 Vomiting, Dose 3 | 0 | 0 | 0
  Related Vomiting, Dose 3 | 1 | 0 | 0
  Grade 3 Related Vomiting, Dose 3 | 0 | 0 | 0
  Medically Attended Vomiting, Dose 3 | 0 | 0 | 0

10. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: as for outcome 7
Time Frame: During the 7-day (Days 0-6) post-vaccination period, across doses
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 62 | 64 | 64
Participants
  Any Abdominal pain, Across doses | 13 | 10 | 4
  Grade 3 Abdominal pain, Across doses | 1 | 2 | 0
  Related Abdominal pain, Across doses | 3 | 3 | 0
  Grade 3 Related Abdominal pain, Across doses | 0 | 1 | 0
  Medically Attended Abdominal pain, Across doses | 3 | 1 | 0
  Any Anorexia, Across doses | 11 | 10 | 7
  Grade 3 Anorexia, Across doses | 1 | 0 | 0
  Related Anorexia, Across doses | 5 | 4 | 0
  Grade 3 Related Anorexia, Across doses | 0 | 0 | 0
  Medically Attended Anorexia, Across doses | 0 | 1 | 0
  Any Diarrhoea, Across doses | 17 | 19 | 14
  Grade 3 Diarrhoea, Across doses | 1 | 0 | 1
  Related Diarrhoea, Across doses | 5 | 4 | 2
  Grade 3 Related Diarrhoea, Across doses | 0 | 0 | 0
  Medically Attended Diarrhoea, Across doses | 2 | 0 | 0
  Any Fatigue, Across doses | 43 | 38 | 20
  Grade 3 Fatigue, Across doses | 8 | 4 | 3
  Related Fatigue, Across doses | 24 | 24 | 9
  Grade 3 Related Fatigue, Across doses | 3 | 2 | 1
  Medically Attended Fatigue, Across doses | 1 | 1 | 0
  Any Headache, Across doses | 32 | 33 | 21
  Grade 3 Headache, Across doses | 4 | 4 | 1
  Related Headache, Across doses | 15 | 17 | 11
  Grade 3 Related Headache, Across doses | 3 | 2 | 0
  Medically Attended Headache, Across doses | 2 | 2 | 1
  Any Myalgia, Across doses | 33 | 32 | 12
  Grade 3 Myalgia, Across doses | 4 | 5 | 1
  Related Myalgia, Across doses | 22 | 21 | 4
  Grade 3 Related Myalgia, Across doses | 2 | 4 | 0
  Medically Attended Myalgia, Across doses | 0 | 2 | 1
  Any Nausea, Across doses | 17 | 14 | 8
  Grade 3 Nausea, Across doses | 1 | 0 | 0
  Related Nausea, Across doses | 7 | 4 | 2
  Grade 3 Related Nausea, Across doses | 0 | 0 | 0
  Medically Attended Nausea, Across doses | 1 | 0 | 0
  Any Sweating, Across doses | 11 | 20 | 10
  Grade 3 Sweating, Across doses | 1 | 2 | 0
  Related Sweating, Across doses | 6 | 7 | 1
  Grade 3 Related Sweating, Across doses | 1 | 1 | 0
  Medically Attended Sweating, Across doses | 0 | 1 | 0
  Any Temperature, Across doses | 14 | 9 | 6
  Grade 3 Temperature, Across doses | 2 | 0 | 0
  Related Temperature, Across doses | 9 | 4 | 0
  Grade 3 Related Temperature, Across doses | 1 | 0 | 0
  Medically Attended Temperature, Across doses | 1 | 1 | 1
  Any Vomiting, Across doses | 3 | 2 | 3
  Grade 3 Vomiting, Across doses | 0 | 0 | 0
  Related Vomiting, Across doses | 2 | 0 | 0
  Grade 3 Related Vomiting, Across doses | 0 | 0 | 0
  Medically Attended Vomiting, Across doses | 0 | 0 | 0

11. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 (G3) AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination. Unsolicited AEs were tabulated following Dose 1 and Dose 2 vaccinations.
Time Frame: During the 28-Day (Days 0-27) period following Dose 1 and Dose 2
Population: The analysis was performed on the Total Vaccinated cohort, which included subjects with at least one vaccine administration documented. For the purpose of the analysis, 3D_HIV Group and 2D_HIV Group were combined into a single group (HIV Group), since Dose 1 and 2 vaccinations were identical for both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 126 | 64
Participants
  Any AE(s) | 58 | 29
  Grade 3 AE(s) | 9 | 3
  Related AE(s) | 6 | 2
  Grade 3 Related AE(s) | 1 | 0
  Medically Attended AE(s) | 17 | 13

12. Primary Outcome: Number of Subjects With Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 (G3) AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination. Unsolicited AEs were tabulated following Dose 3 and across doses.
Time Frame: During the 28-Day (Days 0-27) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 56 | 60 | 56
Participants
  Any AE(s) | 30 | 42 | 34
  Grade 3 AE(s) | 3 | 7 | 3
  Related AE(s) | 2 | 6 | 2
  Grade 3 Related AE(s) | 0 | 1 | 0
  Medically Attended AE(s) | 11 | 14 | 15

13. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (up to Week 48)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 62 | 64 | 64
Participants | 1 | 3 | 2

14. Primary Outcome: Number of Subjects With Potentially Immune-Mediated Diseases (pIMDs)
Description: Potentially Immune-Mediated Diseases (pIMDs) are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
Time Frame: During the entire study period (up to Week 48)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 62 | 64 | 64
Participants | 0 | 1 | 0

15. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: Among the biochemical and haematological parameters with abnormal values were alanine aminotransferase [ALT], albumin [ALB], alkaline phosphatase [ALP], aspartate aminotransferase [AST], bilirubin (total) [BIL], creatinine [CRE], eosinophils [EOS], eosinophils/100 leukocytes [EOS/100LEU], bicarbonate [BIC], haemoglobin [HGB], potassium [PTS], lymphocytes [LYM], lymphocytes/100 leukocytes [LYM/100LEU], sodium [SDI], neutrophils [NEU], neutrophils/100 leukocytes [NEU/100LEU], platelet count [PLC], prothrombin time-international normalized ratio [PTT] and white blood cell count [WBC]. Assessed grades (G) for laboratory parameters were 0, 1 (mild), 2 (moderate), 3 (severe) and 4 (potentially life-threatening), according to DAIDS (division of AIDS table for grading the severity of adult and pediatric adverse events -Version 1.0).
Time Frame: At Screening
Population: The analysis was performed on the Total Vaccinated cohort, which included subjects with at least one vaccine administration documented. For the purpose of the analysis, 3D_HIV Group and 2D_HIV Group were combined into a single group (HIV Group), since the screening timepoint was identical for both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 126 | 64
Participants
  ALT, Grade 0 | 115 | 63
  ALT, Grade 1 | 9 | 1
  ALT, Grade 2 | 2 | 0
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 0 | 0
  ALB, Grade 0 | 126 | 64
  ALB, Grade 1 | 0 | 0
  ALB, Grade 2 | 0 | 0
  ALB, Grade 3 | 0 | 0
  ALB, Grade 4 | 0 | 0
  ALP, Grade 0 | 125 | 64
  ALP, Grade 1 | 1 | 0
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grade 0 | 120 | 63
  AST, Grade 1 | 6 | 1
  AST, Grade 2 | 0 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0
  BIL, Grade 0 | 123 | 63
  BIL, Grade 1 | 2 | 0
  BIL, Grade 2 | 1 | 1
  BIL, Grade 3 | 0 | 0
  BIL, Grade 4 | 0 | 0
  CRE, Grade 0 | 124 | 62
  CRE, Grade 1 | 2 | 1
  CRE, Grade 2 | 0 | 1
  CRE, Grade 3 | 0 | 0
  CRE, Grade 4 | 0 | 0
  EOS, Grade 0 | 124 | 64
  EOS, Grade 1 | 0 | 0
  EOS, Grade 2 | 0 | 0
  EOS, Grade 3 | 0 | 0
  EOS, Grade 4 | 0 | 0
  EOS/100LEU, Grade 0 | 124 | 64
  EOS/100LEU, Grade 1 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0
  BIC, Grade 0 | 118 | 59
  BIC, Grade 1 | 8 | 5
  BIC, Grade 2 | 0 | 0
  BIC, Grade 3 | 0 | 0
  BIC, Grade 4 | 0 | 0
  HGB, Grade 0 | 126 | 64
  HGB, Grade 1 | 0 | 0
  HGB, Grade 2 | 0 | 0
  HGB, Grade 3 | 0 | 0
  HGB, Grade 4 | 0 | 0
  PTS, Grade 0 | 126 | 64
  PTS, Grade 1 | 0 | 0
  PTS, Grade 2 | 0 | 0
  PTS, Grade 3 | 0 | 0
  PTS, Grade 4 | 0 | 0
  LYM, Grade 0 | 124 | 64
  LYM, Grade 1 | 0 | 0
  LYM, Grade 2 | 0 | 0
  LYM, Grade 3 | 0 | 0
  LYM, Grade 4 | 0 | 0
  LYM/100LEU, Grade 0 | 124 | 64
  LYM/100LEU, Grade 1 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0
  SDI, Grade 0 | 115 | 63
  SDI, Grade 1 | 11 | 1
  SDI, Grade 2 | 0 | 0
  SDI, Grade 3 | 0 | 0
  SDI, Grade 4 | 0 | 0
  NEU, Grade 0 | 119 | 64
  NEU, Grade 1 | 3 | 0
  NEU, Grade 2 | 2 | 0
  NEU, Grade 3 | 0 | 0
  NEU, Grade 4 | 0 | 0
  NEU/100LEU, Grade 0 | 124 | 64
  NEU/100LEU, Grade 1 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0
  PLC, Grade 0 | 122 | 63
  PLC, Grade 1 | 2 | 0
  PLC, Grade 2 | 0 | 1
  PLC, Grade 3 | 0 | 0
  PLC, Grade 4 | 0 | 0
  PTT, Grade 0 | 116 | 59
  PTT, Grade 1 | 10 | 4
  PTT, Grade 2 | 0 | 0
  PTT, Grade 3 | 0 | 0
  PTT, Grade 4 | 0 | 0
  WBC, Grade 0 | 126 | 64
  WBC, Grade 1 | 0 | 0
  WBC, Grade 2 | 0 | 0
  WBC, Grade 3 | 0 | 0
  WBC, Grade 4 | 0 | 0

16. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: as for outcome 15
Time Frame: Pre-vaccination, at Week 0
Population: The analysis was performed on the Total Vaccinated cohort, which included subjects with at least one vaccine administration documented. For the purpose of the analysis, 3D_HIV Group and 2D_HIV Group were combined into a single group (HIV Group), since Dose 1 vaccination was identical for both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 126 | 64
Participants
  ALT, Grade 0 | 117 | 62
  ALT, Grade 1 | 6 | 2
  ALT, Grade 2 | 3 | 0
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 0 | 0
  ALB, Grade 0 | 125 | 64
  ALB, Grade 1 | 1 | 0
  ALB, Grade 2 | 0 | 0
  ALB, Grade 3 | 0 | 0
  ALB, Grade 4 | 0 | 0
  ALP, Grade 0 | 125 | 64
  ALP, Grade 1 | 1 | 0
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grade 0 | 121 | 61
  AST, Grade 1 | 3 | 3
  AST, Grade 2 | 2 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0
  BIL, Grade 0 | 125 | 63
  BIL, Grade 1 | 1 | 0
  BIL, Grade 2 | 0 | 1
  BIL, Grade 3 | 0 | 0
  BIL, Grade 4 | 0 | 0
  CRE, Grade 0 | 125 | 61
  CRE, Grade 1 | 0 | 3
  CRE, Grade 2 | 1 | 0
  CRE, Grade 3 | 0 | 0
  CRE, Grade 4 | 0 | 0
  EOS, Grade 0 | 126 | 64
  EOS, Grade 1 | 0 | 0
  EOS, Grade 2 | 0 | 0
  EOS, Grade 3 | 0 | 0
  EOS, Grade 4 | 0 | 0
  EOS/100LEU, Grade 0 | 126 | 64
  EOS/100LEU, Grade 1 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0
  BIC, Grade 0 | 100 | 47
  BIC, Grade 1 | 26 | 17
  BIC, Grade 2 | 0 | 0
  BIC, Grade 3 | 0 | 0
  BIC, Grade 4 | 0 | 0
  HGB, Grade 0 | 126 | 64
  HGB, Grade 1 | 0 | 0
  HGB, Grade 2 | 0 | 0
  HGB, Grade 3 | 0 | 0
  HGB, Grade 4 | 0 | 0
  PTS, Grade 0 | 126 | 64
  PTS, Grade 1 | 0 | 0
  PTS, Grade 2 | 0 | 0
  PTS, Grade 3 | 0 | 0
  PTS, Grade 4 | 0 | 0
  LYM, Grade 0 | 126 | 64
  LYM, Grade 1 | 0 | 0
  LYM, Grade 2 | 0 | 0
  LYM, Grade 3 | 0 | 0
  LYM, Grade 4 | 0 | 0
  LYM/100LEU, Grade 0 | 126 | 64
  LYM/100LEU, Grade 1 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0
  SDI, Grade 0 | 114 | 59
  SDI, Grade 1 | 11 | 5
  SDI, Grade 2 | 1 | 0
  SDI, Grade 3 | 0 | 0
  SDI, Grade 4 | 0 | 0
  NEU, Grade 0 | 123 | 62
  NEU, Grade 1 | 2 | 0
  NEU, Grade 2 | 1 | 2
  NEU, Grade 3 | 0 | 0
  NEU, Grade 4 | 0 | 0
  NEU/100LEU, Grade 0 | 126 | 64
  NEU/100LEU, Grade 1 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0
  PLC, Grade 0 | 121 | 63
  PLC, Grade 1 | 5 | 0
  PLC, Grade 2 | 0 | 1
  PLC, Grade 3 | 0 | 0
  PLC, Grade 4 | 0 | 0
  PTT, Grade 0 | 118 | 55
  PTT, Grade 1 | 7 | 9
  PTT, Grade 2 | 1 | 0
  PTT, Grade 3 | 0 | 0
  PTT, Grade 4 | 0 | 0
  WBC, Grade 0 | 125 | 63
  WBC, Grade 1 | 0 | 0
  WBC, Grade 2 | 1 | 1
  WBC, Grade 3 | 0 | 0
  WBC, Grade 4 | 0 | 0

17. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: as for outcome 15
Time Frame: At Week 4
Population: The analysis was performed on the Total Vaccinated cohort, which included subjects with at least one vaccine administration documented. For the purpose of the analysis, 3D_HIV Group and 2D_HIV Group were combined into a single group (HIV Group), since Dose 1 and Dose 2 vaccinations were identical for both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 126 | 64
Participants
  ALT, Grade 0 | 114 | 62
  ALT, Grade 1 | 10 | 0
  ALT, Grade 2 | 2 | 1
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 0 | 0
  ALB, Grade 0 | 125 | 63
  ALB, Grade 1 | 1 | 0
  ALB, Grade 2 | 0 | 0
  ALB, Grade 3 | 0 | 0
  ALB, Grade 4 | 0 | 0
  ALP, Grade 0 | 124 | 63
  ALP, Grade 1 | 2 | 0
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grade 0 | 119 | 61
  AST, Grade 1 | 5 | 2
  AST, Grade 2 | 2 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0
  BIL, Grade 0 | 125 | 63
  BIL, Grade 1 | 1 | 0
  BIL, Grade 2 | 0 | 0
  BIL, Grade 3 | 0 | 0
  BIL, Grade 4 | 0 | 0
  CRE, Grade 0 | 121 | 61
  CRE, Grade 1 | 5 | 2
  CRE, Grade 2 | 0 | 0
  CRE, Grade 3 | 0 | 0
  CRE, Grade 4 | 0 | 0
  EOS, Grade 0 | 126 | 63
  EOS, Grade 1 | 0 | 0
  EOS, Grade 2 | 0 | 0
  EOS, Grade 3 | 0 | 0
  EOS, Grade 4 | 0 | 0
  EOS/100LEU, Grade 0 | 126 | 63
  EOS/100LEU, Grade 1 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0
  BIC, Grade 0 | 99 | 48
  BIC, Grade 1 | 27 | 15
  BIC, Grade 2 | 0 | 0
  BIC, Grade 3 | 0 | 0
  BIC, Grade 4 | 0 | 0
  HGB, Grade 0 | 126 | 63
  HGB, Grade 1 | 0 | 0
  HGB, Grade 2 | 0 | 0
  HGB, Grade 3 | 0 | 0
  HGB, Grade 4 | 0 | 0
  PTS, Grade 0 | 124 | 63
  PTS, Grade 1 | 2 | 0
  PTS, Grade 2 | 0 | 0
  PTS, Grade 3 | 0 | 0
  PTS, Grade 4 | 0 | 0
  LYM, Grade 0 | 126 | 63
  LYM, Grade 1 | 0 | 0
  LYM, Grade 2 | 0 | 0
  LYM, Grade 3 | 0 | 0
  LYM, Grade 4 | 0 | 0
  LYM/100LEU, Grade 0 | 126 | 63
  LYM/100LEU, Grade 1 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0
  SDI, Grade 0 | 119 | 60
  SDI, Grade 1 | 7 | 3
  SDI, Grade 2 | 0 | 0
  SDI, Grade 3 | 0 | 0
  SDI, Grade 4 | 0 | 0
  NEU, Grade 0 | 122 | 62
  NEU, Grade 1 | 4 | 1
  NEU, Grade 2 | 0 | 0
  NEU, Grade 3 | 0 | 0
  NEU, Grade 4 | 0 | 0
  NEU/100LEU, Grade 0 | 126 | 63
  NEU/100LEU, Grade 1 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0
  PLC, Grade 0 | 123 | 62
  PLC, Grade 1 | 2 | 0
  PLC, Grade 2 | 1 | 1
  PLC, Grade 3 | 0 | 0
  PLC, Grade 4 | 0 | 0
  PTT, Grade 0 | 115 | 54
  PTT, Grade 1 | 11 | 9
  PTT, Grade 2 | 0 | 0
  PTT, Grade 3 | 0 | 0
  PTT, Grade 4 | 0 | 0
  WBC, Grade 0 | 126 | 63
  WBC, Grade 1 | 0 | 0
  WBC, Grade 2 | 0 | 0
  WBC, Grade 3 | 0 | 0
  WBC, Grade 4 | 0 | 0

18. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: as for outcome 15
Time Frame: At Week 6
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 126 | 64
Participants
  ALT, Grade 0 | 117 | 60
  ALT, Grade 1 | 5 | 2
  ALT, Grade 2 | 3 | 0
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 0 | 0
  ALB, Grade 0 | 124 | 62
  ALB, Grade 1 | 1 | 0
  ALB, Grade 2 | 0 | 0
  ALB, Grade 3 | 0 | 0
  ALB, Grade 4 | 0 | 0
  ALP, Grade 0 | 123 | 62
  ALP, Grade 1 | 2 | 0
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grade 0 | 118 | 61
  AST, Grade 1 | 6 | 1
  AST, Grade 2 | 1 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0
  BIL, Grade 0 | 121 | 62
  BIL, Grade 1 | 4 | 0
  BIL, Grade 2 | 0 | 0
  BIL, Grade 3 | 0 | 0
  BIL, Grade 4 | 0 | 0
  CRE, Grade 0 | 119 | 60
  CRE, Grade 1 | 6 | 2
  CRE, Grade 2 | 0 | 0
  CRE, Grade 3 | 0 | 0
  CRE, Grade 4 | 0 | 0
  EOS, Grade 0 | 125 | 62
  EOS, Grade 1 | 0 | 0
  EOS, Grade 2 | 0 | 0
  EOS, Grade 3 | 0 | 0
  EOS, Grade 4 | 0 | 0
  EOS/100LEU, Grade 0 | 125 | 62
  EOS/100LEU, Grade 1 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0
  BIC, Grade 0 | 92 | 39
  BIC, Grade 1 | 33 | 23
  BIC, Grade 2 | 0 | 0
  BIC, Grade 3 | 0 | 0
  BIC, Grade 4 | 0 | 0
  HGB, Grade 0 | 125 | 62
  HGB, Grade 1 | 0 | 0
  HGB, Grade 2 | 0 | 0
  HGB, Grade 3 | 0 | 0
  HGB, Grade 4 | 0 | 0
  PTS, Grade 0 | 124 | 60
  PTS, Grade 1 | 1 | 2
  PTS, Grade 2 | 0 | 0
  PTS, Grade 3 | 0 | 0
  PTS, Grade 4 | 0 | 0
  LYM, Grade 0 | 125 | 62
  LYM, Grade 1 | 0 | 0
  LYM, Grade 2 | 0 | 0
  LYM, Grade 3 | 0 | 0
  LYM, Grade 4 | 0 | 0
  LYM/100LEU, Grade 0 | 125 | 62
  LYM/100LEU, Grade 1 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0
  SDI, Grade 0 | 117 | 58
  SDI, Grade 1 | 7 | 4
  SDI, Grade 2 | 1 | 0
  SDI, Grade 3 | 0 | 0
  SDI, Grade 4 | 0 | 0
  NEU, Grade 0 | 121 | 62
  NEU, Grade 1 | 3 | 0
  NEU, Grade 2 | 1 | 0
  NEU, Grade 3 | 0 | 0
  NEU, Grade 4 | 0 | 0
  NEU/100LEU, Grade 0 | 125 | 62
  NEU/100LEU, Grade 1 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0
  PLC, Grade 0 | 122 | 61
  PLC, Grade 1 | 3 | 0
  PLC, Grade 2 | 0 | 0
  PLC, Grade 3 | 0 | 1
  PLC, Grade 4 | 0 | 0
  PTT, Grade 0 | 118 | 51
  PTT, Grade 1 | 7 | 11
  PTT, Grade 2 | 0 | 0
  PTT, Grade 3 | 0 | 0
  PTT, Grade 4 | 0 | 0
  WBC, Grade 0 | 125 | 62
  WBC, Grade 1 | 0 | 0
  WBC, Grade 2 | 0 | 0
  WBC, Grade 3 | 0 | 0
  WBC, Grade 4 | 0 | 0

19. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: as for outcome 15
Time Frame: At Week 16
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 126 | 64
Participants
  ALT, Grade 0 | 113 | 60
  ALT, Grade 1 | 10 | 0
  ALT, Grade 2 | 1 | 1
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 0 | 0
  ALB, Grade 0 | 123 | 61
  ALB, Grade 1 | 1 | 0
  ALB, Grade 2 | 0 | 0
  ALB, Grade 3 | 0 | 0
  ALB, Grade 4 | 0 | 0
  ALP, Grade 0 | 122 | 61
  ALP, Grade 1 | 2 | 0
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grade 0 | 117 | 59
  AST, Grade 1 | 6 | 2
  AST, Grade 2 | 1 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0
  BIL, Grade 0 | 124 | 59
  BIL, Grade 1 | 0 | 1
  BIL, Grade 2 | 0 | 1
  BIL, Grade 3 | 0 | 0
  BIL, Grade 4 | 0 | 0
  CRE, Grade 0 | 119 | 60
  CRE, Grade 1 | 5 | 1
  CRE, Grade 2 | 0 | 0
  CRE, Grade 3 | 0 | 0
  CRE, Grade 4 | 0 | 0
  EOS, Grade 0 | 124 | 61
  EOS, Grade 1 | 0 | 0
  EOS, Grade 2 | 0 | 0
  EOS, Grade 3 | 0 | 0
  EOS, Grade 4 | 0 | 0
  EOS/100LEU, Grade 0 | 124 | 61
  EOS/100LEU, Grade 1 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0
  BIC, Grade 0 | 93 | 47
  BIC, Grade 1 | 31 | 14
  BIC, Grade 2 | 0 | 0
  BIC, Grade 3 | 0 | 0
  BIC, Grade 4 | 0 | 0
  HGB, Grade 0 | 122 | 61
  HGB, Grade 1 | 2 | 0
  HGB, Grade 2 | 0 | 0
  HGB, Grade 3 | 0 | 0
  HGB, Grade 4 | 0 | 0
  PTS, Grade 0 | 123 | 61
  PTS, Grade 1 | 1 | 0
  PTS, Grade 2 | 0 | 0
  PTS, Grade 3 | 0 | 0
  PTS, Grade 4 | 0 | 0
  LYM, Grade 0 | 124 | 61
  LYM, Grade 1 | 0 | 0
  LYM, Grade 2 | 0 | 0
  LYM, Grade 3 | 0 | 0
  LYM, Grade 4 | 0 | 0
  LYM/100LEU, Grade 0 | 124 | 61
  LYM/100LEU, Grade 1 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0
  SDI, Grade 0 | 121 | 58
  SDI, Grade 1 | 3 | 3
  SDI, Grade 2 | 0 | 0
  SDI, Grade 3 | 0 | 0
  SDI, Grade 4 | 0 | 0
  NEU, Grade 0 | 121 | 60
  NEU, Grade 1 | 2 | 1
  NEU, Grade 2 | 1 | 0
  NEU, Grade 3 | 0 | 0
  NEU, Grade 4 | 0 | 0
  NEU/100LEU, Grade 0 | 124 | 61
  NEU/100LEU, Grade 1 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0
  PLC, Grade 0 | 119 | 60
  PLC, Grade 1 | 4 | 1
  PLC, Grade 2 | 1 | 0
  PLC, Grade 3 | 0 | 0
  PLC, Grade 4 | 0 | 0
  PTT, Grade 0 | 111 | 55
  PTT, Grade 1 | 13 | 6
  PTT, Grade 2 | 0 | 0
  PTT, Grade 3 | 0 | 0
  PTT, Grade 4 | 0 | 0
  WBC, Grade 0 | 124 | 61
  WBC, Grade 1 | 0 | 0
  WBC, Grade 2 | 0 | 0
  WBC, Grade 3 | 0 | 0
  WBC, Grade 4 | 0 | 0

20. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: as for outcome 15
Time Frame: At Week 28
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 126 | 64
Participants
  ALT, Grade 0 | 112 | 57
  ALT, Grade 1 | 5 | 2
  ALT, Grade 2 | 3 | 1
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 1 | 0
  ALB, Grade 0 | 121 | 60
  ALB, Grade 1 | 0 | 0
  ALB, Grade 2 | 0 | 0
  ALB, Grade 3 | 0 | 0
  ALB, Grade 4 | 0 | 0
  ALP, Grade 0 | 121 | 60
  ALP, Grade 1 | 0 | 0
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grade 0 | 115 | 57
  AST, Grade 1 | 4 | 3
  AST, Grade 2 | 1 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 1 | 0
  BIL, Grade 0 | 119 | 59
  BIL, Grade 1 | 1 | 0
  BIL, Grade 2 | 1 | 1
  BIL, Grade 3 | 0 | 0
  BIL, Grade 4 | 0 | 0
  CRE, Grade 0 | 119 | 59
  CRE, Grade 1 | 2 | 0
  CRE, Grade 2 | 0 | 1
  CRE, Grade 3 | 0 | 0
  CRE, Grade 4 | 0 | 0
  EOS, Grade 0 | 121 | 60
  EOS, Grade 1 | 0 | 0
  EOS, Grade 2 | 0 | 0
  EOS, Grade 3 | 0 | 0
  EOS, Grade 4 | 0 | 0
  EOS/100LEU, Grade 0 | 121 | 60
  EOS/100LEU, Grade 1 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0
  BIC, Grade 0 | 92 | 45
  BIC, Grade 1 | 29 | 15
  BIC, Grade 2 | 0 | 0
  BIC, Grade 3 | 0 | 0
  BIC, Grade 4 | 0 | 0
  HGB, Grade 0 | 120 | 59
  HGB, Grade 1 | 1 | 1
  HGB, Grade 2 | 0 | 0
  HGB, Grade 3 | 0 | 0
  HGB, Grade 4 | 0 | 0
  PTS, Grade 0 | 120 | 60
  PTS, Grade 1 | 1 | 0
  PTS, Grade 2 | 0 | 0
  PTS, Grade 3 | 0 | 0
  PTS, Grade 4 | 0 | 0
  LYM, Grade 0 | 121 | 60
  LYM, Grade 1 | 0 | 0
  LYM, Grade 2 | 0 | 0
  LYM, Grade 3 | 0 | 0
  LYM, Grade 4 | 0 | 0
  LYM/100LEU, Grade 0 | 121 | 60
  LYM/100LEU, Grade 1 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0
  SDI, Grade 0 | 115 | 57
  SDI, Grade 1 | 6 | 3
  SDI, Grade 2 | 0 | 0
  SDI, Grade 3 | 0 | 0
  SDI, Grade 4 | 0 | 0
  NEU, Grade 0 | 115 | 58
  NEU, Grade 1 | 3 | 2
  NEU, Grade 2 | 3 | 0
  NEU, Grade 3 | 0 | 0
  NEU, Grade 4 | 0 | 0
  NEU/100LEU, Grade 0 | 121 | 60
  NEU/100LEU, Grade 1 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0
  PLC, Grade 0 | 118 | 59
  PLC, Grade 1 | 2 | 0
  PLC, Grade 2 | 1 | 1
  PLC, Grade 3 | 0 | 0
  PLC, Grade 4 | 0 | 0
  PTT, Grade 0 | 110 | 54
  PTT, Grade 1 | 11 | 6
  PTT, Grade 2 | 0 | 0
  PTT, Grade 3 | 0 | 0
  PTT, Grade 4 | 0 | 0
  WBC, Grade 0 | 121 | 60
  WBC, Grade 1 | 0 | 0
  WBC, Grade 2 | 0 | 0
  WBC, Grade 3 | 0 | 0
  WBC, Grade 4 | 0 | 0

21. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: as for outcome 15
Time Frame: At Week 30
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | 3D_HIV Group | 2D_HIV Group
Number analyzed (Participants) | 64 | 62 | 64
Participants
  ALT, Grade 0 | 53 | 54 | 57
  ALT, Grade 1 | 5 | 2 | 1
  ALT, Grade 2 | 0 | 1 | 1
  ALT, Grade 3 | 0 | 0 | 0
  ALT, Grade 4 | 0 | 0 | 1
  ALB, Grade 0 | 57 | 57 | 60
  ALB, Grade 1 | 1 | 0 | 0
  ALB, Grade 2 | 0 | 0 | 0
  ALB, Grade 3 | 0 | 0 | 0
  ALB, Grade 4 | 0 | 0 | 0
  ALP, Grade 0 | 58 | 56 | 60
  ALP, Grade 1 | 0 | 1 | 0
  ALP, Grade 2 | 0 | 0 | 0
  ALP, Grade 3 | 0 | 0 | 0
  ALP, Grade 4 | 0 | 0 | 0
  AST, Grade 0 | 55 | 54 | 58
  AST, Grade 1 | 3 | 3 | 1
  AST, Grade 2 | 0 | 0 | 0
  AST, Grade 3 | 0 | 0 | 1
  AST, Grade 4 | 0 | 0 | 0
  BIL, Grade 0 | 55 | 57 | 59
  BIL, Grade 1 | 3 | 0 | 1
  BIL, Grade 2 | 0 | 0 | 0
  BIL, Grade 3 | 0 | 0 | 0
  BIL, Grade 4 | 0 | 0 | 0
  CRE, Grade 0 | 57 | 55 | 59
  CRE, Grade 1 | 1 | 2 | 1
  CRE, Grade 2 | 0 | 0 | 0
  CRE, Grade 3 | 0 | 0 | 0
  CRE, Grade 4 | 0 | 0 | 0
  EOS, Grade 0 | 58 | 57 | 60
  EOS, Grade 1 | 0 | 0 | 0
  EOS, Grade 2 | 0 | 0 | 0
  EOS, Grade 3 | 0 | 0 | 0
  EOS, Grade 4 | 0 | 0 | 0
  EOS/100LEU, Grade 0 | 58 | 57 | 60
  EOS/100LEU, Grade 1 | 0 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0 | 0
  BIC, Grade 0 | 43 | 45 | 45
  BIC, Grade 1 | 15 | 12 | 15
  BIC, Grade 2 | 0 | 0 | 0
  BIC, Grade 3 | 0 | 0 | 0
  BIC, Grade 4 | 0 | 0 | 0
  HGB, Grade 0 | 57 | 56 | 60
  HGB, Grade 1 | 0 | 1 | 0
  HGB, Grade 2 | 0 | 0 | 0
  HGB, Grade 3 | 1 | 0 | 0
  HGB, Grade 4 | 0 | 0 | 0
  PTS, Grade 0 | 58 | 56 | 60
  PTS, Grade 1 | 0 | 1 | 0
  PTS, Grade 2 | 0 | 0 | 0
  PTS, Grade 3 | 0 | 0 | 0
  PTS, Grade 4 | 0 | 0 | 0
  LYM, Grade 0 | 58 | 57 | 60
  LYM, Grade 1 | 0 | 0 | 0
  LYM, Grade 2 | 0 | 0 | 0
  LYM, Grade 3 | 0 | 0 | 0
  LYM, Grade 4 | 0 | 0 | 0
  LYM/100LEU, Grade 0 | 58 | 57 | 60
  LYM/100LEU, Grade 1 | 0 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0 | 0
  SDI, Grade 0 | 51 | 55 | 59
  SDI, Grade 1 | 7 | 2 | 1
  SDI, Grade 2 | 0 | 0 | 0
  SDI, Grade 3 | 0 | 0 | 0
  SDI, Grade 4 | 0 | 0 | 0
  NEU, Grade 0 | 55 | 53 | 58
  NEU, Grade 1 | 3 | 4 | 2
  NEU, Grade 2 | 0 | 0 | 0
  NEU, Grade 3 | 0 | 0 | 0
  NEU, Grade 4 | 0 | 0 | 0
  NEU/100LEU, Grade 0 | 58 | 57 | 60
  NEU/100LEU, Grade 1 | 0 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0 | 0
  PLC, Grade 0 | 58 | 56 | 59
  PLC, Grade 1 | 0 | 1 | 0
  PLC, Grade 2 | 0 | 0 | 1
  PLC, Grade 3 | 0 | 0 | 0
  PLC, Grade 4 | 0 | 0 | 0
  PTT, Grade 0 | 53 | 51 | 56
  PTT, Grade 1 | 5 | 6 | 4
  PTT, Grade 2 | 0 | 0 | 0
  PTT, Grade 3 | 0 | 0 | 0
  PTT, Grade 4 | 0 | 0 | 0
  WBC, Grade 0 | 58 | 57 | 60
  WBC, Grade 1 | 0 | 0 | 0
  WBC, Grade 2 | 0 | 0 | 0
  WBC, Grade 3 | 0 | 0 | 0
  WBC, Grade 4 | 0 | 0 | 0

22. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: as for outcome 15
Time Frame: At Week 38
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | 3D_HIV Group | 2D_HIV Group
Number analyzed (Participants) | 64 | 62 | 64
Participants
  ALT, Grade 0 | 53 | 52 | 61
  ALT, Grade 1 | 4 | 3 | 1
  ALT, Grade 2 | 0 | 2 | 1
  ALT, Grade 3 | 1 | 0 | 0
  ALT, Grade 4 | 0 | 0 | 0
  ALB, Grade 0 | 57 | 57 | 63
  ALB, Grade 1 | 0 | 0 | 0
  ALB, Grade 2 | 1 | 0 | 0
  ALB, Grade 3 | 0 | 0 | 0
  ALB, Grade 4 | 0 | 0 | 0
  ALP, Grade 0 | 58 | 55 | 63
  ALP, Grade 1 | 0 | 2 | 0
  ALP, Grade 2 | 0 | 0 | 0
  ALP, Grade 3 | 0 | 0 | 0
  ALP, Grade 4 | 0 | 0 | 0
  AST, Grade 0 | 55 | 52 | 61
  AST, Grade 1 | 2 | 4 | 2
  AST, Grade 2 | 1 | 1 | 0
  AST, Grade 3 | 0 | 0 | 0
  AST, Grade 4 | 0 | 0 | 0
  BIL, Grade 0 | 56 | 57 | 61
  BIL, Grade 1 | 1 | 0 | 1
  BIL, Grade 2 | 1 | 0 | 1
  BIL, Grade 3 | 0 | 0 | 0
  BIL, Grade 4 | 0 | 0 | 0
  CRE, Grade 0 | 56 | 54 | 61
  CRE, Grade 1 | 2 | 3 | 2
  CRE, Grade 2 | 0 | 0 | 0
  CRE, Grade 3 | 0 | 0 | 0
  CRE, Grade 4 | 0 | 0 | 0
  EOS, Grade 0 | 58 | 57 | 63
  EOS, Grade 1 | 0 | 0 | 0
  EOS, Grade 2 | 0 | 0 | 0
  EOS, Grade 3 | 0 | 0 | 0
  EOS, Grade 4 | 0 | 0 | 0
  EOS/100LEU, Grade 0 | 58 | 57 | 63
  EOS/100LEU, Grade 1 | 0 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0 | 0
  BIC, Grade 0 | 46 | 47 | 51
  BIC, Grade 1 | 11 | 10 | 12
  BIC, Grade 2 | 1 | 0 | 0
  BIC, Grade 3 | 0 | 0 | 0
  BIC, Grade 4 | 0 | 0 | 0
  HGB, Grade 0 | 57 | 56 | 63
  HGB, Grade 1 | 0 | 1 | 0
  HGB, Grade 2 | 0 | 0 | 0
  HGB, Grade 3 | 0 | 0 | 0
  HGB, Grade 4 | 1 | 0 | 0
  PTS, Grade 0 | 57 | 57 | 61
  PTS, Grade 1 | 1 | 0 | 2
  PTS, Grade 2 | 0 | 0 | 0
  PTS, Grade 3 | 0 | 0 | 0
  PTS, Grade 4 | 0 | 0 | 0
  LYM, Grade 0 | 58 | 57 | 63
  LYM, Grade 1 | 0 | 0 | 0
  LYM, Grade 2 | 0 | 0 | 0
  LYM, Grade 3 | 0 | 0 | 0
  LYM, Grade 4 | 0 | 0 | 0
  LYM/100LEU, Grade 0 | 58 | 57 | 63
  LYM/100LEU, Grade 1 | 0 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0 | 0
  SDI, Grade 0 | 54 | 54 | 61
  SDI, Grade 1 | 4 | 3 | 2
  SDI, Grade 2 | 0 | 0 | 0
  SDI, Grade 3 | 0 | 0 | 0
  SDI, Grade 4 | 0 | 0 | 0
  NEU, Grade 0 | 56 | 54 | 59
  NEU, Grade 1 | 2 | 2 | 3
  NEU, Grade 2 | 0 | 1 | 1
  NEU, Grade 3 | 0 | 0 | 0
  NEU, Grade 4 | 0 | 0 | 0
  NEU/100LEU, Grade 0 | 58 | 57 | 63
  NEU/100LEU, Grade 1 | 0 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0 | 0
  PLC, Grade 0 | 58 | 55 | 59
  PLC, Grade 1 | 0 | 2 | 3
  PLC, Grade 2 | 0 | 0 | 1
  PLC, Grade 3 | 0 | 0 | 0
  PLC, Grade 4 | 0 | 0 | 0
  PTT, Grade 0 | 51 | 52 | 55
  PTT, Grade 1 | 7 | 5 | 7
  PTT, Grade 2 | 0 | 0 | 0
  PTT, Grade 3 | 0 | 0 | 1
  PTT, Grade 4 | 0 | 0 | 0
  WBC, Grade 0 | 58 | 56 | 63
  WBC, Grade 1 | 0 | 1 | 0
  WBC, Grade 2 | 0 | 0 | 0
  WBC, Grade 3 | 0 | 0 | 0
  WBC, Grade 4 | 0 | 0 | 0

23. Primary Outcome: Number of Subjects With Abnormal Haematological and Biochemical Values
Description: as for outcome 15
Time Frame: At Week 48
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | 3D_HIV Group | 2D_HIV Group
Number analyzed (Participants) | 64 | 62 | 64
Participants
  ALT, Grade 0 | 52 | 55 | 61
  ALT, Grade 1 | 3 | 1 | 2
  ALT, Grade 2 | 2 | 1 | 0
  ALT, Grade 3 | 1 | 0 | 0
  ALT, Grade 4 | 0 | 0 | 0
  ALB, Grade 0 | 58 | 56 | 63
  ALB, Grade 1 | 0 | 1 | 0
  ALB, Grade 2 | 0 | 0 | 0
  ALB, Grade 3 | 0 | 0 | 0
  ALB, Grade 4 | 0 | 0 | 0
  ALP, Grade 0 | 57 | 55 | 63
  ALP, Grade 1 | 1 | 2 | 0
  ALP, Grade 2 | 0 | 0 | 0
  ALP, Grade 3 | 0 | 0 | 0
  ALP, Grade 4 | 0 | 0 | 0
  AST, Grade 0 | 54 | 56 | 63
  AST, Grade 1 | 2 | 1 | 0
  AST, Grade 2 | 2 | 0 | 0
  AST, Grade 3 | 0 | 0 | 0
  AST, Grade 4 | 0 | 0 | 0
  BIL, Grade 0 | 56 | 57 | 63
  BIL, Grade 1 | 1 | 0 | 0
  BIL, Grade 2 | 1 | 0 | 0
  BIL, Grade 3 | 0 | 0 | 0
  BIL, Grade 4 | 0 | 0 | 0
  CRE, Grade 0 | 55 | 54 | 62
  CRE, Grade 1 | 3 | 3 | 1
  CRE, Grade 2 | 0 | 0 | 0
  CRE, Grade 3 | 0 | 0 | 0
  CRE, Grade 4 | 0 | 0 | 0
  EOS, Grade 0 | 58 | 57 | 63
  EOS, Grade 1 | 0 | 0 | 0
  EOS, Grade 2 | 0 | 0 | 0
  EOS, Grade 3 | 0 | 0 | 0
  EOS, Grade 4 | 0 | 0 | 0
  EOS/100LEU, Grade 0 | 58 | 57 | 63
  EOS/100LEU, Grade 1 | 0 | 0 | 0
  EOS/100LEU, Grade 2 | 0 | 0 | 0
  EOS/100LEU, Grade 3 | 0 | 0 | 0
  EOS/100LEU, Grade 4 | 0 | 0 | 0
  BIC, Grade 0 | 49 | 43 | 51
  BIC, Grade 1 | 9 | 14 | 12
  BIC, Grade 2 | 0 | 0 | 0
  BIC, Grade 3 | 0 | 0 | 0
  BIC, Grade 4 | 0 | 0 | 0
  HGB, Grade 0 | 58 | 56 | 63
  HGB, Grade 1 | 0 | 1 | 0
  HGB, Grade 2 | 0 | 0 | 0
  HGB, Grade 3 | 0 | 0 | 0
  HGB, Grade 4 | 0 | 0 | 0
  PTS, Grade 0 | 58 | 57 | 61
  PTS, Grade 1 | 0 | 0 | 2
  PTS, Grade 2 | 0 | 0 | 0
  PTS, Grade 3 | 0 | 0 | 0
  PTS, Grade 4 | 0 | 0 | 0
  LYM, Grade 0 | 58 | 57 | 63
  LYM, Grade 1 | 0 | 0 | 0
  LYM, Grade 2 | 0 | 0 | 0
  LYM, Grade 3 | 0 | 0 | 0
  LYM, Grade 4 | 0 | 0 | 0
  LYM/100LEU, Grade 0 | 58 | 57 | 63
  LYM/100LEU, Grade 1 | 0 | 0 | 0
  LYM/100LEU, Grade 2 | 0 | 0 | 0
  LYM/100LEU, Grade 3 | 0 | 0 | 0
  LYM/100LEU, Grade 4 | 0 | 0 | 0
  SDI, Grade 0 | 55 | 56 | 58
  SDI, Grade 1 | 3 | 1 | 5
  SDI, Grade 2 | 0 | 0 | 0
  SDI, Grade 3 | 0 | 0 | 0
  SDI, Grade 4 | 0 | 0 | 0
  NEU, Grade 0 | 57 | 53 | 60
  NEU, Grade 1 | 0 | 4 | 3
  NEU, Grade 2 | 1 | 0 | 0
  NEU, Grade 3 | 0 | 0 | 0
  NEU, Grade 4 | 0 | 0 | 0
  NEU/100LEU, Grade 0 | 58 | 57 | 63
  NEU/100LEU, Grade 1 | 0 | 0 | 0
  NEU/100LEU, Grade 2 | 0 | 0 | 0
  NEU/100LEU, Grade 3 | 0 | 0 | 0
  NEU/100LEU, Grade 4 | 0 | 0 | 0
  PLC, Grade 0 | 58 | 56 | 62
  PLC, Grade 1 | 0 | 0 | 0
  PLC, Grade 2 | 0 | 1 | 1
  PLC, Grade 3 | 0 | 0 | 0
  PLC, Grade 4 | 0 | 0 | 0
  PTT, Grade 0 | 48 | 55 | 58
  PTT, Grade 1 | 8 | 2 | 5
  PTT, Grade 2 | 0 | 0 | 0
  PTT, Grade 3 | 2 | 0 | 0
  PTT, Grade 4 | 0 | 0 | 0
  WBC, Grade 0 | 58 | 57 | 63
  WBC, Grade 1 | 0 | 0 | 0
  WBC, Grade 2 | 0 | 0 | 0
  WBC, Grade 3 | 0 | 0 | 0
  WBC, Grade 4 | 0 | 0 | 0

24. Secondary Outcome: Geometric Mean Change in HIV-1 Viral Load (LV) From Baseline
Description: Changes from baseline in HIV-1 viral load (ratio of each value over baseline value) were obtained using crude values and expressed in RNA copies/mL. Baseline of HIV-1 viral load was defined as the geometric mean of values measured in blood samples taken at Screening and at Week 0. The HIV type 1, represents the more aggressive virus form, largely responsible for the AIDS pandemic. Changes from baseline were measured at Week 1 to 28 for the HIV Group, Weeks 30 and 38 for the 3D_HIV Group and 2D_HIV Group and from Week 1 to Week 38 for the Control Group.
Time Frame: At Weeks 1, 4, 6, 16, 28, 30 and 38
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: RNA copies/mL
Arm/Group | HIV Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 124 | 53 | 58 | 60
RNA copies/mL
  HIV-1 VL, Week 1: number analyzed (Participants) | 78 | 0 | 0 | 40
  HIV-1 VL, Week 1 | 1.0 (0.18) |  |  | 0.9 (0.18)
  HIV-1 VL, Week 4: number analyzed (Participants) | 124 | 0 | 0 | 58
  HIV-1 VL, Week 4 | 1.1 (0.28) |  |  | 1.1 (0.32)
  HIV-1 VL, Week 6: number analyzed (Participants) | 118 | 0 | 0 | 60
  HIV-1 VL, Week 6 | 1.1 (0.26) |  |  | 1.2 (0.37)
  HIV-1 VL, Week 16: number analyzed (Participants) | 121 | 0 | 0 | 56
  HIV-1 VL, Week 16 | 1.1 (0.31) |  |  | 1.1 (0.28)
  HIV-1 VL, Week 28: number analyzed (Participants) | 116 | 0 | 0 | 54
  HIV-1 VL, Week 28 | 1.2 (0.35) |  |  | 1.2 (0.36)
  HIV-1 VL, Week 30: number analyzed (Participants) | 0 | 53 | 58 | 54
  HIV-1 VL, Week 30 |  | 1.1 (0.24) | 1.2 (0.38) | 1.2 (0.34)
  HIV-1 VL, Week 38: number analyzed (Participants) | 0 | 49 | 57 | 52
  HIV-1 VL, Week 38 |  | 0.9 (0.28) | 1.2 (0.32) | 1.2 (0.43)

25. Secondary Outcome: Geometric Mean Change in HIV-1 VL From Baseline
Description: Changes from baseline in HIV-1 viral load (difference of each value minus baseline value) were obtained using log10-transformed values and expressed in log10-RNA copies/mL. Baseline of HIV-1 viral load was defined as geometric mean of values measured in blood samples taken at Screening and at Week 0. The HIV type 1, represents the more aggressive virus form, largely responsible for the AIDS pandemic. Changes from baseline were measured at Week 1 to 29 for the HIV Group, Weeks 30 and 38 for the 3D_HIV Group and 2D_HIV Group and from Week 1 to Week 38 for the Control Group.
Time Frame: At Weeks 1, 4, 6, 16, 28, 30 and 38
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: log10(RNA copies/mL)
Arm/Group | HIV Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 124 | 53 | 58 | 60
log10(RNA copies/mL)
  HIV-1 VL, Week 1: number analyzed (Participants) | 78 | 0 | 0 | 40
  HIV-1 VL, Week 1 | 0.0 (0.18) |  |  | -0.1 (0.18)
  HIV-1 VL, Week 4: number analyzed (Participants) | 124 | 0 | 0 | 58
  HIV-1 VL, Week 4 | 0.0 (0.28) |  |  | 0.1 (0.32)
  HIV-1 VL, Week 6: number analyzed (Participants) | 118 | 0 | 0 | 60
  HIV-1 VL, Week 6 | 0.1 (0.26) |  |  | 0.1 (0.37)
  HIV-1 VL, Week 16: number analyzed (Participants) | 121 | 0 | 0 | 56
  HIV-1 VL, Week 16 | 0.0 (0.31) |  |  | 0.0 (0.28)
  HIV-1 VL, Week 28: number analyzed (Participants) | 116 | 0 | 0 | 54
  HIV-1 VL, Week 28 | 0.1 (0.35) |  |  | 0.1 (0.36)
  HIV-1 VL, Week 30: number analyzed (Participants) | 0 | 53 | 58 | 54
  HIV-1 VL, Week 30 |  | 0.0 (0.24) | 0.1 (0.38) | 0.1 (0.34)
  HIV-1 VL, Week 38: number analyzed (Participants) | 0 | 49 | 57 | 52
  HIV-1 VL, Week 38 |  | 0.0 (0.28) | 0.1 (0.32) | 0.1 (0.43)

26. Secondary Outcome: Levels of HIV-1 Viral Load (VL)
Description: HIV-1 VL, using crude values, was expressed in RNA copies/mL and measured from Screening to Week 28 for the HIV Group, Weeks 30, 38 and 48 for the 3D_HIV Group and 2D_HIV Group and from Screening to Week 48 for the Control Group.
Time Frame: At Screening, Pre-vaccination and at Weeks 1, 4, 6, 16, 28, 30, 38 and 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: RNA Copies/mL
Arm/Group | HIV Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 125 | 53 | 58 | 60
RNA Copies/mL
  HIV-1 VL, Screening: number analyzed (Participants) | 125 | 0 | 0 | 60
  HIV-1 VL, Screening | 13797 [6823 to 28493] |  |  | 12882.5 [6441.5 to 27468.5]
  HIV-1 VL, Pre-vaccination: number analyzed (Participants) | 122 | 0 | 0 | 58
  HIV-1 VL, Pre-vaccination | 12982 [5800 to 29086] |  |  | 12688.5 [6882 to 26514]
  HIV-1 VL, Week 1: number analyzed (Participants) | 78 | 0 | 0 | 40
  HIV-1 VL, Week 1 | 14939 [5486 to 24432] |  |  | 11936 [6142 to 21405.5]
  HIV-1 VL, Week 4: number analyzed (Participants) | 124 | 0 | 0 | 58
  HIV-1 VL, Week 4 | 14242.5 [6151 to 32192.5] |  |  | 11627.5 [7010 to 25070]
  HIV-1 VL, Week 6: number analyzed (Participants) | 118 | 0 | 0 | 60
  HIV-1 VL, Week 6 | 17019 [6676 to 32848] |  |  | 15117.5 [6488.5 to 35630]
  HIV-1 VL, Week 16: number analyzed (Participants) | 121 | 0 | 0 | 56
  HIV-1 VL, Week 16 | 15045 [6040 to 28436] |  |  | 14605 [5698.5 to 33234]
  HIV-1 VL, Week 28: number analyzed (Participants) | 116 | 0 | 0 | 54
  HIV-1 VL, Week 28 | 12552.5 [6970.5 to 32604.5] |  |  | 13208 [5910 to 28274]
  HIV-1 VL, Week 30: number analyzed (Participants) | 0 | 53 | 58 | 54
  HIV-1 VL, Week 30 |  | 14703 [7365 to 25970] | 13902 [6977 to 29316] | 12855.5 [5996 to 32574]
  HIV-1 VL, Week 38: number analyzed (Participants) | 0 | 49 | 57 | 52
  HIV-1 VL, Week 38 |  | 12248 [6977 to 23435] | 14739 [8367 to 28182] | 12264.5 [5068 to 27001]
  HIV-1 VL, Week 48: number analyzed (Participants) | 0 | 46 | 55 | 50
  HIV-1 VL, Week 48 |  | 11004.5 [5910 to 25624] | 18415 [6741 to 38871] | 15266.5 [6000 to 39189]

27. Secondary Outcome: Levels of HIV-1 VL
Description: HIV-1 VL, using log10 transformed values, was expressed in log10-RNA copies/mL and measured from Screening to Week 28 for the HIV Group, Weeks 30, 38 and 48 for the 3D_HIV Group and 2D_HIV Group and from Screening to Week 48 for the Control Group.
Time Frame: At Screening, Pre-vaccination and at Weeks 1, 4, 6, 16, 28, 30, 38 and 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log10 (RNA Copies/mL)
Arm/Group | HIV Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 125 | 53 | 58 | 60
log10 (RNA Copies/mL)
  HIV-1 VL, Screening: number analyzed (Participants) | 125 | 0 | 0 | 60
  HIV-1 VL, Screening | 4.14 [3.834 to 4.455] |  |  | 4.11 [3.809 to 4.438]
  HIV-1 VL, Pre-vaccination: number analyzed (Participants) | 122 | 0 | 0 | 58
  HIV-1 VL, Pre-vaccination | 4.113 [3.763 to 4.464] |  |  | 4.103 [3.838 to 4.423]
  HIV-1 VL, Week 1: number analyzed (Participants) | 78 | 0 | 0 | 40
  HIV-1 VL, Week 1 | 4.174 [3.739 to 4.388] |  |  | 4.077 [3.788 to 4.331]
  HIV-1 VL, Week 4: number analyzed (Participants) | 124 | 0 | 0 | 58
  HIV-1 VL, Week 4 | 4.153 [3.789 to 4.508] |  |  | 4.065 [3.846 to 4.399]
  HIV-1 VL, Week 6: number analyzed (Participants) | 118 | 0 | 0 | 60
  HIV-1 VL, Week 6 | 4.231 [3.825 to 4.517] |  |  | 4.179 [3.811 to 4.551]
  HIV-1 VL, Week 16: number analyzed (Participants) | 121 | 0 | 0 | 56
  HIV-1 VL, Week 16 | 4.177 [3.781 to 4.454] |  |  | 4.163 [3.755 to 4.52]
  HIV-1 VL, Week 28: number analyzed (Participants) | 116 | 0 | 0 | 54
  HIV-1 VL, Week 28 | 4.099 [3.843 to 4.513] |  |  | 4.12 [3.772 to 4.451]
  HIV-1 VL, Week 30: number analyzed (Participants) | 0 | 53 | 58 | 54
  HIV-1 VL, Week 30 |  | 4.167 [3.867 to 4.414] | 4.143 [3.844 to 4.467] | 4.108 [3.778 to 4.513]
  HIV-1 VL, Week 38: number analyzed (Participants) | 0 | 49 | 57 | 52
  HIV-1 VL, Week 38 |  | 4.088 [3.844 to 4.37] | 4.168 [3.923 to 4.45] | 4.089 [3.705 to 4.429]
  HIV-1 VL, Week 48: number analyzed (Participants) | 0 | 46 | 55 | 50
  HIV-1 VL, Week 48 |  | 4.04 [3.772 to 4.409] | 4.265 [3.829 to 4.59] | 4.184 [3.778 to 4.593]

28. Secondary Outcome: Percentage of Subjects With Plasmatic HIV-1 Viral Load Decrease Higher Than (>) 1
Description: The proportion of subjects with >1 decrease of HIV-1 VL, was determined using log10-transformed values.
Time Frame: At Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 46 | 55 | 50
Percentage of participants | 0.00 | 0.00 | 0.00

29. Secondary Outcome: Cluster of Differentiation 4 (CD4) Absolute Cell Count
Description: Result determination, using crude values, was done from Screening to Week 28 for the HIV Group, Weeks 30, 38 and 48 for the 3D_HIV Group and 2D_HIV Group and from Screening (SCR) to Week (W) 48 for the Control Group.
Time Frame: At Screening, Pre-vaccination and at Weeks 1, 4, 6, 16, 28, 30, 38 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CD4 cells/cubic millimeter
Arm/Group | HIV Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 125 | 53 | 58 | 60
CD4 cells/cubic millimeter
  CD4, Screening: number analyzed (Participants) | 125 | 0 | 0 | 60
  CD4, Screening | 677.072 (164.31) |  |  | 688.2 (141.74)
  CD4, Pre-vaccination: number analyzed (Participants) | 122 | 0 | 0 | 59
  CD4, Pre-vaccination | 687.566 (184.41) |  |  | 712.407 (251.98)
  CD4, Week 1: number analyzed (Participants) | 78 | 0 | 0 | 42
  CD4, Week 1 | 723.91 (228.73) |  |  | 711.905 (226.84)
  CD4, Week 4: number analyzed (Participants) | 124 | 0 | 0 | 60
  CD4, Week 4 | 676.992 (182.96) |  |  | 688.717 (186.24)
  CD4, Week 6: number analyzed (Participants) | 121 | 0 | 0 | 60
  CD4, Week 6 | 691.174 (195.35) |  |  | 687.883 (202.79)
  CD4, Week 16: number analyzed (Participants) | 121 | 0 | 0 | 56
  CD4, Week 16 | 674.215 (213.69) |  |  | 674.75 (186.63)
  CD4, Week 28: number analyzed (Participants) | 116 | 0 | 0 | 54
  CD4, Week 28 | 630.836 (172.16) |  |  | 667.981 (183.53)
  CD4, Week 30: number analyzed (Participants) | 0 | 53 | 58 | 54
  CD4, Week 30 |  | 649.377 (193.66) | 654.448 (202.71) | 662.481 (181.76)
  CD4, Week 38: number analyzed (Participants) | 0 | 49 | 57 | 52
  CD4, Week 38 |  | 660.306 (202.04) | 635.561 (174.15) | 653.154 (176.71)
  CD4, Week 48: number analyzed (Participants) | 0 | 46 | 55 | 50
  CD4, Week 48 |  | 636.957 (175.72) | 650.418 (206.12) | 601.9 (186.81)

30. Secondary Outcome: Mean Change in CD4 Cell Count From Baseline
Description: Baseline for CD4 cell count analysis was defined as the mean of values measured in blood taken at Screening and at pre vaccination (PRE). Result determination, using crude values, was done from week 1 to 28 for the HIV Group, weeks 30, 38 and 48 for the 3D_HIV Group and 2D_HIV Group and from week 1 to week 48 for the Control Group.
Time Frame: At Weeks 1, 4, 6, 16, 28, 30, 38 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CD4 cells/cubic millimeter
Arm/Group | HIV Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 124 | 53 | 58 | 60
CD4 cells/cubic millimeter
  CD4, Week 1: number analyzed (Participants) | 78 | 0 | 0 | 42
  CD4, Week 1 | 4.633 (16.53) |  |  | 0.589 (17.98)
  CD4, Week 4: number analyzed (Participants) | 124 | 0 | 0 | 60
  CD4, Week 4 | -0.201 (17.97) |  |  | -1.212 (18.58)
  CD4, Week 6: number analyzed (Participants) | 121 | 0 | 0 | 60
  CD4, Week 6 | 2.066 (19.97) |  |  | -1.713 (19.68)
  CD4, Week 16: number analyzed (Participants) | 121 | 0 | 0 | 56
  CD4, Week 16 | -0.52 (20.82) |  |  | -2.568 (19.68)
  CD4, Week 28: number analyzed (Participants) | 116 | 0 | 0 | 54
  CD4, Week 28 | -5.782 (19.13) |  |  | -4.421 (16.06)
  CD4, Week 30: number analyzed (Participants) | 0 | 53 | 58 | 54
  CD4, Week 30 |  | -5.641 (19.17) | -2.417 (20.31) | -4.403 (19.88)
  CD4, Week 38: number analyzed (Participants) | 0 | 49 | 57 | 52
  CD4, Week 38 |  | -4.224 (22.97) | -4.626 (20.01) | -5.936 (16.85)
  CD4, Week 48: number analyzed (Participants) | 0 | 46 | 55 | 50
  CD4, Week 48 |  | -9.859 (18.66) | -3.915 (19.56) | -13.82 (18.67)

31. Secondary Outcome: Percentage of Subjects With ART (Anti-Retroviral Therapy) Initiation and HIV-related Clinical Events
Description: Only actual ART initiations were reported under the category "ART initiation". HIV-related clinical events were defined as: clinical disease progression, or confirmed VL > 100.000 copies/mL, or confirmed CD4 cell count < 350 cells/ cubic millimeter (mm3).
Time Frame: During the entire study period (up to Week 48)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
Number analyzed (Participants) | 61 | 64 | 60
Percentage of participants
  ART initiation | 8.2 | 6.3 | 8.3
  HIV related clinical events | 9.8 | 10.9 | 10.0

32. Secondary Outcome: Magnitude of Antigen Specific Cluster of Differentiation-40 Ligand (CD40L)+CD4+ T-cells Expressing at Least Interleukin-2 (IL-2)
Description: Magnitude was defined as the frequency of proteins 17, 24, Nef, reverse transcriptase (RT) - specific CD40L+CD4+ T-cells and F4co-Computed [frequency of CD4+ T-cells expressing markers in the response to the F4co fusion protein was estimated by adding individual frequencies of CD4+ T-cells to each of the 4 antigens (Nef, p17, p24, RT)] CD40L+CD4+ T-cells expressing at least interleukin- 2 (IL-2), as assessed by Intracellular Cytokine Staining (ICS).
Time Frame: During the entire study period - up to Week 48 (Pre-vaccination, Weeks 6, 28, 30 and 48 for the 3D_HIV Group, 2D_HIV Group and Control Group and at Pre-vaccination, Weeks 6 and 28 for the HIV Group)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom CMI assay or humoral results were available against at least one study vaccine antigen component after vaccination.
Measure: Median (Inter-Quartile Range); unit: CD40L+CD+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
CD40L+CD+ T-cells/million cells
  F4co-Computed, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  F4co-Computed, Pre-vaccination | 430.0 [288.0 to 714.0] | 469.0 [285.0 to 679.0] | 435.0 [285.0 to 690.0] | 364.0 [239.0 to 680.0]
  F4co-Computed, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  F4co-Computed, Week 6 | 2559.5 [1123.5 to 3879.5] | 1686.0 [823.5 to 2629.0] | 2014.5 [896.5 to 3456.5] | 557.5 [298.5 to 789.5]
  F4co-Computed, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  F4co-Computed, Week 28 | 818.0 [527.0 to 1333.0] | 677.5 [331.5 to 1179.5] | 751.0 [454.0 to 1329.0] | 345.0 [188.0 to 607.0]
  F4co-Computed, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  F4co-Computed, Week 30 | 2495.5 [1478.0 to 5418.0] | 681.0 [328.0 to 1387.0] |  | 521.0 [278.0 to 705.0]
  F4co-Computed, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  F4co-Computed, Week 48 | 937.0 [499.0 to 2490.0] | 534.5 [280.0 to 1243.5] |  | 365.0 [198.0 to 591.0]
  Nef, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  Nef, Pre-vaccination | 43.0 [28.0 to 81.0] | 42.0 [20.0 to 86.0] | 43.0 [21.0 to 86.0] | 46.0 [4.0 to 93.0]
  Nef, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  Nef, Week 6 | 521.0 [153.5 to 832.0] | 219.0 [126.0 to 524.0] | 259.0 [142.0 to 704.5] | 45.5 [11.0 to 80.0]
  Nef, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  Nef, Week 28 | 157.0 [60.0 to 361.0] | 97.5 [50.0 to 217.5] | 122.0 [54.0 to 243.0] | 29.0 [17.0 to 66.0]
  Nef, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  Nef, Week 30 | 672.0 [320.0 to 1340.0] | 104.0 [40.0 to 228.0] |  | 42.0 [5.0 to 90.0]
  Nef, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  Nef, Week 48 | 166.0 [76.0 to 620.5] | 96.0 [29.0 to 197.0] |  | 26.0 [4.0 to 86.0]
  p17, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p17, Pre-vaccination | 111.5 [44.0 to 152.0] | 92.0 [32.0 to 197.0] | 97.0 [38.0 to 168.0] | 105.0 [59.0 to 169.0]
  p17, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p17, Week 6 | 226.0 [101.0 to 576.0] | 226.0 [115.0 to 300.0] | 226.0 [114.0 to 345.0] | 130.5 [70.0 to 174.5]
  p17, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p17, Week 28 | 132.0 [62.0 to 243.0] | 109.5 [55.5 to 189.5] | 118.0 [60.0 to 202.0] | 68.0 [30.0 to 158.0]
  p17, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  p17, Week 30 | 173.5 [115.0 to 374.0] | 115.0 [56.0 to 222.0] |  | 106.5 [46.0 to 168.0]
  p17, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p17, Week 48 | 100.0 [71.0 to 222.0] | 120.0 [35.0 to 236.0] |  | 78.5 [30.0 to 140.5]
  p24, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p24, Pre-vaccination | 140.5 [74.0 to 266.0] | 121.0 [59.0 to 212.0] | 127.0 [60.0 to 213.0] | 129.0 [80.0 to 250.0]
  p24, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p24, Week 6 | 271.0 [124.0 to 450.0] | 222.0 [128.5 to 411.0] | 253.0 [128.0 to 449.0] | 127.0 [90.5 to 306.0]
  p24, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p24, Week 28 | 184.0 [71.0 to 374.0] | 159.0 [55.5 to 284.5] | 178.0 [60.0 to 291.0] | 120.0 [34.0 to 238.0]
  p24, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  p24, Week 30 | 256.0 [119.0 to 542.0] | 183.5 [94.5 to 286.5] |  | 155.0 [45.0 to 205.0]
  p24, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p24, Week 48 | 197.0 [122.0 to 355.0] | 129.0 [65.0 to 301.0] |  | 119.5 [67.5 to 229.0]
  RT, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  RT, Pre-vaccination | 158.0 [73.0 to 239.0] | 126.0 [85.0 to 185.0] | 132.0 [81.0 to 210.0] | 116.0 [29.0 to 223.0]
  RT, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  RT, Week 6 | 1160.0 [560.0 to 2161.5] | 837.0 [364.5 to 1689.5] | 1070.5 [461.5 to 1890.0] | 174.0 [82.0 to 322.0]
  RT, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  RT, Week 28 | 297.0 [205.0 to 501.0] | 279.5 [130.5 to 540.5] | 297.0 [185.0 to 534.0] | 101.0 [58.0 to 153.0]
  RT, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  RT, Week 30 | 1155.0 [682.0 to 2958.0] | 245.5 [114.0 to 465.0] |  | 180.5 [92.0 to 270.0]
  RT, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  RT, Week 48 | 365.5 [122.0 to 781.5] | 170.0 [91.0 to 469.0] |  | 120.0 [37.0 to 187.0]

33. Secondary Outcome: Magnitude of Antigen Specific CD40L+CD4+ T-cells Expressing at Least One Cytokine
Description: Magnitude was defined as the frequency of proteins 17, 24, Nef, reverse transcriptase (RT) - specific CD40L+CD4+ T-cells and F4co-Computed [frequency of CD4+ T-cells expressing markers in the response to the F4co fusion protein was estimated by adding individual frequencies of CD4+ T-cells to each of the 4 antigens (Nef, p17, p24, RT)] CD40L+CD4+ T-cells expressing at least interleukin- 2 (IL-2) or another cytokine among interferon-gamma (IFN-γ) and/or tumour necrosis-alpha (TNF-α), as assessed by Intracellular Cytokine Staining (ICS).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: CD40L+CD4+ T-cells/million T-cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
CD40L+CD4+ T-cells/million T-cells
  F4co-Computed, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  F4co-Computed, Pre-vaccination | 1135.5 [745.0 to 1666.0] | 997.0 [625.0 to 1631.0] | 1022.0 [686.0 to 1665.0] | 953.0 [550.0 to 1942.0]
  F4co-Computed, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  F4co-Computed, Week 6 | 3675.0 [2101.0 to 5981.0] | 2506.5 [1502.0 to 4102.5] | 2864.0 [1590.5 to 5248.0] | 1243.0 [689.5 to 1815.0]
  F4co-Computed, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  F4co-Computed, Week 28 | 1587.0 [977.0 to 2345.0] | 1253.0 [810.0 to 2402.5] | 1433.0 [876.0 to 2394.0] | 786.0 [612.0 to 1928.0]
  F4co-Computed, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  F4co-Computed, Week 30 | 4039.0 [2055.0 to 7632.0] | 1108.0 [744.0 to 2718.0] |  | 1157.0 [769.0 to 1792.0]
  F4co-Computed, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  F4co-Computed, Week 48 | 1947.0 [847.0 to 2914.0] | 1039.5 [663.5 to 2032.5] |  | 1251.0 [529.0 to 1637.0]
  Nef, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  Nef, Pre-vaccination | 87.0 [55.0 to 219.0] | 87.0 [57.0 to 176.0] | 87.0 [55.0 to 219.0] | 108.0 [52.0 to 172.0]
  Nef, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  Nef, Week 6 | 599.0 [323.0 to 1289.5] | 392.0 [232.0 to 692.5] | 434.0 [244.0 to 821.0] | 115.0 [39.5 to 188.5]
  Nef, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  Nef, Week 28 | 227.0 [134.0 to 480.0] | 179.5 [93.5 to 308.5] | 208.0 [96.0 to 382.0] | 73.0 [33.0 to 149.0]
  Nef, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  Nef, Week 30 | 763.0 [562.0 to 1705.0] | 204.0 [70.0 to 344.0] |  | 113.0 [42.0 to 230.0]
  Nef, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  Nef, Week 48 | 258.5 [136.5 to 717.5] | 146.0 [78.0 to 394.0] |  | 87.0 [45.0 to 213.5]
  p17, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p17, Pre-vaccination | 249.5 [146.0 to 397.0] | 164.0 [106.0 to 406.0] | 228.0 [127.0 to 406.0] | 263.0 [109.0 to 468.0]
  p17, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p17, Week 6 | 517.0 [244.0 to 835.0] | 379.5 [187.0 to 600.5] | 393.0 [221.0 to 791.0] | 267.0 [199.5 to 475.0]
  p17, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p17, Week 28 | 284.0 [171.0 to 415.0] | 243.5 [101.0 to 493.0] | 281.0 [138.0 to 426.0] | 228.0 [116.0 to 406.0]
  p17, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  p17, Week 30 | 413.0 [252.0 to 654.0] | 242.0 [158.5 to 540.0] |  | 303.0 [142.0 to 444.0]
  p17, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p17, Week 48 | 261.0 [124.0 to 455.0] | 244.0 [97.0 to 484.0] |  | 245.5 [146.0 to 426.0]
  p24, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p24, Pre-vaccination | 459.0 [286.0 to 669.0] | 339.0 [242.0 to 532.0] | 379.0 [250.0 to 591.0] | 379.0 [191.0 to 718.0]
  p24, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p24, Week 6 | 596.0 [333.0 to 985.0] | 452.0 [330.0 to 1016.5] | 486.0 [333.0 to 989.0] | 505.5 [235.0 to 766.5]
  p24, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p24, Week 28 | 439.0 [263.0 to 806.0] | 381.5 [173.0 to 735.0] | 408.0 [205.0 to 748.0] | 277.0 [201.0 to 918.0]
  p24, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  p24, Week 30 | 596.0 [413.0 to 941.0] | 424.5 [233.5 to 915.5] |  | 401.5 [255.0 to 688.0]
  p24, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p24, Week 48 | 486.0 [303.0 to 892.0] | 371.0 [220.0 to 638.0] |  | 404.5 [211.0 to 662.5]
  RT, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  RT, Pre-vaccination | 268.5 [158.0 to 412.0] | 238.0 [140.0 to 335.0] | 247.0 [158.0 to 387.0] | 204.0 [110.0 to 436.0]
  RT, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  RT, Week 6 | 1588.5 [839.0 to 2806.0] | 1074.0 [622.5 to 2123.0] | 1346.0 [739.0 to 2427.5] | 296.0 [137.0 to 428.0]
  RT, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  RT, Week 28 | 378.0 [299.0 to 709.0] | 379.0 [204.5 to 687.0] | 378.0 [232.0 to 709.0] | 204.0 [136.0 to 328.0]
  RT, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  RT, Week 30 | 1629.0 [784.0 to 3596.0] | 327.5 [150.0 to 753.5] |  | 256.0 [153.0 to 471.0]
  RT, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  RT, Week 48 | 451.5 [228.0 to 911.5] | 299.0 [155.0 to 615.0] |  | 222.0 [127.0 to 436.0]

34. Secondary Outcome: Magnitude of Antigen Specific CD40L-CD4+ T-cells Expressing at Least One Cytokine.
Description: Magnitude was defined as the frequency of proteins 17, 24, Nef, reverse transcriptase (RT) - specific CD40L-CD4+ T-cells and F4co-Computed [frequency of CD4+ T-cells expressing markers in the response to the F4co fusion protein was estimated by adding individual frequencies of CD4+ T-cells to each of the 4 antigens (Nef, p17, p24, RT)] CD40L-CD4+ T-cells expressing at least interleukin- 2 (IL-2) or another cytokine among interferon-gamma (IFN-γ) and/or tumour necrosis-alpha (TNF-α), as assessed by Intracellular Cytokine Staining (ICS).
Time Frame: as for outcome 32
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects for whom CMI assay or humoral results were available against at least one study vaccine antigen component after vaccination.
Measure: Median (Inter-Quartile Range); unit: CD40L-CD4+ T-cells/million T-cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
CD40L-CD4+ T-cells/million T-cells
  F4co-Computed, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  F4co-Computed, Pre-vaccination | 874.0 [609.0 to 1535.0] | 973.0 [723.0 to 1480.0] | 945.0 [677.0 to 1518.0] | 1433.0 [766.0 to 2554.0]
  F4co-Computed, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  F4co-Computed, Week 6 | 1189.0 [707.5 to 2215.0] | 1086.5 [839.0 to 2067.5] | 1090.0 [815.0 to 2102.0] | 1227.0 [803.0 to 2323.0]
  F4co-Computed, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  F4co-Computed, Week 28 | 892.0 [605.0 to 1528.0] | 1115.5 [645.5 to 1626.5] | 986.0 [644.0 to 1577.0] | 1118.0 [659.0 to 2782.0]
  F4co-Computed, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  F4co-Computed, Week 30 | 1376.0 [1033.0 to 2230.0] | 1198.0 [650.0 to 2233.0] |  | 1416.0 [749.0 to 2035.0]
  F4co-Computed, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  F4co-Computed, Week 48 | 1193.0 [655.0 to 1592.0] | 1006.5 [628.0 to 1781.5] |  | 1419.0 [717.0 to 2659.0]
  Nef, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  Nef, Pre-vaccination | 148.0 [89.0 to 357.0] | 239.0 [115.0 to 400.0] | 195.0 [100.0 to 400.0] | 263.0 [109.0 to 453.0]
  Nef, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  Nef, Week 6 | 302.0 [122.0 to 376.5] | 301.5 [151.0 to 882.5] | 301.5 [133.5 to 495.5] | 211.5 [78.0 to 342.5]
  Nef, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  Nef, Week 28 | 169.0 [70.0 to 542.0] | 261.5 [109.0 to 409.0] | 241.0 [86.0 to 430.0] | 197.0 [102.0 to 322.0]
  Nef, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  Nef, Week 30 | 245.0 [191.0 to 467.0] | 273.0 [152.0 to 529.0] |  | 250.0 [103.0 to 495.0]
  Nef, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  Nef, Week 48 | 215.0 [111.0 to 393.5] | 174.0 [79.0 to 381.0] |  | 267.5 [100.5 to 576.0]
  p17, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p17, Pre-vaccination | 204.5 [110.0 to 316.0] | 184.0 [108.0 to 337.0] | 188.0 [108.0 to 334.0] | 230.0 [101.0 to 552.0]
  p17, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p17, Week 6 | 229.0 [103.0 to 382.0] | 231.5 [100.0 to 333.5] | 230.0 [103.0 to 365.0] | 293.5 [126.5 to 444.5]
  p17, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p17, Week 28 | 164.0 [103.0 to 334.0] | 238.0 [112.5 to 395.5] | 210.0 [106.0 to 361.0] | 203.0 [101.0 to 405.0]
  p17, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  p17, Week 30 | 279.5 [188.0 to 378.0] | 166.0 [101.0 to 336.5] |  | 229.0 [71.0 to 513.0]
  p17, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p17, Week 48 | 210.0 [82.0 to 292.0] | 177.0 [104.0 to 403.0] |  | 224.5 [108.0 to 461.0]
  p24, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p24, Pre-vaccination | 297.5 [189.0 to 568.0] | 287.0 [169.0 to 593.0] | 294.0 [174.0 to 593.0] | 377.0 [200.0 to 819.0]
  p24, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p24, Week 6 | 287.0 [177.0 to 481.0] | 344.5 [173.5 to 594.0] | 288.0 [175.0 to 587.0] | 428.5 [272.5 to 900.0]
  p24, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p24, Week 28 | 296.0 [141.0 to 521.0] | 340.0 [108.5 to 512.0] | 313.0 [116.0 to 521.0] | 487.0 [236.0 to 836.0]
  p24, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  p24, Week 30 | 389.0 [220.0 to 749.0] | 298.0 [163.0 to 674.0] |  | 492.5 [237.0 to 862.0]
  p24, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p24, Week 48 | 341.0 [150.0 to 580.0] | 369.0 [228.0 to 695.0] |  | 396.5 [218.5 to 1082.0]
  RT, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  RT, Pre-vaccination | 175.5 [101.0 to 292.0] | 194.0 [63.0 to 339.0] | 194.0 [73.0 to 310.0] | 235.0 [84.0 to 432.0]
  RT, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  RT, Week 6 | 369.0 [159.0 to 666.5] | 258.5 [142.0 to 513.0] | 304.0 [148.5 to 637.5] | 144.0 [78.0 to 298.0]
  RT, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  RT, Week 28 | 210.0 [85.0 to 455.0] | 118.0 [64.0 to 316.0] | 148.0 [75.0 to 322.0] | 138.0 [88.0 to 340.0]
  RT, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  RT, Week 30 | 369.0 [185.0 to 631.0] | 162.0 [96.5 to 384.0] |  | 162.0 [74.0 to 338.0]
  RT, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  RT, Week 48 | 270.5 [119.0 to 493.0] | 132.5 [77.0 to 428.0] |  | 158.0 [99.0 to 300.0]

35. Secondary Outcome: Magnitude of Antigen Specific CD4+ T-cells Expressing at Least One Cytokine
Description: Magnitude was defined as the frequency of proteins 17, 24, Nef, reverse transcriptase (RT) - specific CD4+ T-cells and F4co-Computed [frequency of CD4+ T-cells expressing markers in the response to the F4co fusion protein was estimated by adding individual frequencies of CD4+ T-cells to each of the 4 antigens (Nef, p17, p24, RT)] CD4+ T-cells expressing at least interleukin- 2 (IL-2) or another cytokine among interferon-gamma (IFN-γ) and/or tumour necrosis-alpha (TNF-α), as assessed by Intracellular Cytokine Staining (ICS).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
CD4+ T-cells/million cells
  F4co-Computed, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  F4co-Computed, Pre-vaccination | 2360.5 [1515.0 to 3354.0] | 1998.0 [1549.0 to 3083.0] | 2068.0 [1515.0 to 3354.0] | 2420.0 [1334.0 to 3993.0]
  F4co-Computed, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  F4co-Computed, Week 6 | 5024.5 [3128.0 to 7808.5] | 4146.5 [2389.0 to 7608.0] | 4432.0 [2623.5 to 7663.5] | 2711.5 [1518.0 to 3755.0]
  F4co-Computed, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  F4co-Computed, Week 28 | 2885.0 [1932.0 to 3632.0] | 2374.0 [1710.0 to 3617.5] | 2459.0 [1806.0 to 3632.0] | 2052.0 [1413.0 to 5226.0]
  F4co-Computed, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  F4co-Computed, Week 30 | 5376.5 [4123.0 to 9609.0] | 2538.0 [1587.0 to 4652.0] |  | 2593.0 [1415.0 to 3718.0]
  F4co-Computed, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  F4co-Computed, Week 48 | 3266.0 [1851.0 to 4297.0] | 2544.5 [1301.0 to 3816.0] |  | 2398.0 [1866.0 to 3805.0]
  Nef, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  Nef, Pre-vaccination | 284.5 [175.0 to 524.0] | 390.0 [186.0 to 706.0] | 337.0 [175.0 to 594.0] | 386.0 [218.0 to 545.0]
  Nef, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  Nef, Week 6 | 983.5 [502.5 to 1533.5] | 805.0 [553.0 to 1474.5] | 813.0 [508.5 to 1474.5] | 323.5 [171.5 to 644.0]
  Nef, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  Nef, Week 28 | 494.0 [288.0 to 1002.0] | 444.0 [308.0 to 786.0] | 455.0 [288.0 to 942.0] | 283.0 [162.0 to 434.0]
  Nef, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  Nef, Week 30 | 1220.0 [824.0 to 2059.0] | 512.0 [263.0 to 1132.0] |  | 357.0 [177.0 to 673.0]
  Nef, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  Nef, Week 48 | 568.0 [320.0 to 888.0] | 356.0 [233.0 to 721.0] |  | 377.5 [173.0 to 772.5]
  p17, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p17, Pre-vaccination | 463.0 [305.0 to 733.0] | 434.0 [256.0 to 980.0] | 457.0 [256.0 to 809.0] | 578.0 [316.0 to 815.0]
  p17, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p17, Week 6 | 797.0 [434.0 to 1198.0] | 561.5 [356.0 to 1252.0] | 682.0 [386.0 to 1198.0] | 562.0 [370.0 to 949.0]
  p17, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p17, Week 28 | 494.0 [364.0 to 687.0] | 527.5 [330.5 to 866.0] | 494.0 [344.0 to 819.0] | 433.0 [281.0 to 823.0]
  p17, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  p17, Week 30 | 798.0 [519.0 to 1041.0] | 473.0 [308.5 to 930.0] |  | 536.0 [324.0 to 925.0]
  p17, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p17, Week 48 | 525.0 [293.0 to 749.0] | 580.0 [230.0 to 962.0] |  | 498.5 [264.5 to 812.5]
  p24, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p24, Pre-vaccination | 794.5 [533.0 to 1280.0] | 699.0 [400.0 to 1112.0] | 759.0 [471.0 to 1237.0] | 733.0 [526.0 to 1658.0]
  p24, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p24, Week 6 | 902.0 [608.0 to 1291.0] | 1033.0 [529.0 to 1847.0] | 977.0 [533.0 to 1363.0] | 943.0 [605.5 to 1772.5]
  p24, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p24, Week 28 | 784.0 [459.0 to 1223.0] | 670.5 [499.0 to 1158.5] | 726.0 [461.0 to 1201.0] | 883.0 [502.0 to 1885.0]
  p24, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  p24, Week 30 | 988.0 [682.0 to 1504.0] | 708.0 [470.0 to 1535.0] |  | 944.5 [606.0 to 1383.0]
  p24, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p24, Week 48 | 856.0 [590.0 to 1194.0] | 831.0 [471.0 to 1393.0] |  | 891.0 [547.5 to 1562.0]
  RT, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  RT, Pre-vaccination | 494.5 [293.0 to 757.0] | 442.0 [298.0 to 677.0] | 455.0 [293.0 to 757.0] | 474.0 [308.0 to 734.0]
  RT, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  RT, Week 6 | 1916.5 [1208.5 to 3465.0] | 1426.5 [839.0 to 2496.5] | 1680.0 [1011.5 to 2837.5] | 416.0 [284.0 to 653.0]
  RT, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  RT, Week 28 | 599.0 [450.0 to 1206.0] | 667.5 [347.0 to 1015.5] | 634.0 [403.0 to 1081.0] | 384.0 [269.0 to 686.0]
  RT, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  RT, Week 30 | 2138.0 [1186.0 to 3878.0] | 540.0 [330.5 to 1299.0] |  | 477.0 [339.0 to 720.0]
  RT, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  RT, Week 48 | 797.5 [433.5 to 1666.0] | 573.0 [373.0 to 791.0] |  | 470.0 [274.0 to 838.0]

36. Secondary Outcome: Magnitude of Antigen Specific CD8+ T-cells Expressing at Least One Cytokine
Description: Magnitude was defined as the frequency of proteins 17, 24, Nef, reverse transcriptase (RT) - specific CD8+ T-cells and F4co-Computed [frequency of CD8+ T-cells expressing markers in the response to the F4co fusion protein was estimated by adding individual frequencies of CD8+ T-cells to each of the 4 antigens (Nef, p17, p24, RT)] CD8+ T-cells expressing at least interleukin- 2 (IL-2) or another cytokine among interferon-gamma (IFN-γ) and/or tumour necrosis-alpha (TNF-α), as assessed by Intracellular Cytokine Staining (ICS).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
CD8+ T-cells/million cells
  F4co-Computed, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  F4co-Computed, Pre-vaccination | 15895.5 [10567.0 to 28650.0] | 19633.0 [13938.0 to 37746.0] | 17609.0 [11299.0 to 30838.0] | 25819.0 [13977.0 to 41349.0]
  F4co-Computed, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  F4co-Computed, Week 6 | 16727.0 [9665.5 to 23222.5] | 19340.0 [13082.0 to 37413.5] | 17839.5 [12295.0 to 25795.5] | 29786.5 [17947.0 to 46398.0]
  F4co-Computed, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  F4co-Computed, Week 28 | 17526.0 [11559.0 to 29760.0] | 17186.5 [11078.5 to 33554.0] | 17344.0 [11179.0 to 30317.0] | 25798.0 [17168.0 to 36067.0]
  F4co-Computed, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  F4co-Computed, Week 30 | 15659.5 [9940.0 to 23406.0] | 19210.0 [12487.0 to 33548.0] |  | 29064.0 [16232.0 to 37335.0]
  F4co-Computed, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  F4co-Computed, Week 48 | 16143.0 [8304.0 to 26733.0] | 21063.0 [10921.0 to 33207.0] |  | 25564.0 [14771.0 to 35420.0]
  Nef, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  Nef, Pre-vaccination | 3187.0 [1413.0 to 6646.0] | 2453.0 [1447.0 to 8829.0] | 3174.0 [1413.0 to 7329.0] | 3796.0 [1772.0 to 10330.0]
  Nef, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  Nef, Week 6 | 3141.0 [1060.0 to 6597.5] | 3497.5 [1341.5 to 8698.5] | 3141.0 [1178.5 to 6856.0] | 5174.0 [2343.5 to 9489.5]
  Nef, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  Nef, Week 28 | 2641.0 [1087.0 to 6218.0] | 3655.0 [1110.5 to 8598.5] | 3054.0 [1087.0 to 7235.0] | 4332.0 [2158.0 to 8647.0]
  Nef, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  Nef, Week 30 | 2790.0 [1156.0 to 4828.0] | 3387.0 [1497.0 to 8670.0] |  | 3970.5 [2122.0 to 9214.0]
  Nef, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  Nef, Week 48 | 2444.5 [1032.5 to 5241.5] | 2478.0 [1521.0 to 7197.0] |  | 4014.5 [2288.5 to 7700.0]
  p17, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p17, Pre-vaccination | 858.0 [185.0 to 1995.0] | 1212.0 [385.0 to 2891.0] | 991.0 [275.0 to 2670.0] | 2246.0 [648.0 to 7255.0]
  p17, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p17, Week 6 | 829.0 [231.0 to 2702.0] | 1478.5 [275.5 to 3688.5] | 1085.0 [260.0 to 3435.0] | 1681.5 [621.0 to 6251.5]
  p17, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p17, Week 28 | 707.0 [217.0 to 2386.0] | 1419.0 [334.5 to 3422.5] | 1055.0 [271.0 to 2756.0] | 1613.0 [566.0 to 3702.0]
  p17, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  p17, Week 30 | 510.0 [142.0 to 2861.0] | 1467.0 [378.0 to 3265.0] |  | 1524.0 [447.0 to 4659.0]
  p17, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p17, Week 48 | 818.0 [217.0 to 1890.0] | 1669.0 [301.0 to 3477.0] |  | 1494.0 [623.0 to 5155.0]
  p24, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  p24, Pre-vaccination | 5364.0 [2266.0 to 8040.0] | 8630.0 [1356.0 to 12207.0] | 6248.0 [1787.0 to 11204.0] | 8435.0 [2567.0 to 20399.0]
  p24, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  p24, Week 6 | 4972.0 [2291.0 to 8391.0] | 6826.0 [1924.0 to 14308.5] | 5610.0 [2221.0 to 10269.0] | 10328.0 [2723.5 to 23641.5]
  p24, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  p24, Week 28 | 6273.0 [2195.0 to 8487.0] | 5465.5 [1629.0 to 12415.5] | 6181.0 [1654.0 to 11338.0] | 8207.0 [2303.0 to 19305.0]
  p24, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  p24, Week 30 | 5525.0 [1903.0 to 8346.0] | 5064.0 [1472.0 to 13693.0] |  | 8923.5 [3217.0 to 21785.0]
  p24, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  p24, Week 48 | 5900.0 [2042.0 to 8511.0] | 6371.0 [2135.0 to 12114.0] |  | 7410.0 [2127.5 to 18982.5]
  RT, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  RT, Pre-vaccination | 3724.5 [1740.0 to 7216.0] | 3073.0 [1953.0 to 7529.0] | 3556.0 [1826.0 to 7529.0] | 4395.0 [2124.0 to 7654.0]
  RT, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  RT, Week 6 | 3699.5 [1575.0 to 8150.5] | 3418.0 [2058.5 to 7416.0] | 3490.0 [1856.0 to 7732.0] | 4715.0 [2605.0 to 9441.0]
  RT, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  RT, Week 28 | 6187.0 [1597.0 to 9131.0] | 2860.5 [1817.5 to 7713.0] | 3663.0 [1778.0 to 8986.0] | 4292.0 [1921.0 to 7171.0]
  RT, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  RT, Week 30 | 3262.0 [1577.0 to 8040.0] | 3747.5 [2134.5 to 7150.5] |  | 4538.0 [2198.0 to 8225.0]
  RT, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  RT, Week 48 | 3299.5 [1737.5 to 7638.0] | 3462.5 [1950.0 to 8127.0] |  | 4565.0 [2477.0 to 7347.0]

37. Secondary Outcome: Number of Subjects With Response to at Least 1, 2, 3 or 4 Antigens
Description: Breadth was assessed only for the CD4+ T-cells and was measured by evaluating response to at least 1, 2, 3 or all 4 antigens: proteins 17, 24, Nef, reverse transcriptase (RT).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
Participants
  1 antigen, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  1 antigen, Pre-vaccination | 30 | 25 | 55 | 25
  2 antigens, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  2 antigens, Pre-vaccination | 19 | 16 | 35 | 18
  3 antigens, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  3 antigens, Pre-vaccination | 11 | 8 | 19 | 8
  4 antigens, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  4 antigens, Pre-vaccination | 4 | 3 | 7 | 3
  1 antigen, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  1 antigen, Week 6 | 28 | 32 | 60 | 9
  2 antigens, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  2 antigens, Week 6 | 24 | 24 | 48 | 2
  3 antigens, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  3 antigens, Week 6 | 12 | 12 | 24 | 1
  4 antigens, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  4 antigens, Week 6 | 6 | 6 | 12 | 0
  1 antigen, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  1 antigen, Week 28 | 19 | 22 | 41 | 7
  2 antigens, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  2 antigens, Week 28 | 13 | 11 | 24 | 4
  3 antigens, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  3 antigens, Week 28 | 4 | 4 | 8 | 2
  4 antigens, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  4 antigens, Week 28 | 2 | 3 | 5 | 1
  1 antigen, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  1 antigen, Week 30 | 30 | 20 |  | 14
  2 antigens, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  2 antigens, Week 30 | 24 | 11 |  | 5
  3 antigens, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  3 antigens, Week 30 | 15 | 6 |  | 3
  4 antigens, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  4 antigens, Week 30 | 8 | 2 |  | 0
  1 antigen, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  1 antigen, Week 48 | 23 | 19 |  | 13
  2 antigens, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  2 antigens, Week 48 | 17 | 7 |  | 3
  3 antigens, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  3 antigens, Week 48 | 5 | 4 |  | 2
  4 antigens, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  4 antigens, Week 48 | 4 | 1 |  | 0

38. Secondary Outcome: Cytokine Expression Profile of F4co-Computed CD4+ T Cells
Description: The cytokine co-expression profile was defined by the frequency of F4co-Computed CD4+ T-cells [frequency of CD4+ T-cells expressing markers in the response to the F4co fusion protein was estimated by adding individual frequencies of CD4+ T-cells to each of the 4 antigens (Nef, p17, p24, RT)] expressing CD40L and/or IL-2 and/or tumour necrosis factor-alpha (TNF-α) and/or interferon-gamma (IFN-γ).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: F4co-computed CD4+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 41 | 42 | 79 | 37
F4co-computed CD4+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L, Pre-vaccination | 772.0 [183.0 to 1601.0] | 299.5 [73.0 to 1332.0] | 453.0 [130.0 to 1451.0] | 493.0 [33.0 to 1376.5]
  CD40L, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  CD40L, Week 6 | 355.0 [4.0 to 1290.0] | 472.0 [172.0 to 1091.0] | 427.0 [33.0 to 1100.5] | 153.0 [4.0 to 931.0]
  CD40L, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L, Week 28 | 560.5 [133.0 to 1163.0] | 453.0 [4.0 to 938.0] | 506.5 [4.0 to 988.0] | 442.0 [4.0 to 848.0]
  CD40L, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  CD40L, Week 30 | 452.0 [4.0 to 1211.0] | 760.5 [4.0 to 1575.0] |  | 716.5 [103.0 to 1666.0]
  CD40L, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L, Week 48 | 383.0 [4.0 to 831.0] | 481.5 [28.0 to 1966.0] |  | 653.0 [143.0 to 1520.0]
  IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  IL-2, Pre-vaccination | 118.0 [18.0 to 237.0] | 45.5 [4.0 to 108.0] | 70.0 [10.0 to 193.0] | 93.5 [29.5 to 149.0]
  IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  IL-2, Week 6 | 127.0 [25.0 to 222.0] | 72.0 [31.0 to 171.0] | 91.5 [25.0 to 206.5] | 58.0 [20.0 to 126.0]
  IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IL-2, Week 28 | 63.0 [4.0 to 126.0] | 59.0 [8.0 to 245.0] | 63.0 [6.5 to 206.5] | 34.0 [4.0 to 115.0]
  IL-2, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  IL-2, Week 30 | 103.0 [25.0 to 273.0] | 92.5 [9.0 to 155.0] |  | 46.5 [4.0 to 137.5]
  IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  IL-2, Week 48 | 74.0 [5.0 to 165.0] | 58.0 [18.0 to 114.0] |  | 86.0 [6.0 to 139.0]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  TNF-α, Pre-vaccination | 250.0 [103.0 to 528.0] | 251.5 [46.0 to 610.0] | 250.0 [67.0 to 610.0] | 178.5 [82.0 to 639.0]
  TNF-α, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  TNF-α, Week 6 | 346.0 [112.0 to 664.0] | 251.0 [130.0 to 528.0] | 277.5 [129.0 to 644.5] | 166.5 [21.0 to 477.0]
  TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α, Week 28 | 242.0 [79.0 to 423.0] | 135.5 [4.0 to 272.0] | 163.0 [6.5 to 329.5] | 216.0 [83.0 to 392.0]
  TNF-α, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  TNF-α, Week 30 | 389.0 [113.0 to 749.0] | 101.5 [4.0 to 422.5] |  | 223.0 [43.5 to 686.5]
  TNF-α, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  TNF-α, Week 48 | 341.0 [70.0 to 901.0] | 192.5 [20.0 to 317.0] |  | 182.0 [25.0 to 668.0]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  IFN- γ, Pre-vaccination | 352.0 [192.0 to 640.0] | 396.5 [193.0 to 779.0] | 383.0 [192.0 to 654.0] | 446.0 [262.5 to 850.0]
  IFN- γ, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  IFN- γ, Week 6 | 411.0 [242.0 to 808.0] | 448.0 [193.0 to 696.0] | 426.0 [212.0 to 697.5] | 563.5 [301.0 to 999.0]
  IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ, Week 28 | 289.5 [167.0 to 419.0] | 454.0 [218.0 to 642.0] | 377.5 [197.0 to 557.0] | 536.0 [275.0 to 995.0]
  IFN- γ, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  IFN- γ, Week 30 | 439.0 [226.0 to 720.0] | 432.5 [235.0 to 935.0] |  | 479.0 [310.5 to 892.0]
  IFN- γ, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  IFN- γ, Week 48 | 329.0 [158.0 to 553.0] | 418.5 [179.0 to 772.5] |  | 487.0 [325.0 to 1223.0]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_IL-2, Pre-vaccination | 149.0 [105.0 to 227.0] | 149.5 [48.0 to 244.0] | 149.0 [67.0 to 244.0] | 77.5 [20.5 to 138.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  CD40L_IL-2, Week 6 | 499.0 [189.0 to 1192.0] | 320.0 [198.0 to 616.0] | 430.5 [193.5 to 890.0] | 127.5 [8.0 to 208.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IL-2, Week 28 | 199.0 [120.0 to 473.0] | 196.0 [91.0 to 325.0] | 198.0 [108.0 to 360.5] | 56.0 [27.0 to 97.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  CD40L_IL-2, Week 30 | 377.0 [175.0 to 865.0] | 142.5 [108.5 to 299.0] |  | 96.0 [46.0 to 180.5]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_IL-2, Week 48 | 172.0 [52.0 to 335.0] | 218.0 [68.0 to 342.0] |  | 102.0 [17.0 to 166.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_TNF-α, Pre-vaccination | 201.0 [90.0 to 270.0] | 116.0 [10.0 to 290.0] | 154.0 [63.0 to 283.0] | 88.5 [41.0 to 254.5]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  CD40L_TNF-α, Week 6 | 416.0 [212.0 to 683.0] | 275.0 [132.0 to 456.0] | 374.5 [165.5 to 481.5] | 110.0 [63.0 to 256.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α, Week 28 | 152.5 [95.0 to 276.0] | 101.0 [57.0 to 236.0] | 129.5 [70.0 to 255.0] | 130.0 [82.0 to 234.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  CD40L_TNF-α, Week 30 | 413.0 [261.0 to 868.0] | 144.5 [48.5 to 268.5] |  | 195.5 [42.5 to 360.5]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_TNF-α, Week 48 | 164.0 [43.0 to 321.0] | 160.5 [29.5 to 321.0] |  | 201.0 [71.0 to 382.0]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_IFN- γ, Pre-vaccination | 229.0 [133.0 to 392.0] | 208.5 [80.0 to 383.0] | 224.0 [99.0 to 392.0] | 209.0 [115.5 to 609.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  CD40L_IFN- γ, Week 6 | 375.0 [201.0 to 619.0] | 233.0 [118.0 to 608.0] | 280.5 [163.5 to 613.5] | 307.0 [178.0 to 532.0]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ, Week 28 | 180.5 [89.0 to 447.0] | 186.5 [94.0 to 412.0] | 181.5 [91.5 to 437.0] | 239.0 [126.0 to 450.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  CD40L_IFN- γ, Week 30 | 325.0 [230.0 to 593.0] | 195.5 [136.0 to 489.0] |  | 254.5 [162.0 to 470.0]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_IFN- γ, Week 48 | 202.0 [129.0 to 447.0] | 202.0 [82.5 to 371.5] |  | 227.0 [115.0 to 466.0]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  TNF-α_IL-2, Pre-vaccination | 23.0 [4.0 to 54.0] | 4.0 [4.0 to 38.0] | 20.0 [4.0 to 43.0] | 4.0 [4.0 to 31.5]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  TNF-α_IL-2, Week 6 | 54.0 [4.0 to 167.0] | 65.0 [29.0 to 112.0] | 60.0 [16.5 to 138.5] | 4.0 [4.0 to 28.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IL-2, Week 28 | 45.5 [4.0 to 103.0] | 20.5 [4.0 to 75.0] | 27.5 [4.0 to 98.5] | 24.0 [4.0 to 36.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  TNF-α_IL-2, Week 30 | 76.0 [23.0 to 208.0] | 17.0 [4.0 to 59.0] |  | 10.5 [4.0 to 45.5]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  TNF-α_IL-2, Week 48 | 36.0 [4.0 to 128.0] | 4.0 [4.0 to 31.5] |  | 6.0 [4.0 to 38.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  IFN- γ_IL-2, Pre-vaccination | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 28.5]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  IFN- γ_IL-2, Week 6 | 19.0 [4.0 to 45.0] | 27.0 [4.0 to 57.0] | 21.5 [4.0 to 49.0] | 4.0 [4.0 to 4.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ_IL-2, Week 28 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 24.0] | 4.0 [4.0 to 24.0] | 4.0 [4.0 to 17.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  IFN- γ_IL-2, Week 30 | 28.0 [4.0 to 67.0] | 4.0 [4.0 to 30.5] |  | 4.0 [4.0 to 10.5]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  IFN- γ_IL-2, Week 48 | 4.0 [4.0 to 24.0] | 4.0 [4.0 to 46.5] |  | 4.0 [4.0 to 14.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  TNF-α_IFN- γ, Pre-vaccination | 94.0 [55.0 to 156.0] | 92.0 [60.0 to 194.0] | 93.0 [56.0 to 184.0] | 149.5 [97.0 to 331.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  TNF-α_IFN- γ, Week 6 | 132.0 [53.0 to 246.0] | 123.0 [66.0 to 253.0] | 127.0 [59.0 to 247.5] | 165.0 [66.0 to 413.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ, Week 28 | 111.5 [54.0 to 155.0] | 141.5 [36.0 to 253.0] | 129.5 [40.5 to 216.0] | 90.0 [46.0 to 349.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  TNF-α_IFN- γ, Week 30 | 110.0 [50.0 to 195.0] | 127.0 [68.5 to 268.5] |  | 153.5 [46.0 to 355.0]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  TNF-α_IFN- γ, Week 48 | 72.0 [44.0 to 171.0] | 98.5 [41.5 to 263.0] |  | 143.0 [74.0 to 334.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_TNF-α_IL-2, Pre-vaccination | 110.0 [31.0 to 193.0] | 109.5 [40.0 to 203.0] | 110.0 [31.0 to 195.0] | 126.0 [46.5 to 239.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  CD40L_TNF-α_IL-2, Week 6 | 889.0 [498.0 to 1600.0] | 529.0 [307.0 to 1187.0] | 730.5 [316.5 to 1340.5] | 134.0 [57.0 to 234.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IL-2, Week 28 | 312.0 [178.0 to 765.0] | 247.0 [88.0 to 470.0] | 286.5 [138.0 to 576.5] | 114.0 [60.0 to 215.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  CD40L_TNF-α_IL-2, Week 30 | 953.0 [466.0 to 2115.0] | 244.5 [101.5 to 410.0] |  | 182.5 [60.0 to 266.5]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_TNF-α_IL-2, Week 48 | 367.0 [125.0 to 1226.0] | 174.0 [60.5 to 384.0] |  | 81.0 [24.0 to 131.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_IFN- γ_IL-2, Pre-vaccination | 46.0 [19.0 to 72.0] | 45.0 [4.0 to 104.0] | 46.0 [18.0 to 79.0] | 43.0 [23.0 to 110.5]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  CD40L_IFN- γ_IL-2, Week 6 | 331.0 [109.0 to 533.0] | 208.0 [88.0 to 462.0] | 253.0 [89.5 to 500.5] | 68.5 [26.0 to 129.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ_IL-2, Week 28 | 88.0 [27.0 to 129.0] | 87.5 [33.0 to 163.0] | 87.5 [32.5 to 137.5] | 37.0 [4.0 to 83.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  CD40L_IFN- γ_IL-2, Week 30 | 336.0 [131.0 to 462.0] | 77.5 [18.5 to 218.0] |  | 55.0 [24.0 to 101.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_IFN- γ_IL-2, Week 48 | 92.0 [26.0 to 170.0] | 58.0 [10.5 to 156.5] |  | 53.0 [6.0 to 112.0]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 149.0 [40.0 to 304.0] | 152.5 [44.0 to 248.0] | 150.0 [40.0 to 297.0] | 154.5 [96.5 to 349.5]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  CD40L_TNF-α_IFN- γ, Week 6 | 341.0 [132.0 to 596.0] | 264.0 [112.0 to 433.0] | 289.0 [125.5 to 521.5] | 172.5 [62.0 to 324.0]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ, Week 28 | 123.5 [87.0 to 253.0] | 131.0 [69.0 to 268.0] | 131.0 [79.0 to 267.5] | 154.0 [48.0 to 265.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  CD40L_TNF-α_IFN- γ, Week 30 | 291.0 [201.0 to 509.0] | 149.5 [86.0 to 283.0] |  | 142.0 [86.5 to 326.5]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_TNF-α_IFN- γ, Week 48 | 187.0 [76.0 to 323.0] | 129.5 [42.0 to 290.5] |  | 121.0 [60.0 to 378.0]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 4.0 [4.0 to 27.0] | 4.0 [4.0 to 22.0] | 4.0 [4.0 to 24.0] | 4.0 [4.0 to 21.5]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 37
  TNF-α_IFN- γ_IL-2, Week 6 | 40.0 [4.0 to 70.0] | 21.0 [4.0 to 66.0] | 32.5 [4.0 to 69.5] | 4.0 [4.0 to 35.0]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ_IL-2, Week 28 | 13.0 [4.0 to 40.0] | 10.5 [4.0 to 53.0] | 12.0 [4.0 to 42.0] | 4.0 [4.0 to 27.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 37
  TNF-α_IFN- γ_IL-2, Week 30 | 36.0 [4.0 to 83.0] | 4.0 [4.0 to 25.0] |  | 4.0 [4.0 to 10.5]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 37
  TNF-α_IFN- γ_IL-2, Week 48 | 18.0 [4.0 to 63.0] | 4.0 [4.0 to 29.0] |  | 4.0 [4.0 to 30.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 106.0 [31.0 to 191.0] | 93.0 [22.0 to 181.0] | 95.0 [25.0 to 191.0] | 131.5 [24.5 to 196.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 624.0 [349.0 to 1399.0] | 441.0 [206.0 to 1044.0] | 532.0 [239.5 to 1079.5] | 146.5 [90.0 to 317.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 235.5 [121.0 to 400.0] | 147.0 [61.0 to 347.0] | 205.5 [85.0 to 396.0] | 91.0 [31.0 to 186.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 37 | 36 | 0 | 36
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 747.0 [479.0 to 2069.0] | 110.5 [55.0 to 502.0] |  | 108.0 [35.5 to 189.5]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 367.0 [80.0 to 657.0] | 132.0 [55.5 to 332.0] |  | 72.0 [44.0 to 232.0]

39. Secondary Outcome: Cytokine Expression Profile of Nef Antigen-specific CD4+ T-cells
Description: The cytokine co-expression profile was defined by the frequency of Nef-specific CD4+ T-cells expressing CD40L and/or IL-2 and/or tumour necrosis factor-alpha (TNF-α) and/or interferon-gamma (IFN-γ).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: Nef-specific CD4+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 41 | 42 | 79 | 37
Nef-specific CD4+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L, Pre-vaccination | 1.0 [1.0 to 331.0] | 1.0 [1.0 to 230.0] | 1.0 [1.0 to 280.0] | 1.0 [1.0 to 390.0]
  CD40L, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  CD40L, Week 6 | 1.0 [1.0 to 194.0] | 1.0 [1.0 to 280.0] | 1.0 [1.0 to 194.0] | 1.0 [1.0 to 34.0]
  CD40L, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L, Week 28 | 1.0 [1.0 to 113.0] | 1.0 [1.0 to 210.0] | 1.0 [1.0 to 158.5] | 1.0 [1.0 to 90.0]
  CD40L, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  CD40L, Week 30 | 1.0 [1.0 to 50.0] | 98.5 [1.0 to 357.5] |  | 1.0 [1.0 to 185.0]
  CD40L, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L, Week 48 | 1.0 [1.0 to 75.0] | 1.0 [1.0 to 420.0] |  | 1.0 [1.0 to 218.0]
  IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IL-2, Pre-vaccination | 14.0 [1.0 to 32.0] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 32.0] | 1.0 [1.0 to 30.0]
  IL-2, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  IL-2, Week 6 | 22.0 [1.0 to 59.0] | 7.0 [1.0 to 43.0] | 14.0 [1.0 to 45.0] | 1.0 [1.0 to 27.0]
  IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IL-2, Week 28 | 4.0 [1.0 to 45.0] | 1.0 [1.0 to 46.0] | 1.5 [1.0 to 45.5] | 1.0 [1.0 to 28.0]
  IL-2, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  IL-2, Week 30 | 19.0 [1.0 to 108.0] | 1.0 [1.0 to 44.5] |  | 1.0 [1.0 to 30.5]
  IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  IL-2, Week 48 | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 26.0] |  | 1.0 [1.0 to 15.0]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α, Pre-vaccination | 18.0 [1.0 to 94.0] | 1.0 [1.0 to 104.0] | 1.0 [1.0 to 104.0] | 1.0 [1.0 to 149.0]
  TNF-α, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  TNF-α, Week 6 | 31.0 [1.0 to 135.0] | 37.5 [1.0 to 164.0] | 32.0 [1.0 to 137.0] | 1.0 [1.0 to 43.0]
  TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α, Week 28 | 5.0 [1.0 to 58.0] | 1.0 [1.0 to 50.0] | 1.0 [1.0 to 53.0] | 1.0 [1.0 to 52.0]
  TNF-α, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  TNF-α, Week 30 | 43.5 [1.0 to 181.0] | 7.5 [1.0 to 109.0] |  | 1.0 [1.0 to 120.0]
  TNF-α, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  TNF-α, Week 48 | 82.5 [1.0 to 203.5] | 1.0 [1.0 to 63.0] |  | 1.0 [1.0 to 187.5]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IFN- γ, Pre-vaccination | 84.0 [38.0 to 124.0] | 62.5 [11.0 to 323.0] | 83.0 [22.0 to 178.0] | 87.0 [21.0 to 229.0]
  IFN- γ, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  IFN- γ, Week 6 | 101.0 [31.0 to 216.0] | 105.5 [41.0 to 182.0] | 103.0 [31.0 to 195.0] | 81.0 [31.0 to 202.0]
  IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ, Week 28 | 24.0 [1.0 to 174.0] | 114.5 [24.0 to 197.0] | 67.0 [1.0 to 179.5] | 101.0 [49.0 to 161.0]
  IFN- γ, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  IFN- γ, Week 30 | 83.0 [31.0 to 144.0] | 118.5 [31.5 to 201.0] |  | 99.5 [50.0 to 238.5]
  IFN- γ, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  IFN- γ, Week 48 | 61.5 [15.0 to 107.0] | 69.0 [24.0 to 160.0] |  | 79.0 [6.0 to 180.5]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IL-2, Pre-vaccination | 1.0 [1.0 to 44.0] | 2.0 [1.0 to 39.0] | 1.0 [1.0 to 40.0] | 1.0 [1.0 to 24.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  CD40L_IL-2, Week 6 | 111.0 [19.0 to 262.0] | 65.5 [1.0 to 190.0] | 78.0 [1.0 to 244.0] | 16.0 [1.0 to 41.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IL-2, Week 28 | 25.0 [1.0 to 104.0] | 9.5 [1.0 to 60.0] | 21.5 [1.0 to 73.5] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  CD40L_IL-2, Week 30 | 112.5 [57.0 to 259.0] | 1.0 [1.0 to 70.0] |  | 1.0 [1.0 to 10.0]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_IL-2, Week 48 | 1.0 [1.0 to 84.5] | 15.0 [1.0 to 78.0] |  | 1.0 [1.0 to 33.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α, Pre-vaccination | 6.0 [1.0 to 43.0] | 7.5 [1.0 to 57.0] | 6.0 [1.0 to 50.0] | 1.0 [1.0 to 7.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 37
  CD40L_TNF-α, Week 6 | 75.0 [1.0 to 155.0] | 42.0 [4.0 to 82.0] | 46.0 [1.0 to 127.0] | 1.0 [1.0 to 32.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α, Week 28 | 2.5 [1.0 to 38.0] | 3.0 [1.0 to 41.0] | 3.0 [1.0 to 39.5] | 1.0 [1.0 to 26.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 37
  CD40L_TNF-α, Week 30 | 141.0 [20.0 to 218.0] | 1.0 [1.0 to 39.5] |  | 1.0 [1.0 to 50.5]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 37
  CD40L_TNF-α, Week 48 | 22.5 [1.0 to 63.5] | 11.0 [1.0 to 49.0] |  | 1.0 [1.0 to 32.0]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IFN- γ, Pre-vaccination | 1.0 [1.0 to 28.0] | 7.5 [1.0 to 36.0] | 1.0 [1.0 to 31.0] | 20.0 [1.0 to 43.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  CD40L_IFN- γ, Week 6 | 31.0 [1.0 to 89.0] | 31.0 [1.0 to 55.0] | 31.0 [1.0 to 79.0] | 1.0 [1.0 to 22.0]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ, Week 28 | 1.0 [1.0 to 36.0] | 12.5 [1.0 to 31.0] | 1.0 [1.0 to 35.0] | 1.0 [1.0 to 48.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  CD40L_IFN- γ, Week 30 | 59.0 [23.0 to 133.0] | 1.0 [1.0 to 36.5] |  | 7.5 [1.0 to 42.5]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_IFN- γ, Week 48 | 10.0 [1.0 to 46.0] | 1.0 [1.0 to 31.0] |  | 1.0 [1.0 to 32.5]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  TNF-α_IL-2, Week 6 | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IL-2, Week 28 | 15.0 [1.0 to 36.0] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 14.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  TNF-α_IL-2, Week 30 | 7.5 [1.0 to 55.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  TNF-α_IL-2, Week 48 | 1.0 [1.0 to 20.5] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IFN- γ, Pre-vaccination | 1.0 [1.0 to 34.0] | 21.5 [1.0 to 63.0] | 15.0 [1.0 to 46.0] | 20.0 [1.0 to 64.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  TNF-α_IFN- γ, Week 6 | 26.0 [1.0 to 44.0] | 8.0 [1.0 to 65.0] | 19.0 [1.0 to 49.0] | 14.0 [1.0 to 54.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ, Week 28 | 18.0 [1.0 to 43.0] | 3.0 [1.0 to 96.0] | 15.0 [1.0 to 59.5] | 24.0 [1.0 to 60.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  TNF-α_IFN- γ, Week 30 | 14.5 [1.0 to 38.0] | 45.5 [1.0 to 77.5] |  | 17.5 [1.0 to 53.0]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  TNF-α_IFN- γ, Week 48 | 1.0 [1.0 to 44.0] | 13.0 [1.0 to 61.0] |  | 16.0 [1.0 to 74.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 37.0] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 29.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  CD40L_TNF-α_IL-2, Week 6 | 207.0 [62.0 to 394.0] | 110.5 [13.0 to 234.0] | 137.0 [37.0 to 305.0] | 1.0 [1.0 to 18.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IL-2, Week 28 | 74.0 [1.0 to 244.0] | 57.5 [1.0 to 123.0] | 67.5 [1.0 to 166.0] | 1.0 [1.0 to 19.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  CD40L_TNF-α_IL-2, Week 30 | 327.0 [113.0 to 572.0] | 38.5 [1.0 to 107.0] |  | 1.5 [1.0 to 37.0]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_TNF-α_IL-2, Week 48 | 78.5 [6.5 to 329.0] | 32.0 [1.0 to 98.0] |  | 1.0 [1.0 to 19.5]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  CD40L_IFN- γ_IL-2, Week 6 | 44.0 [1.0 to 111.0] | 6.5 [1.0 to 93.0] | 22.0 [1.0 to 102.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 22.5] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  CD40L_IFN- γ_IL-2, Week 30 | 74.5 [18.0 to 169.0] | 1.0 [1.0 to 12.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 29.5] | 1.0 [1.0 to 21.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 37.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  CD40L_TNF-α_IFN- γ, Week 6 | 17.0 [1.0 to 111.0] | 16.5 [1.0 to 57.0] | 17.0 [1.0 to 65.0] | 1.0 [1.0 to 32.0]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ, Week 28 | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 25.5] | 1.0 [1.0 to 27.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  CD40L_TNF-α_IFN- γ, Week 30 | 43.0 [1.0 to 120.0] | 1.0 [1.0 to 23.0] |  | 1.0 [1.0 to 33.0]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ, Week 48 | 1.0 [1.0 to 37.5] | 1.0 [1.0 to 33.0] |  | 1.0 [1.0 to 40.0]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 16.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 38 | 73 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 77.0 [13.0 to 222.0] | 53.0 [22.0 to 103.0] | 66.0 [22.0 to 149.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 26.0 [1.0 to 97.0] | 7.5 [1.0 to 42.0] | 20.0 [1.0 to 53.0] | 1.0 [1.0 to 21.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 36 | 0 | 36
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 142.5 [48.0 to 478.0] | 14.5 [1.0 to 51.5] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 43.0 [1.0 to 150.0] | 1.0 [1.0 to 39.0] |  | 1.0 [1.0 to 1.0]

40. Secondary Outcome: Cytokine Expression Profile of P17 Antigen-specific CD4+ T-cells
Description: The cytokine co-expression profile was defined by the frequency of P17-specific CD4+ T-cells expressing CD40L and/or IL-2 and/or tumour necrosis factor-alpha (TNF-α) and/or interferon-gamma (IFN-γ).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: P17-specific CD4+ T-cells/million T-cell
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 41 | 42 | 79 | 37
P17-specific CD4+ T-cells/million T-cell
  CD40L, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L, Pre-vaccination | 180.0 [1.0 to 440.0] | 1.0 [1.0 to 240.0] | 68.0 [1.0 to 380.0] | 1.0 [1.0 to 311.5]
  CD40L, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L, Week 6 | 1.0 [1.0 to 152.5] | 1.0 [1.0 to 340.0] | 1.0 [1.0 to 212.0] | 1.0 [1.0 to 123.0]
  CD40L, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L, Week 28 | 100.0 [1.0 to 270.0] | 60.5 [1.0 to 200.0] | 80.0 [1.0 to 257.0] | 1.0 [1.0 to 230.0]
  CD40L, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  CD40L, Week 30 | 1.0 [1.0 to 440.0] | 133.0 [1.0 to 420.0] |  | 198.0 [1.0 to 415.0]
  CD40L, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L, Week 48 | 1.0 [1.0 to 390.0] | 72.0 [1.0 to 370.0] |  | 150.0 [1.0 to 385.0]
  IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  IL-2, Pre-vaccination | 1.0 [1.0 to 72.0] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 43.0] | 9.0 [1.0 to 34.0]
  IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  IL-2, Week 6 | 1.5 [1.0 to 34.5] | 20.0 [1.0 to 85.0] | 6.0 [1.0 to 43.0] | 1.0 [1.0 to 45.0]
  IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IL-2, Week 28 | 1.0 [1.0 to 16.0] | 27.5 [1.0 to 63.0] | 1.5 [1.0 to 39.0] | 1.0 [1.0 to 23.0]
  IL-2, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  IL-2, Week 30 | 12.0 [1.0 to 44.0] | 1.0 [1.0 to 33.0] |  | 1.0 [1.0 to 26.5]
  IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IL-2, Week 48 | 1.0 [1.0 to 33.0] | 9.0 [1.0 to 43.0] |  | 1.0 [1.0 to 29.0]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  TNF-α, Pre-vaccination | 24.0 [1.0 to 93.0] | 25.5 [1.0 to 166.0] | 25.0 [1.0 to 130.0] | 13.5 [1.0 to 165.5]
  TNF-α, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  TNF-α, Week 6 | 26.5 [1.0 to 147.0] | 41.5 [1.0 to 99.0] | 36.0 [1.0 to 130.0] | 31.5 [1.0 to 175.0]
  TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α, Week 28 | 57.0 [1.0 to 155.0] | 1.0 [1.0 to 101.0] | 26.0 [1.0 to 122.5] | 27.0 [1.0 to 89.0]
  TNF-α, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  TNF-α, Week 30 | 51.0 [1.0 to 162.0] | 1.0 [1.0 to 82.0] |  | 1.5 [1.0 to 171.5]
  TNF-α, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α, Week 48 | 4.0 [1.0 to 110.0] | 1.0 [1.0 to 88.0] |  | 1.0 [1.0 to 155.5]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  IFN- γ, Pre-vaccination | 51.0 [1.0 to 123.0] | 71.0 [1.0 to 131.0] | 55.0 [1.0 to 127.0] | 76.0 [5.0 to 215.5]
  IFN- γ, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  IFN- γ, Week 6 | 88.5 [7.0 to 135.0] | 75.5 [19.0 to 147.0] | 83.0 [15.0 to 142.0] | 88.0 [28.0 to 255.0]
  IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ, Week 28 | 44.0 [1.0 to 92.0] | 82.0 [22.0 to 158.0] | 65.5 [11.0 to 121.0] | 73.0 [10.0 to 199.0]
  IFN- γ, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  IFN- γ, Week 30 | 77.0 [12.0 to 132.0] | 54.0 [14.0 to 179.0] |  | 57.5 [36.0 to 146.0]
  IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IFN- γ, Week 48 | 72.0 [6.0 to 123.0] | 74.0 [15.0 to 134.0] |  | 84.5 [22.0 to 180.5]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_IL-2, Pre-vaccination | 31.0 [1.0 to 63.0] | 6.0 [1.0 to 44.0] | 23.0 [1.0 to 63.0] | 1.0 [1.0 to 25.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_IL-2, Week 6 | 58.5 [3.0 to 107.0] | 21.5 [1.0 to 65.0] | 33.0 [1.0 to 101.0] | 19.0 [1.0 to 62.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IL-2, Week 28 | 34.5 [1.0 to 69.0] | 20.0 [1.0 to 54.0] | 28.0 [1.0 to 62.5] | 1.0 [1.0 to 27.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  CD40L_IL-2, Week 30 | 56.0 [1.0 to 101.0] | 14.0 [1.0 to 60.0] |  | 1.0 [1.0 to 38.5]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IL-2, Week 48 | 1.0 [1.0 to 37.0] | 42.0 [1.0 to 88.0] |  | 34.5 [1.0 to 63.5]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_TNF-α, Pre-vaccination | 24.0 [1.0 to 74.0] | 16.0 [1.0 to 74.0] | 21.0 [1.0 to 74.0] | 6.5 [1.0 to 38.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_TNF-α, Week 6 | 58.5 [3.0 to 145.0] | 34.5 [1.0 to 88.0] | 45.0 [2.0 to 118.0] | 30.5 [1.0 to 67.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α, Week 28 | 39.5 [1.0 to 102.0] | 6.0 [1.0 to 57.0] | 23.0 [1.0 to 64.5] | 26.0 [1.0 to 47.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  CD40L_TNF-α, Week 30 | 26.0 [1.0 to 68.0] | 22.0 [1.0 to 66.0] |  | 21.5 [1.0 to 85.5]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α, Week 48 | 11.0 [1.0 to 51.0] | 20.0 [1.0 to 78.0] |  | 32.5 [1.0 to 91.5]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_IFN- γ, Pre-vaccination | 41.0 [1.0 to 94.0] | 42.0 [1.0 to 80.0] | 41.0 [1.0 to 94.0] | 48.0 [29.0 to 149.5]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_IFN- γ, Week 6 | 76.0 [28.0 to 126.5] | 42.0 [17.0 to 96.0] | 56.0 [25.0 to 113.0] | 70.0 [44.0 to 149.0]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ, Week 28 | 33.5 [1.0 to 93.0] | 49.0 [1.0 to 132.0] | 41.0 [1.0 to 117.5] | 64.0 [40.0 to 125.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  CD40L_IFN- γ, Week 30 | 79.0 [39.0 to 169.0] | 35.0 [22.0 to 84.0] |  | 56.0 [22.5 to 146.5]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IFN- γ, Week 48 | 44.0 [21.0 to 101.0] | 43.0 [1.0 to 108.0] |  | 49.0 [22.5 to 95.5]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  TNF-α_IL-2, Week 6 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IL-2, Week 28 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  TNF-α_IL-2, Week 30 | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IL-2, Week 48 | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 19.5]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  TNF-α_IFN- γ, Pre-vaccination | 19.0 [1.0 to 40.0] | 1.0 [1.0 to 41.0] | 16.0 [1.0 to 41.0] | 26.5 [1.0 to 61.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  TNF-α_IFN- γ, Week 6 | 7.5 [1.0 to 35.0] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 33.0] | 22.0 [1.0 to 61.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ, Week 28 | 22.0 [1.0 to 34.0] | 23.5 [1.0 to 64.0] | 22.0 [1.0 to 42.5] | 1.00 [1.0 to 44.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  TNF-α_IFN- γ, Week 30 | 1.0 [1.0 to 40.0] | 20.0 [1.0 to 45.0] |  | 14.0 [1.0 to 80.5]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IFN- γ, Week 48 | 2.0 [1.0 to 25.0] | 11.0 [1.0 to 28.0] |  | 24.0 [1.0 to 57.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_TNF-α_IL-2, Pre-vaccination | 4.0 [1.0 to 42.0] | 16.5 [1.0 to 43.0] | 10.0 [1.0 to 43.0] | 26.0 [1.0 to 56.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_TNF-α_IL-2, Week 6 | 88.0 [3.0 to 124.5] | 64.5 [33.0 to 118.0] | 73.5 [24.0 to 122.0] | 25.0 [1.0 to 47.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IL-2, Week 28 | 51.0 [1.0 to 72.0] | 25.0 [1.0 to 66.0] | 31.5 [1.0 to 71.5] | 6.0 [1.0 to 40.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  CD40L_TNF-α_IL-2, Week 30 | 44.0 [2.0 to 156.0] | 33.0 [1.0 to 63.0] |  | 17.0 [1.0 to 50.5]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IL-2, Week 48 | 33.0 [1.0 to 67.0] | 15.0 [1.0 to 68.0] |  | 1.0 [1.0 to 38.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 29.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_IFN- γ_IL-2, Week 6 | 26.5 [1.0 to 68.5] | 25.0 [1.0 to 54.0] | 25.0 [1.0 to 61.0] | 1.0 [1.0 to 18.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 22.0] | 18.5 [1.0 to 34.0] | 12.5 [1.0 to 28.0] | 1.0 [1.0 to 20.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  CD40L_IFN- γ_IL-2, Week 30 | 20.0 [1.0 to 45.0] | 1.0 [1.0 to 35.0] |  | 1.0 [1.0 to 24.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 17.0] |  | 1.0 [1.0 to 21.5]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 37.0 [1.0 to 96.0] | 35.0 [1.0 to 64.0] | 35.0 [1.0 to 85.0] | 37.0 [7.0 to 86.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_TNF-α_IFN- γ, Week 6 | 54.5 [10.5 to 131.5] | 35.0 [1.0 to 86.0] | 42.0 [1.0 to 118.0] | 37.5 [17.0 to 87.0]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ, Week 28 | 32.5 [4.0 to 45.0] | 28.5 [1.0 to 92.0] | 30.5 [1.0 to 54.5] | 26.0 [1.0 to 99.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  CD40L_TNF-α_IFN- γ, Week 30 | 59.0 [38.0 to 95.0] | 40.0 [13.0 to 94.0] |  | 39.5 [1.0 to 88.5]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ, Week 48 | 26.0 [1.0 to 100.0] | 16.0 [1.0 to 55.0] |  | 22.0 [1.0 to 90.0]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 36
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 22.0 [1.0 to 41.0] | 8.5 [1.0 to 50.0] | 20.0 [1.0 to 43.0] | 12.5 [1.0 to 56.5]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 50.0 [2.5 to 121.5] | 71.5 [31.0 to 123.0] | 64.0 [23.0 to 123.0] | 30.5 [3.0 to 63.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 22.5 [1.0 to 34.0] | 8.5 [1.0 to 69.0] | 21.0 [1.0 to 57.5] | 25.0 [1.0 to 45.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 37 | 37 | 0 | 36
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 46.0 [21.0 to 125.0] | 13.0 [1.0 to 105.0] |  | 27.5 [1.0 to 60.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 42.0 [22.0 to 74.0] | 25.0 [1.0 to 51.0] |  | 14.0 [1.0 to 41.0]

41. Secondary Outcome: Cytokine Expression Profile of P24 Antigen-specific CD4+ T-cells
Description: The cytokine co-expression profile was defined by the frequency of P24-specific CD4+ T-cells expressing CD40L and/or IL-2 and/or tumour necrosis factor-alpha (TNF-α) and/or interferon-gamma (IFN-γ).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: P24-specific CD4+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 41 | 42 | 79 | 37
P24-specific CD4+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L, Pre-vaccination | 115.0 [1.0 to 384.0] | 65.0 [1.0 to 404.0] | 114.0 [1.0 to 404.0] | 70.0 [1.0 to 420.0]
  CD40L, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L, Week 6 | 86.0 [1.0 to 345.5] | 140.5 [1.0 to 470.0] | 110.0 [1.0 to 400.0] | 1.0 [1.0 to 470.0]
  CD40L, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L, Week 28 | 125.0 [1.0 to 380.0] | 194.0 [1.0 to 408.0] | 165.0 [1.0 to 394.0] | 15.0 [1.0 to 380.0]
  CD40L, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L, Week 30 | 22.5 [1.0 to 290.0] | 110.0 [1.0 to 398.0] |  | 130.5 [1.0 to 416.0]
  CD40L, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L, Week 48 | 1.0 [1.0 to 282.0] | 160.0 [1.0 to 569.0] |  | 125.0 [1.0 to 490.5]
  IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IL-2, Pre-vaccination | 21.0 [1.0 to 59.0] | 3.0 [1.0 to 49.0] | 5.0 [1.0 to 55.0] | 1.0 [1.0 to 33.0]
  IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  IL-2, Week 6 | 1.0 [1.0 to 58.5] | 6.0 [1.0 to 37.0] | 1.0 [1.0 to 44.0] | 1.0 [1.0 to 24.0]
  IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IL-2, Week 28 | 2.5 [1.0 to 32.0] | 1.0 [1.0 to 44.0] | 1.0 [1.0 to 34.5] | 1.0 [1.0 to 29.0]
  IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  IL-2, Week 30 | 22.0 [1.0 to 74.0] | 1.0 [1.0 to 37.0] |  | 1.0 [1.0 to 32.0]
  IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IL-2, Week 48 | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 32.0] |  | 19.0 [1.0 to 60.5]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α, Pre-vaccination | 79.0 [13.0 to 172.0] | 11.5 [1.0 to 134.0] | 58.0 [1.0 to 168.0] | 21.0 [1.0 to 153.0]
  TNF-α, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  TNF-α, Week 6 | 24.5 [1.0 to 103.0] | 32.5 [1.0 to 126.0] | 32.0 [1.0 to 109.0] | 1.0 [1.0 to 133.0]
  TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α, Week 28 | 34.0 [1.0 to 120.0] | 1.0 [1.0 to 32.0] | 4.5 [1.0 to 64.0] | 39.0 [1.0 to 180.0]
  TNF-α, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  TNF-α, Week 30 | 65.0 [1.0 to 234.0] | 1.0 [1.0 to 148.0] |  | 20.5 [1.0 to 171.0]
  TNF-α, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α, Week 48 | 67.0 [1.0 to 258.0] | 40.0 [1.0 to 89.0] |  | 12.0 [1.0 to 182.5]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IFN- γ, Pre-vaccination | 124.0 [53.0 to 249.0] | 112.0 [46.0 to 275.0] | 124.0 [46.0 to 275.0] | 164.0 [105.0 to 561.0]
  IFN- γ, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  IFN- γ, Week 6 | 139.0 [50.5 to 242.0] | 125.0 [62.0 to 320.0] | 128.5 [59.0 to 267.0] | 233.5 [123.0 to 653.0]
  IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ, Week 28 | 99.5 [53.0 to 199.0] | 118.5 [45.0 to 326.0] | 105.0 [51.5 to 282.5] | 271.0 [75.0 to 494.0]
  IFN- γ, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  IFN- γ, Week 30 | 157.5 [60.0 to 290.0] | 167.0 [61.0 to 375.0] |  | 224.5 [67.5 to 432.5]
  IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IFN- γ, Week 48 | 96.0 [47.0 to 235.0] | 171.0 [74.0 to 323.0] |  | 266.0 [89.5 to 621.0]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IL-2, Pre-vaccination | 43.0 [1.0 to 81.0] | 22.0 [1.0 to 51.0] | 35.0 [1.0 to 67.0] | 22.0 [1.0 to 54.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_IL-2, Week 6 | 45.5 [1.0 to 163.0] | 36.5 [1.0 to 119.0] | 41.5 [1.0 to 129.0] | 17.5 [1.0 to 61.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IL-2, Week 28 | 31.0 [1.0 to 79.0] | 31.5 [1.0 to 86.0] | 31.5 [1.0 to 84.0] | 13.0 [1.0 to 46.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_IL-2, Week 30 | 46.5 [1.0 to 74.0] | 51.0 [12.0 to 83.0] |  | 9.5 [1.0 to 67.0]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IL-2, Week 48 | 30.0 [1.0 to 108.0] | 34.0 [1.0 to 80.0] |  | 2.0 [1.0 to 38.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α, Pre-vaccination | 68.0 [39.0 to 104.0] | 30.0 [1.0 to 73.0] | 58.0 [2.0 to 95.0] | 38.0 [1.0 to 92.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_TNF-α, Week 6 | 55.0 [1.0 to 105.5] | 72.0 [15.0 to 108.0] | 64.5 [8.0 to 108.0] | 26.0 [1.0 to 89.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α, Week 28 | 49.0 [1.0 to 111.0] | 13.0 [1.0 to 61.0] | 29.5 [1.0 to 82.5] | 46.0 [1.0 to 112.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_TNF-α, Week 30 | 86.5 [15.0 to 165.0] | 48.0 [1.0 to 90.0] |  | 61.5 [2.5 to 124.5]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α, Week 48 | 63.0 [1.0 to 130.0] | 6.0 [1.0 to 137.0] |  | 48.0 [14.0 to 109.5]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IFN- γ, Pre-vaccination | 127.0 [60.0 to 200.0] | 96.5 [43.0 to 199.0] | 119.0 [45.0 to 200.0] | 120.0 [48.0 to 319.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_IFN- γ, Week 6 | 122.5 [50.5 to 201.5] | 81.5 [41.0 to 240.0] | 98.0 [43.0 to 218.0] | 129.5 [68.0 to 312.0]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ, Week 28 | 87.5 [46.0 to 203.0] | 94.0 [44.0 to 168.0] | 89.0 [45.0 to 186.0] | 106.0 [61.0 to 210.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_IFN- γ, Week 30 | 113.5 [65.0 to 195.0] | 106.0 [53.0 to 231.0] |  | 137.5 [61.0 to 202.5]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IFN- γ, Week 48 | 79.0 [42.0 to 200.0] | 102.0 [44.0 to 204.0] |  | 99.5 [49.5 to 200.0]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  TNF-α_IL-2, Week 6 | 1.0 [1.0 to 24.0] | 1.5 [1.0 to 29.0] | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IL-2, Week 28 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 13.5] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  TNF-α_IL-2, Week 30 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 14.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IL-2, Week 48 | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 12.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IFN- γ, Pre-vaccination | 22.0 [1.0 to 61.0] | 42.0 [19.0 to 86.0] | 35.0 [1.0 to 80.0] | 53.0 [26.0 to 173.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  TNF-α_IFN- γ, Week 6 | 34.0 [1.0 to 82.0] | 34.0 [1.0 to 64.0] | 34.0 [1.0 to 70.0] | 56.5 [1.0 to 254.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ, Week 28 | 28.0 [1.0 to 65.0] | 41.5 [1.0 to 107.0] | 33.5 [1.0 to 87.5] | 29.0 [1.0 to 223.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  TNF-α_IFN- γ, Week 30 | 26.5 [1.0 to 75.0] | 43.0 [15.0 to 72.0] |  | 52.0 [7.0 to 211.5]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IFN- γ, Week 48 | 24.0 [1.0 to 59.0] | 40.0 [20.0 to 76.0] |  | 46.0 [3.5 to 101.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IL-2, Pre-vaccination | 19.0 [1.0 to 73.0] | 20.5 [1.0 to 55.0] | 20.0 [1.0 to 65.0] | 36.0 [2.0 to 65.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_TNF-α_IL-2, Week 6 | 98.0 [22.5 to 185.0] | 80.0 [51.0 to 162.0] | 87.0 [25.0 to 170.0] | 29.5 [1.0 to 87.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IL-2, Week 28 | 41.5 [1.0 to 130.0] | 36.0 [1.0 to 102.0] | 39.0 [1.0 to 105.0] | 25.0 [1.0 to 55.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_TNF-α_IL-2, Week 30 | 79.5 [29.0 to 172.0] | 44.0 [13.0 to 97.0] |  | 32.5 [1.0 to 98.0]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IL-2, Week 48 | 78.0 [10.0 to 112.0] | 31.0 [1.0 to 103.0] |  | 45.0 [4.0 to 78.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 44.0] | 1.0 [1.0 to 30.0] | 16.0 [1.0 to 32.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_IFN- γ_IL-2, Week 6 | 30.5 [1.0 to 59.5] | 30.0 [1.0 to 63.0] | 30.5 [1.0 to 60.0] | 29.0 [1.0 to 57.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ_IL-2, Week 28 | 19.5 [1.0 to 39.0] | 21.5 [1.0 to 58.0] | 21.5 [1.0 to 43.0] | 2.0 [1.0 to 27.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_IFN- γ_IL-2, Week 30 | 41.0 [1.0 to 91.0] | 14.0 [1.0 to 69.0] |  | 17.0 [1.0 to 41.5]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 55.0] | 21.0 [1.0 to 54.0] |  | 16.0 [1.0 to 55.5]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 59.0 [1.0 to 161.0] | 85.5 [15.0 to 149.0] | 72.0 [1.0 to 150.0] | 71.0 [33.0 to 212.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_TNF-α_IFN- γ, Week 6 | 68.0 [34.0 to 159.5] | 84.5 [30.0 to 147.0] | 74.5 [31.0 to 147.0] | 62.5 [20.0 to 158.0]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ, Week 28 | 70.0 [24.0 to 121.0] | 54.0 [1.0 to 173.0] | 58.5 [10.5 to 125.5] | 59.0 [7.0 to 138.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_TNF-α_IFN- γ, Week 30 | 83.5 [37.0 to 162.0] | 57.0 [1.0 to 125.0] |  | 83.5 [26.0 to 165.0]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ, Week 48 | 64.0 [30.0 to 157.0] | 61.0 [1.0 to 122.0] |  | 68. [28.5 to 133.0]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 16.5] | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 19.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 41.0 [1.0 to 88.0] | 38.0 [1.0 to 67.0] | 40.0 [1.0 to 79.0] | 36.0 [1.0 to 85.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 36 | 38 | 74 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 62.5 [3.5 to 128.5] | 58.0 [1.0 to 120.0] | 59.0 [1.0 to 120.0] | 52.5 [17.0 to 85.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 52.0 [28.0 to 104.0] | 41.0 [1.0 to 88.0] | 49.5 [1.0 to 90.0] | 27.0 [1.0 to 118.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 85.5 [23.0 to 206.0] | 46.0 [1.0 to 118.0] |  | 24.0 [1.0 to 62.5]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 57.0 [1.0 to 143.0] | 53.0 [11.0 to 86.0] |  | 24.0 [1.0 to 84.5]

42. Secondary Outcome: Cytokine Expression Profile of RT Antigen-specific CD4+ T-cells
Description: The cytokine co-expression profile was defined by the frequency of reverse transcriptase (RT)-specific CD4+ T-cells expressing CD40L and/or IL-2 and/or tumour necrosis factor-alpha (TNF-α) and/or interferon-gamma (IFN-γ).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: RT-specific CD4+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 41 | 42 | 79 | 37
RT-specific CD4+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L, Pre-vaccination | 24.0 [1.0 to 701.0] | 78.5 [1.0 to 472.0] | 41.0 [1.0 to 590.0] | 1.0 [1.0 to 380.0]
  CD40L, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  CD40L, Week 6 | 1.0 [1.0 to 460.0] | 40.0 [1.0 to 260.0] | 20.5 [1.0 to 285.0] | 1.0 [1.0 to 150.0]
  CD40L, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L, Week 28 | 1.0 [1.0 to 230.0] | 1.0 [1.0 to 200.0] | 1.0 [1.0 to 206.5] | 1.0 [1.0 to 207.0]
  CD40L, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L, Week 30 | 1.0 [1.0 to 350.0] | 90.0 [1.0 to 441.0] |  | 135.0 [1.0 to 365.0]
  CD40L, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L, Week 48 | 1.0 [1.0 to 359.0] | 44.5 [1.0 to 423.0] |  | 30.0 [1.0 to 328.0]
  IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IL-2, Pre-vaccination | 21.0 [1.0 to 62.0] | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 62.0] | 9.0 [1.0 to 59.0]
  IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  IL-2, Week 6 | 34.0 [1.0 to 121.0] | 12.0 [1.0 to 50.0] | 14.0 [1.0 to 63.5] | 13.0 [1.0 to 35.0]
  IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IL-2, Week 28 | 1.0 [1.0 to 66.0] | 1.0 [1.0 to 50.0] | 1.0 [1.0 to 62.5] | 1.0 [1.0 to 3.0]
  IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  IL-2, Week 30 | 25.5 [1.0 to 101.0] | 5.0 [1.0 to 49.0] |  | 1.0 [1.0 to 48.5]
  IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  IL-2, Week 48 | 20.0 [1.0 to 55.5] | 8.0 [1.0 to 48.0] |  | 4.0 [1.0 to 30.0]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α, Pre-vaccination | 61.0 [17.0 to 106.0] | 18.0 [1.0 to 199.0] | 40.0 [1.0 to 170.0] | 46.0 [1.0 to 233.0]
  TNF-α, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  TNF-α, Week 6 | 78.0 [1.0 to 285.0] | 69.0 [13.0 to 126.0] | 73.5 [1.5 to 172.5] | 1.0 [1.0 to 116.0]
  TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α, Week 28 | 40.0 [1.0 to 136.0] | 1.0 [1.0 to 62.0] | 1.0 [1.0 to 72.0] | 41.0 [1.0 to 112.0]
  TNF-α, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  TNF-α, Week 30 | 85.0 [3.0 to 250.0] | 11.0 [1.0 to 133.0] |  | 41.0 [1.0 to 171.5]
  TNF-α, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  TNF-α, Week 48 | 59.5 [1.0 to 180.0] | 1.0 [1.0 to 87.0] |  | 30.0 [1.0 to 127.0]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IFN- γ, Pre-vaccination | 21.0 [1.0 to 75.0] | 25.5 [1.0 to 108.0] | 23.0 [1.0 to 89.0] | 45.0 [1.0 to 70.0]
  IFN- γ, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  IFN- γ, Week 6 | 85.0 [32.0 to 159.0] | 27.0 [1.0 to 106.0] | 65.0 [10.5 to 144.0] | 28.0 [1.0 to 64.0]
  IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ, Week 28 | 18.5 [1.0 to 96.0] | 27.0 [1.0 to 77.0] | 21.5 [1.0 to 90.5] | 44.0 [9.0 to 97.0]
  IFN- γ, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  IFN- γ, Week 30 | 57.5 [27.0 to 125.0] | 40.0 [3.0 to 90.0] |  | 47.0 [6.0 to 88.5]
  IFN- γ, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  IFN- γ, Week 48 | 42.0 [1.0 to 84.0] | 46.0 [1.0 to 114.0] |  | 55.0 [10.0 to 92.0]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IL-2, Pre-vaccination | 44.0 [1.0 to 108.0] | 43.5 [5.0 to 85.0] | 44.0 [1.0 to 95.0] | 11.0 [1.0 to 49.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  CD40L_IL-2, Week 6 | 183.0 [56.0 to 450.0] | 179.0 [78.0 to 277.0] | 181.0 [66.0 to 380.5] | 27.0 [1.0 to 90.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IL-2, Week 28 | 64.0 [1.0 to 143.0] | 80.0 [20.0 to 148.0] | 77.5 [5.0 to 145.5] | 15.0 [1.0 to 36.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_IL-2, Week 30 | 118.5 [84.0 to 352.0] | 57.0 [5.0 to 153.0] |  | 30.0 [1.0 to 66.0]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_IL-2, Week 48 | 63.0 [12.5 to 126.5] | 45.5 [1.0 to 105.0] |  | 3.0 [1.0 to 62.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α, Pre-vaccination | 36.0 [1.0 to 99.0] | 39.0 [1.0 to 68.0] | 37.0 [1.0 to 86.0] | 30.0 [1.0 to 78.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  CD40L_TNF-α, Week 6 | 156.0 [79.0 to 293.0] | 116.0 [1.0 to 197.0] | 132.5 [46.5 to 219.5] | 32.0 [1.0 to 64.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α, Week 28 | 35.5 [2.0 to 76.0] | 22.5 [1.0 to 95.0] | 30.5 [1.0 to 89.5] | 28.0 [1.0 to 73.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_TNF-α, Week 30 | 175.0 [54.0 to 229.0] | 23.0 [1.0 to 60.0] |  | 36.5 [1.0 to 93.0]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_TNF-α, Week 48 | 39.0 [1.5 to 99.5] | 31.0 [1.0 to 80.0] |  | 39.0 [1.0 to 163.0]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IFN- γ, Pre-vaccination | 26.0 [1.0 to 42.0] | 17.5 [1.0 to 64.0] | 22.0 [1.0 to 58.0] | 23.0 [1.0 to 55.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  CD40L_IFN- γ, Week 6 | 89.0 [44.0 to 192.0] | 76.0 [29.0 to 154.0] | 81.0 [36.0 to 176.5] | 31.0 [1.0 to 67.0]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ, Week 28 | 15.5 [1.0 to 45.0] | 1.0 [1.0 to 54.0] | 5.5 [1.0 to 50.0] | 23.0 [1.0 to 52.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_IFN- γ, Week 30 | 71.0 [22.0 to 177.0] | 22.0 [1.0 to 45.0] |  | 28.0 [1.0 to 61.0]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_IFN- γ, Week 48 | 31.0 [1.0 to 46.0] | 7.5 [1.0 to 36.0] |  | 30.0 [1.0 to 57.0]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  TNF-α_IL-2, Week 6 | 22.0 [1.0 to 57.0] | 24.0 [1.0 to 55.0] | 22.5 [1.0 to 56.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IL-2, Week 28 | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 23.5] | 1.0 [1.0 to 16.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  TNF-α_IL-2, Week 30 | 7.5 [1.0 to 64.0] | 1.0 [1.0 to 16.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  TNF-α_IL-2, Week 48 | 1.0 [1.0 to 39.5] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IFN- γ, Pre-vaccination | 7.0 [1.0 to 37.0] | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 37.0] | 1.0 [1.0 to 48.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  TNF-α_IFN- γ, Week 6 | 35.0 [1.0 to 66.0] | 17.0 [1.0 to 58.0] | 27.5 [1.0 to 61.5] | 1.0 [1.0 to 48.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ, Week 28 | 9.5 [1.0 to 31.0] | 1.0 [1.0 to 34.0] | 1.0 [1.0 to 32.5] | 19.0 [1.0 to 40.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  TNF-α_IFN- γ, Week 30 | 22.0 [1.0 to 75.0] | 16.0 [1.0 to 41.0] |  | 1.0 [1.0 to 35.5]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  TNF-α_IFN- γ, Week 48 | 1.0 [1.0 to 32.5] | 1.0 [1.0 to 13.0] |  | 13.0 [1.0 to 41.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IL-2, Pre-vaccination | 23.0 [1.0 to 59.0] | 25.5 [1.0 to 68.0] | 23.0 [1.0 to 68.0] | 23.0 [1.0 to 70.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  CD40L_TNF-α_IL-2, Week 6 | 476.0 [182.0 to 1046.0] | 315.0 [129.0 to 623.0] | 346.5 [168.0 to 734.5] | 43.0 [1.0 to 91.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IL-2, Week 28 | 142.0 [65.0 to 353.0] | 95.0 [36.0 to 185.0] | 121.5 [40.5 to 227.0] | 49.0 [3.0 to 66.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_TNF-α_IL-2, Week 30 | 491.0 [226.0 to 878.0] | 91.0 [34.0 to 245.0] |  | 76.0 [22.0 to 101.0]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_TNF-α_IL-2, Week 48 | 185.0 [58.5 to 361.5] | 66.0 [2.0 to 120.0] |  | 20.0 [1.0 to 39.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 38.0] | 6.5 [1.0 to 28.0] | 1.0 [1.0 to 32.0] | 9.0 [1.0 to 24.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  CD40L_IFN- γ_IL-2, Week 6 | 141.0 [22.0 to 284.0] | 96.0 [46.0 to 239.0] | 123.5 [26.5 to 261.5] | 14.0 [1.0 to 43.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_IFN- γ_IL-2, Week 28 | 26.5 [1.0 to 45.0] | 17.0 [1.0 to 51.0] | 21.0 [1.0 to 51.0] | 1.0 [1.0 to 27.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_IFN- γ_IL-2, Week 30 | 131.0 [42.0 to 289.0] | 20.0 [1.0 to 57.0] |  | 1.0 [1.0 to 28.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_IFN- γ_IL-2, Week 48 | 21.0 [1.0 to 60.0] | 11.5 [1.0 to 51.0] |  | 1.0 [1.0 to 26.0]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 18.0 [1.0 to 35.0] | 1.5 [1.0 to 22.0] | 14.0 [1.0 to 31.0] | 27.0 [1.0 to 50.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  CD40L_TNF-α_IFN- γ, Week 6 | 141.0 [59.0 to 227.0] | 64.0 [24.0 to 113.0] | 90.0 [30.0 to 175.5] | 1.0 [1.0 to 54.0]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ, Week 28 | 14.5 [1.0 to 47.0] | 17.5 [1.0 to 42.0] | 15.5 [1.0 to 44.0] | 19.0 [1.0 to 77.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_TNF-α_IFN- γ, Week 30 | 71.5 [24.0 to 198.0] | 20.0 [1.0 to 44.0] |  | 22.0 [1.0 to 61.5]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_TNF-α_IFN- γ, Week 48 | 25.5 [1.0 to 56.5] | 21.5 [1.0 to 50.0] |  | 21.0 [1.0 to 54.0]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  TNF-α_IFN- γ_IL-2, Week 6 | 18.0 [1.0 to 45.0] | 1.0 [1.0 to 31.0] | 7.0 [1.0 to 42.5] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 9.0] | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  TNF-α_IFN- γ_IL-2, Week 30 | 7.5 [1.0 to 51.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 41 | 38 | 79 | 37
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 29.0 [1.0 to 59.0] | 14.0 [1.0 to 46.0] | 20.0 [1.0 to 55.0] | 23.0 [1.0 to 70.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 35 | 37 | 72 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 371.0 [203.0 to 837.0] | 262.0 [128.0 to 665.0] | 337.0 [131.0 to 747.5] | 56.0 [14.0 to 108.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 34 | 42 | 76 | 37
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 100.5 [36.0 to 192.0] | 70.0 [1.0 to 172.0] | 85.5 [29.0 to 182.0] | 18.0 [1.0 to 55.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 38 | 37 | 0 | 36
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 459.5 [198.0 to 963.0] | 48.0 [6.0 to 164.0] |  | 34.5 [2.0 to 86.5]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 96.0 [21.0 to 262.5] | 58.0 [1.0 to 121.0] |  | 33.0 [1.0 to 55.0]

43. Secondary Outcome: Cytokine Expression Profile of F4co-Computed CD8+ T Cells
Description: The cytokine co-expression profile was defined by the frequency of F4co-Computed CD8+ T-cells [Frequency of CD8+ T cells expressing markers in the response to the F4co fusion protein was estimated by adding individual frequencies of CD8+ T-cells to each of the 4 antigens (Nef, p17, p24, RT)] expressing CD40L and/or IL-2 and/or TNF-α and/or IFN-γ.
Time Frame: as for outcome 32
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects for whom CMI assay or humoral results were available against at least one study vaccine antigen component after vaccination.
Measure: Median (Inter-Quartile Range); unit: F4co-Computed CD8+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
F4co-Computed CD8+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L, Pre-vaccination | 79.5 [4.0 to 264.0] | 204.0 [20.0 to 367.0] | 100.0 [4.0 to 281.0] | 223.0 [39.0 to 377.0]
  CD40L, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L, Week 6 | 76.0 [5.0 to 185.0] | 110.5 [18.5 to 376.5] | 96.5 [5.5 to 284.5] | 179.5 [21.0 to 265.5]
  CD40L, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L, Week 28 | 167.0 [85.0 to 222.0] | 200.0 [28.5 to 349.0] | 174.0 [55.0 to 275.0] | 108.0 [34.0 to 233.0]
  CD40L, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  CD40L, Week 30 | 197.5 [24.0 to 421.0] | 143.0 [24.0 to 363.0] |  | 95.0 [18.0 to 282.0]
  CD40L, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L, Week 48 | 83.0 [4.0 to 296.0] | 64.0 [4.0 to 224.5] |  | 66.0 [4.0 to 320.0]
  IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IL-2, Pre-vaccination | 71.0 [4.0 to 190.0] | 98.0 [18.0 to 269.0] | 83.0 [7.0 to 236.0] | 81.0 [4.0 to 159.0]
  IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  IL-2, Week 6 | 93.5 [25.5 to 266.0] | 149.0 [51.0 to 265.0] | 119.5 [42.0 to 266.0] | 50.5 [4.0 to 143.0]
  IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IL-2, Week 28 | 192.0 [4.0 to 281.0] | 114.5 [41.0 to 247.5] | 124.0 [20.0 to 272.0] | 80.0 [6.0 to 175.0]
  IL-2, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  IL-2, Week 30 | 80.5 [11.0 to 162.0] | 152.0 [44.0 to 278.0] |  | 74.5 [25.0 to 221.0]
  IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  IL-2, Week 48 | 84.0 [4.0 to 278.0] | 83.5 [6.5 to 155.0] |  | 179.0 [18.0 to 315.0]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α, Pre-vaccination | 183.5 [74.0 to 434.0] | 213.0 [119.0 to 431.0] | 192.0 [82.0 to 434.0] | 314.0 [148.0 to 621.0]
  TNF-α, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  TNF-α, Week 6 | 227.0 [24.0 to 326.0] | 267.5 [144.5 to 543.5] | 244.0 [76.0 to 422.5] | 242.5 [94.0 to 585.5]
  TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α, Week 28 | 195.0 [44.0 to 484.0] | 158.5 [66.0 to 308.5] | 178.0 [66.0 to 454.0] | 227.0 [90.0 to 561.0]
  TNF-α, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  TNF-α, Week 30 | 176.0 [19.0 to 346.0] | 179.0 [22.0 to 416.0] |  | 240.0 [112.0 to 600.0]
  TNF-α, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  TNF-α, Week 48 | 246.0 [82.0 to 463.0] | 200.5 [30.0 to 527.5] |  | 273.0 [21.0 to 508.0]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ, Pre-vaccination | 13049.5 [8790.0 to 23850.0] | 16362.0 [10584.0 to 34174.0] | 15324.0 [8820.0 to 27122.0] | 21932.0 [11820.0 to 34367.0]
  IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  IFN- γ, Week 6 | 15467.0 [8103.0 to 20814.0] | 17126.0 [9396.5 to 35148.0] | 16697.0 [8830.5 to 22174.0] | 25219.0 [14676.0 to 39710.0]
  IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ, Week 28 | 16351.0 [10308.0 to 26108.0] | 14143.0 [8982.0 to 30999.5] | 14770.0 [9056.0 to 27519.0] | 21406.0 [14414.0 to 31530.0]
  IFN- γ, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  IFN- γ, Week 30 | 13512.0 [8067.0 to 20647.0] | 14730.0 [8580.0 to 31970.0] |  | 25319.5 [14013.0 to 32660.0]
  IFN- γ, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  IFN- γ, Week 48 | 14423.0 [7680.0 to 25368.0] | 18658.0 [9160.5 to 27347.0] |  | 20890.0 [12037.0 to 29108.0]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IL-2, Pre-vaccination | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_IL-2, Week 6 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IL-2, Week 28 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  CD40L_IL-2, Week 30 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 16.0]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_IL-2, Week 48 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 4.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α, Pre-vaccination | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 14.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 22.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_TNF-α, Week 6 | 4.0 [4.0 to 17.0] | 4.0 [4.0 to 16.0] | 4.0 [4.0 to 16.0] | 4.0 [4.0 to 14.5]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α, Week 28 | 4.0 [4.0 to 12.0] | 4.0 [4.0 to 14.0] | 4.0 [4.0 to 12.0] | 4.0 [4.0 to 4.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  CD40L_TNF-α, Week 30 | 4.0 [4.0 to 25.0] | 4.0 [4.0 to 15.0] |  | 4.0 [4.0 to 17.0]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_TNF-α, Week 48 | 4.0 [4.0 to 22.0] | 4.0 [4.0 to 20.0] |  | 4.0 [4.0 to 19.0]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ, Pre-vaccination | 19.5 [4.0 to 42.0] | 21.0 [4.0 to 60.0] | 21.0 [4.0 to 51.0] | 35.0 [4.0 to 73.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_IFN- γ, Week 6 | 27.0 [4.0 to 63.5] | 24.0 [4.0 to 52.0] | 25.0 [4.0 to 57.5] | 25.5 [10.0 to 57.0]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ, Week 28 | 23.0 [4.0 to 53.0] | 19.0 [4.0 to 38.0] | 21.0 [4.0 to 44.0] | 22.0 [13.0 to 46.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  CD40L_IFN- γ, Week 30 | 17.0 [4.0 to 37.0] | 4.0 [4.0 to 32.0] |  | 45.5 [19.0 to 82.0]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_IFN- γ, Week 48 | 31.0 [4.0 to 46.0] | 21.5 [4.0 to 45.0] |  | 28.0 [4.0 to 53.0]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IL-2, Pre-vaccination | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  TNF-α_IL-2, Week 6 | 4.0 [4.0 to 9.5] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 20.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IL-2, Week 28 | 4.0 [4.0 to 15.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  TNF-α_IL-2, Week 30 | 4.0 [4.0 to 25.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 15.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  TNF-α_IL-2, Week 48 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 16.5] |  | 4.0 [4.0 to 15.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ_IL-2, Pre-vaccination | 72.0 [21.0 to 191.0] | 102.0 [34.0 to 202.0] | 84.0 [28.0 to 202.0] | 117.0 [61.0 to 380.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  IFN- γ_IL-2, Week 6 | 70.0 [19.5 to 139.5] | 111.0 [33.0 to 204.0] | 84.5 [25.5 to 152.5] | 119.0 [39.5 to 507.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ_IL-2, Week 28 | 76.0 [21.0 to 149.0] | 66.5 [32.0 to 245.5] | 71.0 [23.0 to 229.0] | 100.0 [35.0 to 208.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  IFN- γ_IL-2, Week 30 | 51.0 [19.0 to 137.0] | 103.0 [25.0 to 213.0] |  | 74.5 [38.0 to 298.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  IFN- γ_IL-2, Week 48 | 68.0 [20.0 to 168.0] | 80.0 [29.0 to 192.5] |  | 81.0 [19.0 to 257.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ, Pre-vaccination | 1049.5 [539.0 to 2678.0] | 1820.0 [841.0 to 2671.0] | 1469.0 [572.0 to 2678.0] | 2095.0 [1062.0 to 4440.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  TNF-α_IFN- γ, Week 6 | 957.5 [476.0 to 2395.0] | 1864.5 [1197.5 to 2480.5] | 1610.5 [777.5 to 2458.5] | 2199.0 [1184.0 to 5725.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ, Week 28 | 1563.0 [590.0 to 2732.0] | 1782.5 [629.5 to 3126.5] | 1563.0 [622.0 to 2941.0] | 2012.0 [921.0 to 4006.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  TNF-α_IFN- γ, Week 30 | 985.0 [560.0 to 1981.0] | 1904.0 [706.0 to 3290.0] |  | 2260.0 [826.0 to 5091.0]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  TNF-α_IFN- γ, Week 48 | 993.0 [460.0 to 2222.0] | 1900.0 [764.5 to 3052.5] |  | 1787.0 [843.0 to 5013.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IL-2, Pre-vaccination | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_TNF-α_IL-2, Week 6 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IL-2, Week 28 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  CD40L_TNF-α_IL-2, Week 30 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_TNF-α_IL-2, Week 48 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 4.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ_IL-2, Pre-vaccination | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_IFN- γ_IL-2, Week 6 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ_IL-2, Week 28 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  CD40L_IFN- γ_IL-2, Week 30 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 4.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_IFN- γ_IL-2, Week 48 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 4.0 [4.0 to 20.0] | 4.0 [4.0 to 10.0] | 4.0 [4.0 to 16.0] | 4.0 [4.0 to 36.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_TNF-α_IFN- γ, Week 6 | 4.0 [4.0 to 11.5] | 4.0 [4.0 to 9.5] | 4.0 [4.0 to 10.5] | 4.0 [4.0 to 27.5]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ, Week 28 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 7.5] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 15.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  CD40L_TNF-α_IFN- γ, Week 30 | 4.0 [4.0 to 15.0] | 4.0 [4.0 to 17.0] |  | 4.5 [4.0 to 23.0]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_TNF-α_IFN- γ, Week 48 | 4.0 [4.0 to 19.0] | 4.0 [4.0 to 9.0] |  | 17.0 [4.0 to 37.0]
  TNF-α_IFN_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN_IL-2, Pre-vaccination | 17.0 [4.0 to 50.0] | 36.0 [4.0 to 97.0] | 30.0 [4.0 to 72.0] | 40.0 [4.0 to 125.0]
  TNF-α_IFN_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  TNF-α_IFN_IL-2, Week 6 | 9.5 [4.0 to 41.0] | 18.5 [4.0 to 65.0] | 16.0 [4.0 to 58.0] | 58.0 [11.5 to 176.5]
  TNF-α_IFN_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN_IL-2, Week 28 | 15.0 [4.0 to 52.0] | 19.0 [4.0 to 68.0] | 17.0 [4.0 to 56.0] | 21.0 [4.0 to 117.0]
  TNF-α_IFN_IL-2, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  TNF-α_IFN_IL-2, Week 30 | 4.0 [4.0 to 27.0] | 22.0 [4.0 to 126.0] |  | 30.5 [12.0 to 134.0]
  TNF-α_IFN_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  TNF-α_IFN_IL-2, Week 48 | 33.0 [4.0 to 54.0] | 19.5 [4.0 to 46.0] |  | 26.0 [4.0 to 62.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 34 | 35 | 0 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 4.0 [4.0 to 25.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 4.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 36 | 0 | 31
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] |  | 4.0 [4.0 to 4.0]

44. Secondary Outcome: Cytokine Expression Profile of Nef Antigen-specific CD8+ T-cells
Description: The cytokine co-expression profile was defined by the frequency of Nef-specific CD8+ T-cells expressing CD40L and/or IL-2 and/or TNF-α and/or IFN-γ.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: Nef-specific CD8+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
Nef-specific CD8+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L, Pre-vaccination | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 65.0] | 1.0 [1.0 to 51.0] | 51.0 [1.0 to 143.0]
  CD40L, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L, Week 6 | 1.0 [1.0 to 78.0] | 1.0 [1.0 to 90.0] | 1.0 [1.0 to 84.5] | 1.0 [1.0 to 99.5]
  CD40L, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L, Week 28 | 16.0 [1.0 to 94.0] | 12.5 [1.0 to 91.5] | 16.0 [1.0 to 94.0] | 1.0 [1.0 to 35.0]
  CD40L, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  CD40L, Week 30 | 5.0 [1.0 to 111.0] | 1.0 [1.0 to 80.0] |  | 1.0 [1.0 to 40.0]
  CD40L, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L, Week 48 | 1.0 [1.0 to 39.0] | 1.0 [1.0 to 48.0] |  | 1.0 [1.0 to 65.0]
  IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IL-2, Pre-vaccination | 1.0 [1.0 to 32.0] | 4.0 [1.0 to 55.0] | 1.0 [1.0 to 53.0] | 1.0 [1.0 to 37.0]
  IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  IL-2, Week 6 | 1.0 [1.0 to 73.0] | 6.0 [1.0 to 83.0] | 1.0 [1.0 to 75.0] | 1.0 [1.0 to 23.5]
  IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IL-2, Week 28 | 1.0 [1.0 to 31.0] | 14.0 [1.0 to 69.5] | 1.0 [1.0 to 61.0] | 19.0 [1.0 to 100.0]
  IL-2, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  IL-2, Week 30 | 1.0 [1.0 to 44.0] | 35.0 [1.0 to 89.0] |  | 1.0 [1.0 to 79.0]
  IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  IL-2, Week 48 | 1.0 [1.0 to 42.0] | 1.0 [1.0 to 31.0] |  | 4.5 [1.0 to 66.5]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α, Pre-vaccination | 1.0 [1.0 to 67.0] | 21.0 [1.0 to 81.0] | 1.0 [1.0 to 75.0] | 39.0 [1.0 to 187.0]
  TNF-α, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  TNF-α, Week 6 | 32.0 [1.0 to 78.5] | 31.5 [1.0 to 119.5] | 32.0 [1.0 to 94.0] | 42.5 [1.0 to 119.0]
  TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α, Week 28 | 12.0 [1.0 to 84.0] | 9.5 [1.0 to 64.0] | 12.0 [1.0 to 72.0] | 29.0 [1.0 to 119.0]
  TNF-α, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  TNF-α, Week 30 | 1.0 [1.0 to 83.0] | 1.0 [1.0 to 63.0] |  | 50.0 [1.0 to 143.0]
  TNF-α, Week 48: number analyzed (Participants) | 36 | 40 | 0 | 32
  TNF-α, Week 48 | 18.0 [1.0 to 77.5] | 11.0 [1.0 to 153.0] |  | 26.5 [1.0 to 142.5]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ, Pre-vaccination | 2947.0 [1230.0 to 5976.0] | 2150.0 [1020.0 to 7966.0] | 2646.0 [1049.0 to 6678.0] | 3224.0 [1607.0 to 8951.0]
  IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  IFN- γ, Week 6 | 2942.0 [853.0 to 5634.0] | 2951.0 [1199.5 to 8049.0] | 2942.0 [906.0 to 6203.0] | 4330.0 [2055.0 to 9013.0]
  IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ, Week 28 | 2396.0 [907.0 to 5646.0] | 2850.0 [996.0 to 7154.0] | 2748.0 [959.0 to 6291.0] | 3449.0 [1880.0 to 7427.0]
  IFN- γ, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  IFN- γ, Week 30 | 2586.0 [969.0 to 4509.0] | 2778.0 [1213.0 to 7998.0] |  | 3469.0 [2069.0 to 8384.0]
  IFN- γ, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  IFN- γ, Week 48 | 2236.5 [862.0 to 4932.5] | 2228.0 [961.0 to 6537.0] |  | 3584.0 [2034.5 to 6793.5]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  CD40L_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_TNF-α, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  CD40L_TNF-α, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_TNF-α, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ, Pre-vaccination | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 13.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_IFN- γ, Week 6 | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 7.5] | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 17.5]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ, Week 28 | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 13.5] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 14.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  CD40L_IFN- γ, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 16.0]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_IFN- γ, Week 48 | 1.0 [1.0 to 6.5] | 1.0 [1.0 to 14.0] |  | 1.0 [1.0 to 7.5]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  TNF-α_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  TNF-α_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  TNF-α_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 39.0] | 1.0 [1.0 to 82.0] | 1.0 [1.0 to 59.0] | 16.0 [1.0 to 55.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 27.5] | 11.5 [1.0 to 41.0] | 1.0 [1.0 to 34.0] | 22.5 [1.0 to 46.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 39.0] | 19.5 [1.0 to 71.0] | 17.0 [1.0 to 55.0] | 13.0 [1.0 to 48.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 37.0] | 18.0 [1.0 to 65.0] |  | 12.5 [1.0 to 58.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  IFN- γ_IL-2, Week 48 | 8.0 [1.0 to 38.5] | 19.0 [1.0 to 62.0] |  | 1.0 [1.0 to 34.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ, Pre-vaccination | 157.5 [56.0 to 378.0] | 174.0 [90.0 to 547.0] | 160.0 [75.0 to 383.0] | 259.0 [124.0 to 1318.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  TNF-α_IFN- γ, Week 6 | 152.5 [43.0 to 321.5] | 216.5 [64.5 to 487.0] | 156.5 [46.5 to 407.5] | 345.5 [210.5 to 1302.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ, Week 28 | 161.0 [39.0 to 369.0] | 191.5 [65.5 to 517.5] | 175.0 [61.0 to 515.0] | 333.0 [145.0 to 1010.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  TNF-α_IFN- γ, Week 30 | 138.0 [34.0 to 333.0] | 256.0 [79.0 to 510.0] |  | 292.5 [120.0 to 1380.0]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  TNF-α_IFN- γ, Week 48 | 110.0 [33.0 to 324.5] | 156.0 [48.0 to 553.0] |  | 293.5 [62.0 to 962.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_TNF-α_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  CD40L_TNF-α_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_TNF-α_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  CD40L_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_TNF-α_IFN- γ, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  CD40L_TNF-α_IFN- γ, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 21.0]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 7.0 [1.0 to 22.5]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 9.0] | 1.0 [1.0 to 21.5] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 19.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 13.0] |  | 1.0 [1.0 to 26.0]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 12.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 35 | 0 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]

45. Secondary Outcome: Cytokine Expression Profile of P17 Antigen-specific CD8+ T-cells
Description: The cytokine co-expression profile was defined by the frequency of P17-specific CD8+ T-cells expressing CD40L and/or IL-2 and/or TNF-α and/or IFN-γ.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: P17-specific CD8+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
P17-specific CD8+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L, Pre-vaccination | 1.0 [1.0 to 66.0] | 9.0 [1.0 to 76.0] | 7.0 [1.0 to 74.0] | 20.0 [1.0 to 111.0]
  CD40L, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L, Week 6 | 1.0 [1.0 to 24.0] | 23.0 [1.0 to 113.5] | 2.0 [1.0 to 66.0] | 17.0 [1.0 to 103.5]
  CD40L, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L, Week 28 | 15.0 [1.0 to 112.0] | 42.5 [1.0 to 95.0] | 40.0 [1.0 to 99.0] | 4.0 [1.0 to 66.0]
  CD40L, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  CD40L, Week 30 | 1.0 [1.0 to 95.0] | 3.0 [1.0 to 100.5] |  | 1.0 [1.0 to 38.0]
  CD40L, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L, Week 48 | 1.0 [1.0 to 32.0] | 1.0 [1.0 to 59.0] |  | 1.0 [1.0 to 85.5]
  IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IL-2, Pre-vaccination | 1.0 [1.0 to 63.0] | 29.0 [1.0 to 79.0] | 7.0 [1.0 to 74.0] | 1.0 [1.0 to 57.0]
  IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  IL-2, Week 6 | 17.0 [1.0 to 80.0] | 16.0 [1.0 to 41.5] | 17.0 [1.0 to 51.0] | 4.5 [1.0 to 34.5]
  IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IL-2, Week 28 | 19.0 [1.0 to 83.0] | 37.5 [1.0 to 80.0] | 37.0 [1.0 to 83.0] | 1.0 [1.0 to 81.0]
  IL-2, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  IL-2, Week 30 | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 65.5] |  | 22.0 [1.0 to 57.0]
  IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IL-2, Week 48 | 2.0 [1.0 to 73.0] | 1.0 [1.0 to 35.0] |  | 21.0 [1.0 to 87.0]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α, Pre-vaccination | 11.5 [1.0 to 64.0] | 27.0 [1.0 to 69.0] | 13.0 [1.0 to 69.0] | 29.0 [1.0 to 133.0]
  TNF-α, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  TNF-α, Week 6 | 25.0 [1.0 to 76.0] | 39.5 [1.0 to 79.0] | 29.0 [1.0 to 76.0] | 19.0 [1.0 to 134.0]
  TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α, Week 28 | 1.0 [1.0 to 61.0] | 6.0 [1.0 to 52.5] | 5.0 [1.0 to 60.0] | 1.0 [1.0 to 77.0]
  TNF-α, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  TNF-α, Week 30 | 2.5 [1.0 to 59.0] | 1.0 [1.0 to 39.5] |  | 11.0 [1.0 to 116.0]
  TNF-α, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α, Week 48 | 11.0 [1.0 to 71.0] | 17.0 [1.0 to 86.0] |  | 1.0 [1.0 to 52.5]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ, Pre-vaccination | 497.0 [21.0 to 1794.0] | 901.0 [115.0 to 2700.0] | 811.0 [83.0 to 2603.0] | 1617.0 [524.0 to 6545.0]
  IFN- γ, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  IFN- γ, Week 6 | 642.0 [69.0 to 2471.0] | 1144.0 [207.0 to 3376.0] | 733.0 [112.0 to 3154.0] | 1450.5 [550.0 to 5866.0]
  IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ, Week 28 | 694.0 [35.0 to 2002.0] | 1070.0 [169.5 to 2712.0] | 880.0 [58.0 to 2404.0] | 994.0 [378.0 to 3542.0]
  IFN- γ, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  IFN- γ, Week 30 | 276.0 [61.0 to 2387.0] | 1199.5 [230.5 to 2718.0] |  | 1279.0 [279.0 to 4396.0]
  IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IFN- γ, Week 48 | 406.0 [58.0 to 1670.0] | 1049.0 [100.0 to 2990.0] |  | 1059.0 [190.5 to 4540.5]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  CD40L_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_TNF-α, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  CD40L_TNF-α, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 19.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_IFN- γ, Week 6 | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 5.0]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 12.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  CD40L_IFN- γ, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 16.0]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IFN- γ, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 15.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  TNF-α_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  TNF-α_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 42.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 3.0] | 7.0 [1.0 to 32.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 19.5] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 30.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 16.5] |  | 1.0 [1.0 to 22.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 25.0] |  | 1.0 [1.0 to 15.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ, Pre-vaccination | 47.0 [1.0 to 158.0] | 60.0 [1.0 to 179.0] | 49.0 [1.0 to 173.0] | 164.0 [32.0 to 682.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  TNF-α_IFN- γ, Week 6 | 52.0 [1.0 to 173.0] | 107.0 [1.0 to 346.0] | 66.0 [1.0 to 268.0] | 130.0 [17.5 to 707.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ, Week 28 | 69.0 [1.0 to 146.0] | 61.0 [1.0 to 238.0] | 63.0 [1.0 to 228.0] | 110.0 [1.0 to 468.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  TNF-α_IFN- γ, Week 30 | 67.5 [1.0 to 140.0] | 76.5 [16.5 to 299.5] |  | 128.0 [4.0 to 410.0]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IFN- γ, Week 48 | 66.0 [1.0 to 148.0] | 111.0 [1.0 to 217.0] |  | 130.0 [19.5 to 541.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_TNF-α_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  CD40L_TNF-α_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  CD40L_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_TNF-α_IFN- γ, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  CD40L_TNF-α_IFN- γ, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 13.0]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 13.5]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 11.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 14.0]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 14.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 34 | 36 | 0 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]

46. Secondary Outcome: Cytokine Expression Profile of P24 Antigen-specific CD8+ T-cells
Description: The cytokine co-expression profile was defined by the frequency of P24-specific CD8+ T-cells expressing CD40L and/or IL-2 and/or TNF-α and/or IFN-γ.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: P24-specific CD8+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
P24-specific CD8+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L, Pre-vaccination | 1.0 [1.0 to 64.0] | 26.0 [1.0 to 110.0] | 3.0 [1.0 to 88.0] | 54.0 [1.0 to 86.0]
  CD40L, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L, Week 6 | 1.0 [1.0 to 9.0] | 10.0 [1.0 to 110.5] | 1.0 [1.0 to 74.0] | 26.5 [1.0 to 74.5]
  CD40L, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L, Week 28 | 1.0 [1.0 to 42.0] | 25.5 [1.0 to 129.0] | 7.0 [1.0 to 89.0] | 28.0 [1.0 to 76.0]
  CD40L, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L, Week 30 | 38.0 [1.0 to 147.0] | 18.0 [1.0 to 80.0] |  | 1.5 [1.0 to 105.0]
  CD40L, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L, Week 48 | 1.0 [1.0 to 85.0] | 1.0 [1.0 to 78.0] |  | 1.0 [1.0 to 77.0]
  IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IL-2, Pre-vaccination | 1.0 [1.0 to 31.0] | 2.0 [1.0 to 38.0] | 1.0 [1.0 to 37.0] | 1.0 [1.0 to 20.0]
  IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  IL-2, Week 6 | 1.0 [1.0 to 69.0] | 5.5 [1.0 to 69.0] | 2.0 [1.0 to 69.0] | 1.0 [1.0 to 19.0]
  IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IL-2, Week 28 | 1.0 [1.0 to 64.0] | 21.5 [1.0 to 51.5] | 12.0 [1.0 to 55.0] | 1.0 [1.0 to 41.0]
  IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  IL-2, Week 30 | 8.0 [1.0 to 54.0] | 35.5 [1.0 to 75.0] |  | 1.0 [1.0 to 29.0]
  IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IL-2, Week 48 | 1.0 [1.0 to 64.0] | 4.0 [1.0 to 47.0] |  | 11.0 [1.0 to 62.5]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α, Pre-vaccination | 54.5 [1.0 to 109.0] | 50.0 [1.0 to 139.0] | 51.0 [1.0 to 131.0] | 89.0 [12.0 to 178.0]
  TNF-α, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  TNF-α, Week 6 | 37.0 [1.0 to 111.0] | 82.5 [4.5 to 175.0] | 71.0 [1.0 to 154.0] | 40.0 [4.0 to 128.0]
  TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α, Week 28 | 69.0 [1.0 to 129.0] | 40.5 [1.0 to 70.0] | 47.0 [1.0 to 97.0] | 48.0 [1.0 to 111.0]
  TNF-α, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  TNF-α, Week 30 | 29.0 [1.0 to 165.0] | 19.0 [1.0 to 103.0] |  | 74.5 [1.0 to 154.0]
  TNF-α, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α, Week 48 | 53.0 [1.0 to 140.0] | 37.0 [1.0 to 135.0] |  | 17.5 [1.0 to 182.5]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ, Pre-vaccination | 4897.0 [2034.0 to 7095.0] | 6910.0 [1140.0 to 11555.0] | 5933.0 [1361.0 to 10100.0] | 6749.0 [2530.0 to 17157.0]
  IFN- γ, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  IFN- γ, Week 6 | 4570.0 [1899.0 to 7039.0] | 5096.0 [1217.5 to 13414.5] | 4657.0 [1458.0 to 9252.0] | 9141.5 [2594.0 to 19732.5]
  IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ, Week 28 | 5862.0 [1562.0 to 7767.0] | 4345.0 [1216.5 to 10098.0] | 5268.0 [1444.0 to 9807.0] | 6198.0 [2202.0 to 17804.0]
  IFN- γ, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  IFN- γ, Week 30 | 5056.0 [1670.0 to 8265.0] | 4358.0 [960.0 to 11810.5] |  | 7770.0 [3089.0 to 18585.0]
  IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IFN- γ, Week 48 | 5122.0 [1729.0 to 8072.0] | 4974.0 [1572.0 to 9962.0] |  | 6070.0 [1588.5 to 17183.0]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_TNF-α, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_TNF-α, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ, Pre-vaccination | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 28.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_IFN- γ, Week 6 | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 30.5]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ, Week 28 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 7.5] | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 22.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_IFN- γ, Week 30 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 8.5] |  | 11.5 [1.0 to 42.0]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IFN- γ, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 17.0] |  | 1.0 [1.0 to 14.5]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  TNF-α_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  TNF-α_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ_IL-2, Pre-vaccination | 7.5 [1.0 to 47.0] | 26.0 [1.0 to 61.0] | 19.0 [1.0 to 60.0] | 28.0 [1.0 to 159.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 29.0] | 19.0 [1.0 to 71.5] | 1.0 [1.0 to 54.0] | 22.0 [1.0 to 215.5]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 36.0] | 20.5 [1.0 to 41.5] | 18.0 [1.0 to 38.0] | 22.0 [1.0 to 92.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  IFN- γ_IL-2, Week 30 | 11.0 [1.0 to 39.0] | 18.5 [1.0 to 61.5] |  | 25.0 [1.0 to 132.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 36.0] | 2.0 [1.0 to 56.0] |  | 1.0 [1.0 to 92.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ, Pre-vaccination | 291.5 [182.0 to 693.0] | 586.0 [139.0 to 1045.0] | 319.0 [160.0 to 919.0] | 705.0 [137.0 to 1290.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  TNF-α_IFN- γ, Week 6 | 236.0 [134.0 to 674.0] | 390.5 [167.0 to 1087.5] | 283.0 [139.0 to 884.0] | 751.5 [143.5 to 2159.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ, Week 28 | 471.0 [195.0 to 1020.0] | 492.0 [103.5 to 1038.0] | 471.0 [118.0 to 1022.0] | 484.0 [118.0 to 1604.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  TNF-α_IFN- γ, Week 30 | 246.0 [111.0 to 542.0] | 313.5 [93.5 to 1256.0] |  | 761.0 [177.0 to 1630.0]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IFN- γ, Week 48 | 299.0 [119.0 to 865.0] | 423.0 [128.0 to 1030.0] |  | 497.0 [193.5 to 1362.5]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_TNF-α_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_TNF-α_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 17.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_TNF-α_IFN- γ, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 20.5]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_TNF-α_IFN- γ, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 11.0] |  | 1.0 [1.0 to 14.5]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 37.0]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 21.5] | 1.0 [1.0 to 21.0] | 8.5 [1.0 to 70.0]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 32.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 19.5] |  | 1.0 [1.0 to 27.0]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 9.0] |  | 1.0 [1.0 to 20.5]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 33 | 36 | 69 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 35 | 37 | 0 | 32
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]

47. Secondary Outcome: Cytokine Expression Profile of RT Antigen-specific CD8+ T-cells
Description: The cytokine co-expression profile was defined by the frequency of reverse transcriptase (RT)-specific CD8+ T-cells expressing CD40L and/or IL-2 and/or TNF-α and/or IFN-γ.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: RT-specific CD8+ T-cells/million cells
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 38 | 40 | 75 | 35
RT-specific CD8+ T-cells/million cells
  CD40L, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L, Pre-vaccination | 1.0 [1.0 to 67.0] | 60.0 [1.0 to 137.0] | 1.0 [1.0 to 90.0] | 12.0 [1.0 to 142.0]
  CD40L, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  CD40L, Week 6 | 1.0 [1.0 to 12.5] | 15.0 [1.0 to 97.0] | 1.0 [1.0 to 84.0] | 35.0 [1.0 to 62.0]
  CD40L, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L, Week 28 | 1.0 [1.0 to 50.0] | 1.0 [1.0 to 127.5] | 1.0 [1.0 to 76.0] | 1.0 [1.0 to 66.0]
  CD40L, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L, Week 30 | 19.0 [1.0 to 71.0] | 1.0 [1.0 to 88.0] |  | 1.0 [1.0 to 62.0]
  CD40L, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L, Week 48 | 1.0 [1.0 to 54.5] | 1.0 [1.0 to 94.0] |  | 1.0 [1.0 to 58.0]
  IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IL-2, Pre-vaccination | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 48.0] | 1.0 [1.0 to 48.0] | 1.0 [1.0 to 66.0]
  IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  IL-2, Week 6 | 1.0 [1.0 to 59.5] | 1.0 [1.0 to 77.5] | 1.0 [1.0 to 70.5] | 1.0 [1.0 to 35.0]
  IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IL-2, Week 28 | 1.0 [1.0 to 60.0] | 15.5 [1.0 to 72.0] | 13.0 [1.0 to 70.0] | 2.0 [1.0 to 44.0]
  IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  IL-2, Week 30 | 1.0 [1.0 to 44.0] | 21.5 [1.0 to 83.0] |  | 12.5 [1.0 to 55.0]
  IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  IL-2, Week 48 | 2.0 [1.0 to 61.5] | 1.0 [1.0 to 51.0] |  | 40.0 [1.0 to 109.0]
  TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α, Pre-vaccination | 71.5 [1.0 to 150.0] | 67.0 [12.0 to 143.0] | 68.0 [1.0 to 150.0] | 84.0 [35.0 to 196.0]
  TNF-α, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  TNF-α, Week 6 | 61.0 [1.0 to 125.5] | 70.0 [8.0 to 133.5] | 63.0 [1.0 to 127.0] | 82.0 [16.0 to 157.0]
  TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α, Week 28 | 42.0 [1.0 to 119.0] | 50.0 [1.0 to 162.5] | 48.0 [1.0 to 131.0] | 80.0 [1.0 to 187.0]
  TNF-α, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  TNF-α, Week 30 | 33.0 [1.0 to 102.0] | 76.0 [1.0 to 164.5] |  | 97.0 [1.0 to 187.0]
  TNF-α, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  TNF-α, Week 48 | 63.5 [1.0 to 158.0] | 63.0 [1.0 to 125.0] |  | 109.0 [1.0 to 193.0]
  IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ, Pre-vaccination | 3370.0 [1592.0 to 6581.0] | 2161.0 [1464.0 to 6962.0] | 3138.0 [1464.0 to 6784.0] | 3950.0 [1335.0 to 6877.0]
  IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  IFN- γ, Week 6 | 3474.0 [1187.5 to 6812.0] | 2885.0 [1774.0 to 6141.0] | 3050.5 [1453.0 to 6341.0] | 4012.0 [2452.0 to 8455.0]
  IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ, Week 28 | 5410.0 [1201.0 to 7637.0] | 2355.5 [1355.0 to 5886.0] | 3079.0 [1342.0 to 7349.0] | 3595.0 [1370.0 to 6370.0]
  IFN- γ, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  IFN- γ, Week 30 | 2959.0 [1287.0 to 7160.0] | 2824.5 [1767.0 to 5807.5] |  | 4000.0 [1730.0 to 7055.0]
  IFN- γ, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  IFN- γ, Week 48 | 3081.0 [1341.5 to 6169.0] | 3187.0 [1690.0 to 6150.0] |  | 4294.0 [1579.0 to 6806.0]
  CD40L_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  CD40L_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  CD40L_TNF-α, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_TNF-α, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_TNF-α, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ, Pre-vaccination | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  CD40L_IFN- γ, Week 6 | 1.0 [1.0 to 15.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ, Week 28 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_IFN- γ, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_IFN- γ, Week 48 | 1.0 [1.0 to 18.5] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 11.0]
  TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  TNF-α_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  TNF-α_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  TNF-α_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  IFN- γ_IL-2, Pre-vaccination | 14.5 [1.0 to 60.0] | 17.0 [1.0 to 54.0] | 17.0 [1.0 to 60.0] | 18.0 [1.0 to 64.0]
  IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 36.0] | 28.0 [6.0 to 48.5] | 23.5 [1.0 to 42.5] | 16.0 [1.0 to 47.0]
  IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  IFN- γ_IL-2, Week 28 | 16.0 [1.0 to 62.0] | 7.0 [1.0 to 55.0] | 13.0 [1.0 to 57.0] | 16.0 [1.0 to 50.0]
  IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 52.0] | 11.5 [1.0 to 54.5] |  | 19.0 [1.0 to 45.0]
  IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  IFN- γ_IL-2, Week 48 | 17.0 [1.0 to 36.5] | 8.0 [1.0 to 52.0] |  | 18.0 [1.0 to 47.0]
  TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ, Pre-vaccination | 271.0 [92.0 to 616.0] | 314.0 [119.0 to 814.0] | 300.0 [101.0 to 779.0] | 410.0 [89.0 to 782.0]
  TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  TNF-α_IFN- γ, Week 6 | 301.0 [78.5 to 1025.5] | 360.0 [178.5 to 831.0] | 339.0 [150.0 to 925.0] | 471.0 [149.0 to 925.0]
  TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ, Week 28 | 372.0 [129.0 to 1249.0] | 455.0 [118.0 to 843.0] | 454.0 [119.0 to 1080.0] | 366.0 [205.0 to 812.0]
  TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  TNF-α_IFN- γ, Week 30 | 232.0 [97.0 to 745.0] | 542.5 [183.0 to 1006.5] |  | 490.0 [207.0 to 1040.0]
  TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  TNF-α_IFN- γ, Week 48 | 250.5 [109.0 to 725.0] | 483.5 [166.0 to 1020.0] |  | 404.0 [174.0 to 725.0]
  CD40L_TNF-α_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  CD40L_TNF-α_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_TNF-α_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_TNF-α_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  CD40L_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  CD40L_TNF-α_IFN- γ, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_TNF-α_IFN- γ, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_TNF-α_IFN- γ, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 25.0]
  TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 16.5] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 21.0] | 10.0 [1.0 to 27.0]
  TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 16.0]
  TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 5.0 [1.0 to 26.5] |  | 1.0 [1.0 to 30.0]
  TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 10.5] | 1.0 [1.0 to 18.0] |  | 1.0 [1.0 to 17.0]
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination: number analyzed (Participants) | 38 | 37 | 75 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Pre-vaccination | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 6: number analyzed (Participants) | 32 | 36 | 68 | 33
  CD40L_TNF-α_IFN- γ_IL-2, Week 6 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 28: number analyzed (Participants) | 31 | 40 | 71 | 35
  CD40L_TNF-α_IFN- γ_IL-2, Week 28 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 30: number analyzed (Participants) | 35 | 36 | 0 | 34
  CD40L_TNF-α_IFN- γ_IL-2, Week 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]
  CD40L_TNF-α_IFN- γ_IL-2, Week 48: number analyzed (Participants) | 36 | 38 | 0 | 31
  CD40L_TNF-α_IFN- γ_IL-2, Week 48 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] |  | 1.0 [1.0 to 1.0]

48. Secondary Outcome: Number of Seropositive Subjects for Anti-P17 Antibodies
Description: Seropositivity rates for antibodies against P17 antigen were assessed using the Enzyme-Linked Immunosorbent Assay (ELISA), with a reference cut-off value greater than or equal to (≥) 187 milli-ELISA units per milliliter (mEL.U/mL).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 44 | 45 | 89 | 40
Participants
  Anti-P17, Pre-vaccination | 35 | 38 | 73 | 34
  Anti-P17, Week 6: number analyzed (Participants) | 44 | 43 | 87 | 40
  Anti-P17, Week 6 | 39 | 37 | 76 | 33
  Anti-P17, Week 28: number analyzed (Participants) | 44 | 45 | 89 | 39
  Anti-P17, Week 28 | 37 | 38 | 75 | 32
  Anti-P17, Week 30: number analyzed (Participants) | 43 | 42 | 0 | 38
  Anti-P17, Week 30 | 41 | 35 |  | 31
  Anti-P17, Week 48: number analyzed (Participants) | 39 | 43 | 0 | 37
  Anti-P17, Week 48 | 31 | 33 |  | 31

49. Secondary Outcome: Number of Seropositive Subjects for Anti-P24 Antibodies
Description: Seropositivity rates for antibodies against P24 antigen were assessed using the Enzyme-Linked Immunosorbent Assay (ELISA), with a reference cut-off value greater than or equal to (≥) 119 milli-ELISA units per milliliter (mEL.U/mL).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 44 | 45 | 89 | 40
Participants
  Anti-P24, Pre-vaccination | 42 | 45 | 87 | 38
  Anti-P24, Week 6: number analyzed (Participants) | 44 | 43 | 87 | 40
  Anti-P24, Week 6 | 43 | 43 | 86 | 38
  Anti-P24, Week 28: number analyzed (Participants) | 44 | 45 | 89 | 39
  Anti-P24, Week 28 | 43 | 44 | 87 | 37
  Anti-P24, Week 30: number analyzed (Participants) | 43 | 42 | 0 | 38
  Anti-P24, Week 30 | 43 | 41 |  | 36
  Anti-P24, Week 48: number analyzed (Participants) | 39 | 43 | 0 | 37
  Anti-P24, Week 48 | 39 | 42 |  | 35

50. Secondary Outcome: Number of Seropositive Subjects for Anti-Nef Antibodies
Description: Seropositivity rates for antibodies against Nef antigen were assessed using the Enzyme-Linked Immunosorbent Assay (ELISA), with a reference cut-off value greater than or equal to (≥) 494 milli-ELISA units per milliliter (mEL.U/mL).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 44 | 45 | 89 | 40
Participants
  Anti-Nef, Pre-vaccination | 22 | 28 | 50 | 21
  Anti-Nef, Week 6: number analyzed (Participants) | 44 | 43 | 87 | 40
  Anti-Nef, Week 6 | 38 | 35 | 73 | 17
  Anti-Nef, Week 28: number analyzed (Participants) | 44 | 45 | 89 | 39
  Anti-Nef, Week 28 | 24 | 31 | 55 | 20
  Anti-Nef, Week 30: number analyzed (Participants) | 43 | 42 | 0 | 38
  Anti-Nef, Week 30 | 42 | 28 |  | 20
  Anti-Nef, Week 48: number analyzed (Participants) | 39 | 43 | 0 | 37
  Anti-Nef, Week 48 | 33 | 27 |  | 18

51. Secondary Outcome: Number of Seropositive Subjects for Anti-RT Antibodies
Description: Seropositivity rates for antibodies against RT antigen were assessed using the Enzyme-Linked Immunosorbent Assay (ELISA), with a reference cut-off value greater than or equal to (≥) 125 milli-ELISA units per milliliter (mEL.U/mL).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 44 | 45 | 89 | 40
Participants
  Anti-RT, Pre-vaccination: number analyzed (Participants) | 40 | 42 | 82 | 39
  Anti-RT, Pre-vaccination | 40 | 42 | 82 | 39
  Anti-RT, Week 6: number analyzed (Participants) | 43 | 42 | 85 | 40
  Anti-RT, Week 6 | 43 | 42 | 85 | 40
  Anti-RT, Week 28: number analyzed (Participants) | 44 | 45 | 89 | 38
  Anti-RT, Week 28 | 44 | 45 | 89 | 38
  Anti-RT, Week 30: number analyzed (Participants) | 42 | 41 | 0 | 38
  Anti-RT, Week 30 | 42 | 41 |  | 38
  Anti-RT, Week 48: number analyzed (Participants) | 38 | 41 | 0 | 37
  Anti-RT, Week 48 | 38 | 41 |  | 37

52. Secondary Outcome: Number of Seropositive Subjects for Anti-F4co Antibodies
Description: Seropositivity rates for antibodies against F4co antigen were assessed using the Enzyme-Linked Immunosorbent Assay (ELISA), with a reference cut-off value greater than or equal to (≥) 42 milli-ELISA units per milliliter (mEL.U/mL).
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | 3D_HIV Group | 2D_HIV Group | HIV Group | Control Group
Number analyzed (Participants) | 44 | 45 | 89 | 40
Participants
  Anti-F4co, Pre-vaccination | 44 | 45 | 89 | 40
  Anti-F4co, Week 6: number analyzed (Participants) | 44 | 43 | 87 | 40
  Anti-F4co, Week 6 | 44 | 43 | 87 | 40
  Anti-F4co, Week 28: number analyzed (Participants) | 44 | 45 | 89 | 39
  Anti-F4co, Week 28 | 44 | 45 | 89 | 39
  Anti-F4co, Week 30: number analyzed (Participants) | 43 | 42 | 0 | 38
  Anti-F4co, Week 30 | 43 | 42 |  | 38
  Anti-F4co, Week 48: number analyzed (Participants) | 39 | 43 | 0 | 37
  Anti-F4co, Week 48 | 39 | 43 |  | 37

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 28-day (Days 0-27) post-vaccination period; SAEs: during the entire study period (Week 0 to Week 48).
Arm/Group | 3D_HIV Group | 2D_HIV Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/62 | 3/64 | 2/64
Other Adverse Events (participants affected / at risk) | 60/62 | 60/64 | 42/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3D_HIV Group (N=62) | 2D_HIV Group (N=64) | Control Group (N=64)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3D_HIV Group (N=62) | 2D_HIV Group (N=64) | Control Group (N=64)
Abdominal pain (Gastrointestinal disorders) | 13 (18) | 10 (13) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 11 (13) | 10 (11) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 18 (23) | 20 (29) | 15 (19)
Erythema (Skin and subcutaneous tissue disorders) | 18 (23) | 14 (19) | 0 (0)
Fatigue (General disorders) | 43 (83) | 39 (66) | 20 (34)
Headache (Nervous system disorders) | 32 (57) | 33 (57) | 22 (32)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 (21) | 20 (27) | 10 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 33 (61) | 33 (55) | 13 (21)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 17 (24) | 15 (18) | 8 (8)
Pain (General disorders) | 58 (146) | 57 (115) | 14 (20)
Pyrexia (General disorders) | 14 (18) | 9 (11) | 7 (8)
Swelling (General disorders) | 4 (6) | 8 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.